# Incidence of melanoma and non-melanoma skin cancer in people with vitiligo: A case-control study in the UK, 2009-2020: Statistical Analysis Plan and Protocol

| <b>Document version</b> | 1.3 |
|-------------------------|-------------|
| Date | 5 July 2021 |

## Contents

| List of abbreviations | 4 |
|---------------------------------------------------------------|----|
| 1. Introduction | 5 |
| 1.1 Background | 5 |
| 1.2. Purposes of analyses | 6 |
| 2. Study objectives and endpoints | 7 |
| 2.1 Study objectives | 7 |
| 2.2 Primary objectives | 7 |
| 2.3 Secondary objectives: | 7 |
| 2.4 Primary endpoint | 7 |
| 2.5 Secondary endpoints | 8 |
| 2.6 Other exploratory analyses | 8 |
| 3 General Study Design and Plan | 8 |
| 3.1 Study Design | 8 |
| 3.2 Data source and Read codes | 8 |
| 3.3 Data extraction | 8 |
| 3.4 Inclusion-Exclusion Criteria and General Study Population | 9 |
| Definition of vitiligo cases | 9 |
| 3.5 Baseline characteristics | 9 |
| 4 Sample size calculations | 10 |
| 5 Populations to be analysed | 10 |
| 5.1 Inclusion Criteria | 10 |
| 5.2 Exclusion Criteria | 10 |
| 5.3 Matching process | 10 |
| 6 Statistical Analysis | 11 |
| 6.1 Statistical principles | 11 |

| 6.2 Primary Endpoint Analysis | 11 |
|----------------------------------|----|
| 6.3 Secondary Objective Analysis | 12 |
| 6.4 Sensitivity analysis | 12 |
| 6.5 Missing data | 13 |
| 7 Study Limitations | 13 |
| 8 Statistical software | 13 |
| 9 Ethics | 14 |
| References | 15 |
| Appendix 1 | 17 |
| Appendix 2 | 32 |
| Appendix 3 | 33 |
| Appendix 4 | 36 |

# List of abbreviations

| Abbreviation | Full Form |
|---|---|
| ADEPT | Anonymised Data Ethics Protocols and Transparency |
| AK | Actinic keratoses |
| BCC | Basal cell carcinoma |
| BMI | Body mass index |
| CI | Confidence Interval |
| GEP | Good Epidemiological Practice |
| GP | General Practitioner |
| GPP | Guidelines for Good Pharmacoepidemiology Practices |
| HR | Hazard Ratio |
| IEA | International Epidemiological Association |
| IMD | Index of multiple deprivation |
| IQR | Interquartile range |
| ISPE | International Society for Pharmacoepidemiology |
| NMSC | Nonmelanoma skin cancers |
| OPCRD | Optimum Patient Care Research Database |
| RECORD | Reporting of studies conducted using observational routinely collected data |
| SCC | Squamous cell carcinoma |
| SD | Standard deviation |
| SES | Socio-economic status |
| UK | United Kingdom |
| UV | Ultraviolet |

### 1. Introduction

### 1.1 Background

Vitiligo is an acquired depigmenting cutaneous disease with an incidence of 0.5 to 2% worldwide. It is characterised by white patches of skin resulting from the destruction of melanocytes from the epidermis (1). Although the exact cause of the condition remains to be established, autoimmunity is an important hypothesis of the aetiology of vitiligo. It has been demonstrated that CD8+ T-cells play a major role in the destruction of melanocytes, through the recognition of melanocyte differentiation antigens (2).

Genetic studies of vitiligo have greatly advanced understanding of the pathobiology of the condition and provided insights regarding to susceptibility to skin cancer. Genome-wide association analyses have found that vitiligo is associated with polymorphisms in the TYR gene, which codes for tyrosinase, the main enzyme in melanin synthesis. The TYR allele that is associated with susceptibility to vitiligo may confer a degree of protection against melanoma because of the anti-tyrosinase immunity (3). In addition, human leukocyte antigen A2 which is the risk allele for the development of vitiligo was found to be associated with regressing melanoma, supporting the inverse relationship between vitiligo and melanoma (4).

Although the genetic and autoimmunity profiles in vitiligo may protect against the development of melanoma and nonmelanoma skin cancers (NMSC), an absence of melanin in lesional skin and prolonged phototherapy treatment may cause concern about the development of skin cancer in this population (5). In a retrospective cohort study of 479 patients with vitiligo, an overall higher incidence of NMSC in the white vitiligo cohort than the white US rates was reported (6). This finding was supported by a recent, nationwide, control-matched cohort study conducted in Korea assessing 131,245 patients. The authors reported that, taking into account of the important cofounders (e.g. ultraviolet treatment), people with vitiligo were 3.4 and 1.3 times more likely to get melanoma and nonmelanoma skin cancer (NMSC), respectively, than those without vitiligo (7).

In contrast to the above-mentioned studies, Teulings and colleagues (8), in a large comparative cohort, Dutch, survey-based study in 2013, found a 3-fold lower probability of developing melanoma and NMSC in those with vitiligo. Stratification of the results into subgroups of patients treated with narrowband ultraviolet (UV) B, and psoralen and UV-A did not find increased lifetime prevalence of melanoma or NMSC. A subsequent study conducted in Italy by Paradisi and colleagues (9) also reported that patients with vitiligo had a significantly lower probability of developing melanoma or NMSC than those with a non-dermatological condition. However, a markedly higher risk (14.1% vs 3.2%) was noted in patients treated with phototherapy compared with the control group.

Overall, the risk of melanoma and NMSC in vitiligo is still being debated and further research is needed in this field.

### 1.2. Purposes of analyses

To the best of our knowledge, there have not been any large population-based studies in the UK assessing the incidence of melanoma and NMSC in patients with vitiligo compared with people without the condition. The purpose of this study is therefore to fill this data gap, and to examine whether the susceptibility to melanoma and NMSC may vary between different patient subgroups, e.g. ethnicity, those who undergo phototherapy or treatment with the new targeted biologic immunosuppressive therapies. Such new insights will be valuable for clinicians in advising patients with vitiligo on sun-related behaviour and treatment options in the UK.

# 2. Study objectives and endpoints

# 2.1 Study objectives

The overall purpose of this study is to examine whether the risk of skin cancer is higher in people diagnosed with vitiligo compared to people without vitiligo.

### 2.2 Primary objectives

- Describe the risk of new onset skin cancer in adults diagnosed with vitiligo in a contemporary real-world population compared with matched controls without vitiligo.
- Describe the risk of new onset skin cancer in adults diagnosed with vitiligo by sociodemographic subgroups.

## 2.3 Secondary objectives:

- Describe the prevalence of skin cancer in adults diagnosed with vitiligo compared with matched controls without vitiligo.
- Describe the prevalence of individual skin cancer types in adults diagnosed with vitiligo compared with matched controls without vitiligo.
- Describe the risk of new onset actinic keratoses (AK) in adults diagnosed with vitiligo compared with matched controls without vitiligo.
- Examine the prevalence of AK in adults diagnosed with vitiligo compared with matched controls without vitiligo.

# 2.4 Primary endpoint

- The skin cancer outcome comprises of the composite of melanoma and NMSC.
   NMSC comprises squamous cell carcinoma (SCC) and basal cell carcinoma (BCC).
   When more than one of melanoma, SCC and BCC occur, the skin cancer diagnosis date will be the earliest of these cancers.
- The primary endpoint is time to first diagnosis of new onset skin cancer during the study follow up period.

### 2.5 Secondary endpoints

- The prevalence (those diagnosed prior to the study period) of any skin cancer and each individual skin cancer in each study group.
- The secondary endpoint for new onset AK is the time to first diagnosis of AK during the study follow up period.

### 2.6 Other exploratory analyses

If there is sufficient information in the primary care record, we will examine the possibility of comparing the primary endpoints in those people with a documented history of immunotherapy use (compared the those without) and those people with a documented history of phototherapy treatment (compared the those without). Data on phototherapy treatment may be insufficient to enable comparisons, if this is the case, this will be reported as a limitation of the study.

# 3 General Study Design and Plan

### 3.1 Study Design

A matched-cohort design will be used to compare the risk of new onset skin cancers. The study will use a case-control design to compare the prevalence of skin cancers.

#### 3.2 Data source and Read codes

This study will use routinely collected and collated data from the Optimum Patient Care Research Database (OPCRD). (10) This database incorporates pseudonymised primary care records from up to 700 GP practices distributed across England, Wales, Scotland and Northern Ireland. The current OPCRD cohort size is over 5 million actively registered people, and historic records available for 10.1 million people.

#### 3.3 Data extraction

Individual patient data is anonymised at the point of data extraction. Queries will be executed to extract relevant data from the OPCRD using the Read code listed in Appendix 1. All data will remain in anonymised form and will be held on a secure server. The data will not be used for any purposes other than for the research which is described in the

respective protocols and which has been approved by OPC. The sponsor, Pfizer Ltd, will not have access to the individual anonymised patient data.

### 3.4 Inclusion-Exclusion Criteria and General Study Population

### Definition of vitiligo cases

We will identify all people diagnosed with vitiligo using diagnostic Read and SNOMED CT codes which are specific to vitiligo (Appendix 1). A diagnostic algorithm will be used to facilitate robust case identification of vitiligo. This algorithm will identify anyone with a vitiligo specific diagnosis code followed by exclusion of anyone with a diagnosis code for an alternative depigmenting disorder coded within a one-year period (six months before or after their first vitiligo diagnosis code). The list of alternative depigmenting disorders is shown in Appendix 2. We will include people diagnosed with vitiligo prior to the study period (referred to as prevalent vitiligo) and people newly diagnosed with vitiligo during the study period (referred to as incident vitiligo) as vitiligo cases for the risk of new onset of skin cancers analysis. Only people with incident vitiligo will be included as cases in prevalence analysis.

The study index date for people diagnosed with vitiligo will be the latest of; the start date of follow-up (1st Jan 2010), date of registration with GP plus six months, or the date of diagnosis of vitiligo.

### 3.5 Baseline characteristics

A fully list of the study variables is provided in Appendix 3. Sociodemographic groups will be defined by age category (18-44, 45-64, ≥65), sex, socio-economic status (SES), and ethnicity. SES will be defined using the official national deprivation measure; index of multiple deprivation (IMD).(11) This will be calculated at the point of data extraction, using patient postcode, with the resultant scores stratified by deprivation quintile according to the national distribution. Ethnicity will be grouped into major ethnic groups to be consistent with the UK official census categories: White, Black African/Caribbean, Asian, Mixed, and Other(12, 13). Other clinical covariates comprised BMI category, smoking status, alcohol use, and common comorbidities (hypertension, hyperlipidaemia, type 2 diabetes, atrial fibrillation, angina, myocardial infarction, stroke, heart failure,

chronic kidney disease stages 3-5, chronic obstructive pulmonary disease, asthma, chronic liver disease, and dementia). These will be identified using clinical codes and test results recorded in the patient record.

## 4 Sample size calculations

No previous UK population-based studies have examined skin cancer risk in people with vitiligo to provide an estimation of effect size to inform our sample size calculation. Assuming 80% power, a 1:1 ratio of vitiligo cases to controls, and an overall probability of melanoma over the study period of 0.45% (a conservative estimate based on a previous analysis of melanoma incidence in the general population (14)) a sample size of 6,177 will be required to detect a minimum clinically relevant effect size of a 80% decreased risk of melanoma in the vitiligo cohort compared to population controls. We anticipate c.22,500 people in our study cohort will be defined as vitiligo cases, these will be 1:1 matched to population controls providing a study cohort well in excess of this required sample size.

# 5 Populations to be analysed

### **5.1 Inclusion Criteria**

All eligible adult patients (aged ≥18) registered with GP practices contributing data to OPCRD between January 1, 2010 and December 31, 2020, are eligible for inclusion in the study. People diagnosed with vitiligo prior to the study period (prevalent vitiligo) and people newly diagnosed with vitiligo during the study period (incident vitiligo) will be included as cases.

#### 5.2 Exclusion Criteria

People actively registered with the GP practice at that date without a history of vitiligo require a minimum one-year registration with their GP practice.

# 5.3 Matching process

Each adult with vitiligo (prevalent or incident) will be 1:1 matched at their index date using, nearest neighbour matching (30) with an unaffected control (people without vitiligo prior to or during the study period). Matching variables will comprise age, sex,

duration of practice registration and within primary care practice where numbers allow. After matching, the index date for each control will be set at the index date of their matched counterpart.

# **6 Statistical Analysis**

### 6.1 Statistical principles

The mean, standard deviation (sd) and any other statistical measures, will be reported to one decimal place. Continuous data will be summarised in the form of means, sd, median, interquartile range (IQR) and range as appropriate. Categorical data will be summarised using frequencies and proportions. Chi-squared and t-tests will be performed to compare the frequency of dichotomous variables and the values of continuous variables where relevant. 95% CIs will be reported for main effect sizes. Statistical significance will be assessed using p<0.05. Actual p-values will be reported except for p-values less than 3 decimal places which will be reported as "<0.001". P-values >0.1 will be reported to one decimal place, p-values between 0.01 and 0.1 will be reported to three decimal places.

The assessment of any associations with baseline characteristics and the primary endpoint will be assessed using Cox proportional hazards models. A standard set of features will be used in all multivariable models as listed in section 6.2.

Assumptions of statistical approaches will be assessed, and transformations used if necessary (although it is not anticipated that the data will violate model assumptions).

# **6.2 Primary Endpoint Analysis**

Risk of new onset skin cancer will be assessed prospectively in vitiligo cases (prevalent and incident vitiligo, refer to section 3.4) and matched controls from the index date. Endpoints will be identified using the clinical codes described in Appendix 4. Only vitiligo cases where both the vitiligo case and their matched counterpart do not have skin cancer at their index date will be included. We will then estimate risk of skin cancer over the study period starting from the index date for both vitiligo cases and controls, The end of follow-up will be defined as the earliest of the study end-date (December 31, 2020), the

date of patient transfer from an included general practice, date of death, or the date an individual first developed skin cancer. Risk of developing skin cancer will then be examined using time to failure analysis. Initially, unadjusted Cox proportional hazards models, stratified by matched set (vitiligo cases versus matched controls), will be used to provide overall hazard ratios (HRs) as summary estimates for the association of the presence of vitiligo with the time to skin cancer. Models will subsequently be adjusted for baseline sociodemographic, history of immunotherapy use or phototherapy treatment, prior vitiligo disease duration, and comorbidities (hypertension, hyperlipidaemia, type 2 diabetes, atrial fibrillation, angina, myocardial infarction, stroke, heart failure, chronic kidney disease stages 3-5, chronic obstructive pulmonary disease, asthma, chronic liver disease, and dementia) in multivariable analysis.

This primary endpoint analysis will be repeated in sociodemographic subgroups defined by age, sex, SES and ethnicity.

### **6.3 Secondary Objective Analysis**

Prevalence of skin cancer and each individual cancer type (melanoma, SCC, BCC and AK) will be examined in incident vitiligo cases (refer to section 3.4) and compared to matched controls without vitiligo. Prevalence will be estimated at the index date for both cases and matched controls.

Risk of new onset as described in the primary endpoint analysis will be repeated for each individual cancer type (melanoma, SCC, BCC and AK).

# **6.4 Sensitivity analysis**

To evaluate the magnitude of potential bias from including, as matched controls, people who are registered with GP practices but who do not attend their practice, we also repeated the primary analysis including only controls with a least one primary care consultation in the year preceding their index date.

As part of developing the vitiligo case definition we will explore the numbers of people excluded by each alternative diagnosis. If an alternative diagnosis is found to be common and lead to exclusion of a large proportion of the potential cohort (e.g. >10%) then

sensitivity analysis will be performed to identify any effect of removing that particular exclusion criteria on: 1) the study cohort demographics and 2) any associations with the outcome measures. These analyses may lead to an updated case definition which will be reported in full in the final project manuscript.

### 6.5 Missing data

This study will use the missing indicator variable method as missing data are considered likely not to be missing at random, meaning multiple imputation approaches will lack validity.

Patient will need to be excluded from analyses based on a matched design if they have incomplete data in the fields (age, sex) required to run the matching process. In similar studies, the exclusion rate due to incomplete data has been low (15, 16).

# 7 Study Limitations

Although the data is derived from a validated and nationally representative sample of the UK, results should not be extrapolated to dissimilar populations. Important limitations of the study include the reliance on comprehensive code lists to identify any given baseline or outcome variable. This limitation is common to all studies using routinely recorded data and will be mitigated through the use of a validated approach for defining baseline and outcome parameters. (17)

Limitations exist in the amount of clinical detail presently recorded in routine primary care electronic health records. Routine primary care databases offer the benefit of large cohorts at the expense of granularity; a limitation that is universal in epidemiological studies of this type. Some analyses will be restricted to people in whom complete information is available which may introduce selection bias as a result. Finally, the data presented will be observational in nature and although attempts will be made to reduce confounding by statistical adjustment where relevant, it is not possible to exclude the possibility of residual confounding as part of the explanation for any findings.

### 8 Statistical software

All statistical analyses will be performed using R software version 3.4.1.

### 9 Ethics

This study requires approval by the Anonymised Data Ethics Protocols and Transparency (ADEPT) Committee. It has been uploaded to ClinicalTrials.gov.

This study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value, and rigor and follow generally accepted research practices described in Guidelines for Good Pharmacoepidemiology Practices (GPP) issued by the International Society for Pharmacoepidemiology (ISPE), and Good Epidemiological Practice (GEP) guidelines issued by the International Epidemiological Association (IEA). Study reporting will be conducted in accordance with the RECORD (Reporting of studies conducted using observational routinely collected data) guidelines.(18)

### References

- 1. Steiner D, Bedin V, Moraes MB, Villas RT, Steiner T. Vitiligo. Anais Brasileiros de Dermatologia. 2004;79:335-51.
- 2. Ongenae K, Van Geel N, Naeyaert JM. Evidence for an autoimmune pathogenesis of vitiligo. Pigment Cell Res. 2003;16(2):90-100.
- 3. Bishop DT, Demenais F, Iles MM, Harland M, Taylor JC, Corda E, et al. Genome-wide association study identifies three loci associated with melanoma risk. Nat Genet. 2009;41(8):920-5.
- 4. Liu JB, Li M, Chen H, Zhong SQ, Yang S, Du WD, et al. Association of vitiligo with HLA-A2: a meta-analysis. J Eur Acad Dermatol Venereol. 2007;21(2):205-13.
- 5. Rodrigues M. Skin Cancer Risk (Nonmelanoma Skin Cancers/Melanoma) in Vitiligo Patients. Dermatologic Clinics. 2017;35(2):129-34.
- 6. Hexsel CL, Eide MJ, Johnson CC, Krajenta R, Jacobsen G, Hamzavi I, et al. Incidence of nonmelanoma skin cancer in a cohort of patients with vitiligo. Journal of the American Academy of Dermatology. 2009;60(6):929-33.
- 7. Kim HS, Kim HJ, Hong ES, Kim KB, Lee JD, Kang TU, et al. The incidence and survival of melanoma and nonmelanoma skin cancer in patients with vitiligo: a nationwide population-based matched cohort study in Korea. British Journal of Dermatology.n/a(n/a).
- 8. Teulings HE, Overkamp M, Ceylan E, Nieuweboer-Krobotova L, Bos JD, Nijsten T, et al. Decreased risk of melanoma and nonmelanoma skin cancer in patients with vitiligo: a survey among 1307 patients and their partners. Br J Dermatol. 2013;168(1):162-71.
- 9. Paradisi A, Tabolli S, Didona B, Sobrino L, Russo N, Abeni D. Markedly reduced incidence of melanoma and nonmelanoma skin cancer in a nonconcurrent cohort of 10,040 patients with vitiligo. J Am Acad Dermatol. 2014;71(6):1110-6.
- 10. OPCRD. OPCRD The Optimum Patient Care Research Database 2016 [Available from: <a href="http://optimumpatientcare.org/opcrd/">http://optimumpatientcare.org/opcrd/</a>.
- 11. Department for Communities and Local Government. The English Indices of Deprivation. 2015.2015. Available from: <a href="https://www.gov.uk/government/statistics/english-indices-of-deprivation-2015">https://www.gov.uk/government/statistics/english-indices-of-deprivation-2015</a>.
- 12. Office for National Statistics. Ethnicity2018 2nd January 2020. Available from: <a href="https://www.ons.gov.uk/peoplepopulationandcommunity/culturalidentity/ethnicity">https://www.ons.gov.uk/peoplepopulationandcommunity/culturalidentity/ethnicity</a>.
- 13. Tippu Z, Correa A, Liyanage H, Burleigh D, McGovern A, Van Vlymen J, et al. Ethnicity Recording in Primary Care Computerised Medical Record Systems: An Ontological Approach. J Innov Health Inform. 2017;23(4):920.
- 14. Memon A, Bannister P, Rogers I, Sundin J, Al-Ayadhy B, James PW, et al. Changing epidemiology and age-specific incidence of cutaneous malignant melanoma in England: An analysis of the national cancer registration data by age, gender and anatomical site, 1981–2018. The Lancet Regional Health Europe. 2021;2.
- 15. Kumar S, de Lusignan S, McGovern A, Correa A, Hriskova M, Gatenby P, et al. Ischaemic stroke, haemorrhage, and mortality in older patients with chronic kidney disease newly started on anticoagulation for atrial fibrillation: a population based study from UK primary care. Bmj. 2018;360:k342.
- 16. Rayner LH, Mcgovern A, Sherlock J, Gatenby P, Correa A, Creagh-Brown B, et al. The impact of therapy on the risk of asthma in type 2 diabetes. Clin Respir J. 2019;13(5):299-305.
- 17. de Lusignan S, Liaw ST, Michalakidis G, Jones S. Defining datasets and creating data dictionaries for quality improvement and research in chronic disease using routinely collected data: an ontology-driven approach. Informatics in primary care. 2011;19(3):127-34.

18. Benchimol EI, Smeeth L, Guttmann A, Harron K, Moher D, Petersen I, et al. The REporting of studies Conducted using Observational Routinely-collected health Data (RECORD) statement. PLoS Med. 2015;12(10):e1001885.

Codes to be used to identify cases of vitiligo and important exclusion conditions (see also Appendix 2).

Read and SNOMED codes to be used to identify cases of vitiligo

| | Term | |
|---|---|---|
| Read V2 Code | ID | Description |
| M2951 | All | Vitiligo |
| M293. | All | Hypopigmentation disorder |
| F4E53 | All | Vitiligo of eyelid |
| M295. | All | Leucoderma |
| M295z | All | Leucoderma NOS |
| | Term | |
| Read CTV3 Code | ID | Description |
| M2951 | All | Vitiligo |
| M293. | All | Hypopigmentation disorder |
| F4E53 | All | Vitiligo of eyelid |
| M295. | All | Acquired hypomelanosis |
| M295z | All | Leucoderma NOS |
| | Term | |
| SNOMED Code | ID | Description |
| 56727007 | | Vitiligo (disorder) |
| 87666009 | | Vitiligo of eyelid (disorder) |
| 721539008 | | Vitiligo of eyelid and periocular area (disorder) |
| 403271008 | | Kobner vitiligo (disorder) |
| 403270009 | | Trichrome vitiligo (disorder) |
| 403267005 | | Localised vitiligo (disorder) |
| 403268000 | | Segmental vitiligo (disorder) |
| 402621008 | | Idiopathic vitiligo (disorder) |
| 403269008 | | Generalised vitiligo (disorder) |
| 33093100011910 | | |
| 6 | | Vitiligo of skin of left eyelid and periocular area (disorder) |
| 33093100011910 | | |
| 4 | | Vitiligo of skin of right eyelid and periocular area (disorder) |
| 33091100011910 | | Vitiligo of skin of left upper eyelid and periocular area |
| 1 | | (disorder) |
| 33088100011910 | | Vitiligo of skin of right upper eyelid and periocular area |
| 1 | | (disorder) |
| 726608002 | | Spastic paraparesis, vitiligo, premature greying, |
| 22005000 | | characteristic facies syndrome |
| 23006000 | | Hypopigmentation of skin (disorder) |
| 89031001 | | Hypopigmentation (morphological abnormality) |
| 68210006 | | Hypopigmentation of eyelid |

| 18655006 | Dipigmentation |
|-----------|----------------------------------------|
| 23267004 | Achromia of skin (disorder) |
| 402807009 | Circumscribed hypomelanosis (disorder) |

Read codes and SNOMED codes to be used to identify alternative depigmenting disorders for exclusion

| Congenital and Genetic Hypomelanoses | | |
|---|---|---|
| | Term | |
| Read V2 Code | ID | Description |
| C302A | All | Piebaldism |
| PK5 | All | Tuberous sclerosis |
| PKy54 | All | Waardenburg's syndrome |
| C3029 | All | Hermansky-Pudlak |
| PKy92 | All | Menke's syndrome |
| | Term | |
| Read CTV3 Code | ID | Description |
| X78Ve | All | Hypomelanosis of Ito |
| XaZqX | All | Piebaldism |
| PK5 | All | Tuberous sclerosis |
| X78E7 | All | Ash leaf spot, tuberous sclerosis |
| X78E8 | All | Shargreen patch |
| X78E9 | All | Adenoma sebaceum |
| X20Ex | All | Hermansky-Pudlak syndrome |
| X20ij | All | Griscelli syndrome with immunodeficiency |
| PKy92 | All | Menkes syndrome |
| | Term | |
| SNOMED Code | ID | Description |
| 218358001 | | Incontinentia pigmenti achromians syndrome (disorder) |
| 718122005 | | Piebaldism (disorder) |
| 7199000 | | Tuberous sclerosus syndrome (disorder) |
| 254243001 | | Ash leaf spot, tuberous sclerosis (disorder) |
| 36025004 | | Fibrous skin tumor of tuberous sclerosis (disorder) |
| 254244007 | | Shagreen patch (disorder) |
| 9311003 | | Hermansky-Pudlak syndrome (disorder) |
| 37548006 | | Hypopigmentation-immunodeficiency disease (disorder) |
| 59178007 | | Menkes kinky-hair syndrome (disorder) |
| 47434006 | | Waardenburg's syndrome (disorder) |
| 715052000 | | Waardenburg syndrome co-occurrent with Hirschsprung |
| 715952000 | | disease (disorder) |
| 773575001 | | Ocular albinism with congenital sensorineural deafness (disorder) |

| 765325002 | | Peripheral demyelinating neuropathy, central dysmyelinating leukodystrophy, Waardenburg syndrome, Hirschsprung disease (disorder) |
|---|---|---|
| Post-inflammatory | Hypomela | noses |
| Read V2 Code | Term<br>ID | Description |
| M2920 | All | Post inflammatory hypopigmentation |
| M170. | All | Lichen planus |
| M1700 | All | Lichen planus actinicus |
| M1701 | All | Lichen planus annularis |
| M1702 | All | Lichen planus atrophicus |
| M1703 | All | Lichen planus bullosus |
| M1704 | All | Lichen planus hypertrophicus |
| M1705 | All | Lichen planus linearis |
| M1707 | All | Lichen planus obtusus |
| M1708 | All | Subacute active lichen planus |
| M1709 | All | Follicular lichen planus |
| M170z | All | Lichen planus NOS |
| M17y0 | All | Lichen ruber moniliforme |
| M1650 | All | Pityriasis alba |
| M2102 | All | Lichen sclerosus and atrophicus |
| K276. | All | Balanitis xerotica obliterans |
| Read CTV3 Code | Term<br>ID | Description |
| Xa0WM | All | Post inflammatory hypopigmentation |
| M170. | All | Lichen planus |
| X507Y | All | Confluent lichen planus |
| X507Z | All | Micropaplular lichen planus |
| X507a | All | Guttate lichen planus |
| X507b | All | Follicular lichen planus |
| M1703 | All | Bullous lichen planus |
| M1701 | All | Annular lichen planus |
| M1704 | All | Hypertrophic lichen planus |

| M1702 | All | Atrophic lichen planus |
|-------|-----|------------------------------------------------------|
| M1705 | All | Linear lichen planus |
| X507c | All | Zosteriform lichen planus |
| M1700 | All | Acintic lichen planus |
| X507d | All | Post inflammatory hyperpigmentation in lichen planus |
| X507e | All | Wickham's striae in lichen planus |
| X507f | All | Lichen planus - lupus erythematosus overlap |
| X507g | All | Lichen planus pemphigoides |
| X507h | All | Site-specific lichen planus |
| X507i | All | Lichen planus of scalp |
| X507j | All | Lichen planus of palms and soles |
| X507k | All | Ulcerative lichen planus of palms and soles |
| X507n | All | Mutilating lichen planus of fingers and toes |
| X507l | All | Lichen planus of nail |
| X507w | All | Genital lichen planus |
| X408F | All | Lichen planus of vuvla |
| X507y | All | Erosive lichen planus of vulva |
| X507z | All | Lichen planus of penis |
| X5080 | All | Lichen planus of glans penis |
| M1707 | All | Lichen planus obtusus |
| M1708 | All | Subacute active lichen planus |
| M170z | All | Lichen planus NOS |
| Myu32 | All | [X]Other lichen planus |
| M17y0 | All | Lichen ruber moniliforme |
| M1650 | All | Pityriasis alba |
| M2102 | All | Lichen sclerosus |
| X50FC | All | Genital lichen sclerosus |
| K276. | All | Balanitis xerotica obliterans |
| X50FE | All | Lichen sclerosus of vulva |
| X50FF | All | Extra genital lichen sclerosus |
| X50FG | All | Guttate lichen sclerosus |

| SNOMED Code | Term<br>ID | Description |
|---|---|---|
| 277787003 | | Post-inflammatory hypopigmentation (disorder) |
| 403272001 | | Post-infective hypomelanosis (disorder) |
| 403276003 | | Acquired hypomelanosis of uncertain etiology (disorder) |
| 4776004 | | Lichen planus (disorder) |
| 263797007 | | Lichen planus-like (qualifier value) |
| 4459000 | | Linear lichen planus (disorder) |
| 6111009 | | Bullous lichen planus (disorder) |
| 238666005 | | Lichen planus of lips (disorder) |
| 201001005 | | Lichen planus obtusus (disorder) |
| 200999007 | | Actinic lichen planus (disorder) |
| 238658001 | | Lichen planus of nail (disorder) |
| 238668006 | | Genital lichen planus (disorder) |
| 201000006 | | Annular lichen planus (disorder) |
| 238647005 | | Guttate lichen planus (disorder) |
| 237112004 | | Lichen planus of vulva (disorder) |
| 400108007 | | Flexural lichen planus (disorder) |
| 238655003 | | Lichen planus of scalp (disorder) |
| 44509000 | | Linear lichen planus (disorder) |
| 25858008 | | Atrophic lichen planus (disorder) |
| 238670002 | | Lichen planus of penis (disorder) |
| 238645002 | | Confluent lichen planus (disorder) |
| 717061002 | | Lichen planus pigmentosus (disorder) |
| 238648000 | | Zosteriform lichen planus (disorder) |
| 238653005 | | Lichen planus pemphigoides (disorder) |
| 68266006 | | Hypertrophic lichen planus (disorder) |
| 238646001 | | Micropapular lichen planus (disorder) |
| 64540004 | | Lichen planopilaris (disorder) |
| 238654004 | | Site-specific lichen planus (disorder) |
| 238652000 | | Lichen planus-lupus erythematosus overlap (disorder) |
| 403198004 | | Lichenoid actinic keratosis (disorder) |
| 723003004 | | Acute eruptive lichen planus (disorder) |
| 238671003 | | Lichen planus of glans penis (disorder) |
| 68266006 | | Hypertrophic lichen planus (disorder) |
| 201002003 | | Subacute active lichen planus (disorder) |
| 720493003 | | Annular atrophic lichen planus (disorder) |
| 120493003 | | Annual acrophic lichen planus (disorder) |

| 238651007 | | Wickham's striae in lichen planus (disorder) |
|---|---|---|
| 201001005 | | Lichen planus obtusus (disorder) |
| 402349005 | | Chronic lichen planus (disorder) |
| 238668006 | | Genital lichen planus (disorder) |
| 238656002 | | Lichen planus of palms and soles (disorder) |
| 402352002 | | Poikiloderma due to lichen planus (disorder) |
| 721171007 | | Hypertrophic lichen planus of vulva (disorder) |
| 402348002 | | Köbner reaction from lichen planus (disorder) |
| 238657006 | | Ulcerative lichen planus of palms and soles (disorder) |
| 238660004 | | Mutilating lichen planus of fingers and toes (disorder) |
| 726476005 | | Lichen planus co-occurrent with onycholysis (disorder) |
| | | Post-inflammatory hyperpigmentation in lichen planus |
| 238649008 | | (disorder) |
| 402296004 | | Pityriasis alba (disorder) |
| 402298003 | | Diffuse pityriasis alba (disorder) |
| 402297008 | | Localised pityriasis alba (disorder) |
| 25674000 | | Lichen sclerosus et atrophicus (disorder) |
| 402423004 | | Adult lichen sclerosus (disorder) |
| 782666006 | | Lichen sclerosus of anus (disorder) |
| 238934003 | | Guttate lichen sclerosus (disorder) |
| 238932004 | | Genital lichen sclerosus (disorder) |
| 700082001 | | Lichen sclerosus of penis (disorder) |
| 26348009 | | Lichen sclerosus et atrophicus of the vulva (disorder) |
| 402424005 | | Childhood lichen sclerosus (disorder) |
| 403566002 | | Anogenital lichen sclerosus (disorder) |
| 238933009 | | Extragenital lichen sclerosus (disorder) |
| 402714001 | | Lichen sclerosus of male genitalia (disorder) |
| 402715000 | | Lichen sclerosus of female genitalia (disorder) |
| 402422009 | | Bullous extragenital lichen sclerosus (disorder) |
| 721199003 | | Prepubertal lichen sclerosus of vulva (disorder) |
| 403568001 | | Localized extragenital lichen sclerosus (disorder) |
| 402421002 | | Generalized extragenital lichen sclerosus (disorder) |
| 403564004 | | Lichen sclerosus of penis, childhood form (disorder) |
| 111023000 | | Lichen sclerosus et atrophicus, bullous type (disorder) |
| 403565003 | | Vulval lichen sclerosus, childhood form (disorder) |
| 198033005 | | Balanitis xerotica obliterans (disorder) |
| Post Traumatic Leul | koderma | |
| | Term | |
| SNOMED Code | ID | Description |
| 402622001 | | Hypomelanosis due to scarring (disorder) |
| 18655006 | | Depigmentation (morphologic abnormality) |
| 23006000 | | Hypopigmentation of skin (disorder) |
| 398656003 | | Acquired hypomelanotic disorder (disorder) |
| Para-Malignant Hypomelanoses | | |

| Term | |
|------|-------------------------------------------------------------|
| ID | Description |
| All | Mycosis fungoides |
| All | Mycosis fungoides of unspecified site |
| All | Mycosis fungoides of lymph nodes of head, face and neck |
| All | Mycosis fungoides of intrathoracic lymph nodes |
| All | Mycosis fungoides of intra-abdominal lymph nodes |
| All | Mycosis fungoides of lymph nodes of axilla and upper limb |
| All | Mycosis fungoides of lymph nodes of inguinal region and leg |
| All | Mycosis fungoides of intrapelvic lymph nodes |
| All | Mycosis fungoides of spleen |
| All | Mycosis fungoides of lymph nodes of multiple sites |
| All | Mycosis fungoides NOS |
| All | [M]Mycosis fungoides |
| All | [M]Mycosis fungoides |
| All | [M]Sezary's disease |
| All | [M]Mycosis fungoides NOS |
| All | Oth and unspecif peripheral & cutaneous T-cell lymphomas |
| All | Subcutaneous panniculitis like T-cell lymphoma |
| All | [M]Cutaneous lymphoma |
| All | Sezary's disease |
| All | Sezary's disease of unspecified site |
| All | Sezary's disease of lymph nodes of head, face and neck |
| All | Sezary's disease of intrathoracic lymph nodes |
| All | Sezary's disease of intra-abdominal lymph nodes |
| All | Sezary's disease of lymph nodes of axilla and upper limb |
| All | Sezary's disease of lymph nodes of inguinal region and leg |
| All | Sezary's disease of intrapelvic lymph nodes |
| All | Sezary's disease of spleen |
| All | Sezary's disease of lymph nodes of multiple sites |
| All | Sezary's disease NOS |
| All | Amelanotic melanoma |
| Term | |
| ID | Description |
| All | Mycosis fungoides |
| All | Poikiloderma vasculare atrophicans |
| All | Mycosis fungoides of skin |
| All | Mycosis fungoides of unspecified site |
| All | Mycosis fungoides of lymph nodes of head, face and neck |
| All | Mycosis fungoides of intrathoracic lymph nodes |
| All | Mycosis fungoides of intra-abdominal lymph nodes |
| | Mycosis fungoides of lymph nodes of axilla and upper limb |
| | Mycosis fungoides of lymph nodes of inguinal region and leg |
| All | Mycosis fungoides of intrapelvic lymph nodes |
| | All |

| | · |
|---|---|
| All | Mycosis fungoides of lymph nodes of multiple sites |
| All | Mycosis fungoides NOS |
| All | Sezary's disease |
| All | Sezary's disease of unspecified site |
| All | Sezary's disease of lymph nodes of head, face and neck |
| All | Sezary's disease of intrathoracic lymph nodes |
| All | Sezary's disease of intra-abdominal lymph nodes |
| All | Sezary's disease of lymph nodes of axilla and upper limb |
| All | Sezary's disease of lymph nodes of inguinal region and leg |
| All | Sezary's disease of intrapelvic lymph nodes |
| All | Sezary's disease of spleen |
| All | Sezary's disease of lymph nodes of multiple sites |
| All | Sezary's disease NOS |
| All | Sezary's disease of skin |
| All | Cutaneous lymphoma |
| All | Cutaneous follicle centre lymphoma |
| All | Cutaneous/peripheral T-cell lymphoma |
| All | Subcutaneous panniculitis like T-cell lymphoma |
| | [X]0th and unspecif peripheral & cutaneous T-cell |
| All | lymphomas |
| | Primary cutaneous CD30 antigen positive large T-cell |
| All | lymphoma |
| All | Amelanotic malignant melanoma of skin |
| Term | |
| ID | Description |
| | Mycosis fungoides (morphologic abnormality) |
| | Mycosis fungoides (disorder) |
| | , , , , , |
| | Classic mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) Folliculotropic mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) Folliculotropic mycosis fungoides (disorder) |
| | Classic mycosis fungoides (disorder) Bullous mycosis fungoides (disorder) Mycosis fungoides of spleen (disorder) Spongiotic mycosis fungoides (disorder) History of mycosis fungoides (situation) Follicular mycosis fungoides (morphologic abnormality) Tumour stage mycosis fungoides (disorder) Syrngotropic mycosis fungoides (disorder) Granulomatous mycosis fungoides (disorder) Erythrodermic mycosis fungoides (disorder) Hypomelanocytic mycosis fungoides (disorder) Folliculotropic mycosis fungoides (disorder) Pokilodermatous mycosis fungoides (disorder) |
| | All |

| | Mycosis fungoides of intra-abdominal lymph nodes |
|---|---|
| 94707004 | (disorder) |
| 34707004 | Mycosis fungoides of lymph nodes of multiple sites |
| 188627002 | (disorder) |
| 100027002 | Lymphomatoid papulosis-associated mycosis fungoides |
| 404111002 | (disorder) |
| 10 122302 | Lymphomatoid papulosis type B mycosis fungoides-like |
| 404104001 | (disorder) |
| | Mycosis fungoides of extranodal AND/OR solid organ site |
| 94715001 | (disorder) |
| 94709001 | Mycosis fungoides of intrathoracic lymph nodes (disorder) |
| 5 W 00002 | Mycosis fungoides of lymph nodes of head, face AND/OR |
| 94711005 | neck (disorder) |
| | Mycosis fungoides of lymph nodes of axilla AND/OR upper |
| 94710006 | limb (disorder) |
| | Mycosis fungoides of lymph nodes of multiple sites |
| 188627002 | (disorder) |
| | Mycosis fungoides of lymph nodes of inguinal region |
| 94712003 | AND/OR lower limb (disorder) |
| | Cutaneous T-cell lymphoma, no International Classifcation |
| | of Diseases for oncology subtype (morphologic |
| 28054005 | abnormality) |
| 40012207 | Primary cutaneous T-cell lymphoma (disorder) |
| 277613000 | Cutaneous/peripheral T-cell lymphoma (disorder) |
| 404128004 | CD-30 negative cutanoeus T-cell lymphoma (disorder) |
| | Primary cutaneous T-cell lymphoma - category |
| 419283005 | (morphologic abnormality) |
| | Primary cutaneous CD30 antigen positive T-cell |
| 128804002 | lymphoproliferative disorder (morphologic abnormality) |
| | Primary cutaneous gamma-delta T-cell lymphoma |
| 450908002 | (morphologic abnormality) |
| 12257100011910 | |
| 6 | History of primary cutaneous T-cell lymphoma (situation) |
| | Primary cutaneous large T-cell lymphoma - category |
| 419018000 | (morphologic abnormality) |
| 402880009 | Primary cutaneous large T-cell lymphoma (disorder) |
| | Subcutaneous panniculitic cutaneous T-cell lymphoma |
| 404133000 | (disorder) |
| 404128004 | CD-30 negative cutaneous T-cell lymphoma (disorder) |
| | Primary cutaneous acral CD8 positive T-cell lymphoma |
| 787198005 | (morphologic abnormality) |
| | Primary cutaneous anaplastic large T-cell lymphoma, CD30 |
| 397352006 | positive (morphologic abnormality) |
| | Primary cutaneous gamma-delta-positive T-cell lymphoma |
| 733627006 | (disorder) |

| | CD-30 negative anaplastic large T-cell cutaneous lymphoma |
|---|---|
| 404129007 | (disorder) |
| 12257100011910 | (a.soruc.) |
| 6 | History of malignant cutaneous T-cell lymphoma (situation) |
| | CD-30 negative pleomorphic large T-cell cutaneous |
| 404130002 | lymphoma (disorder) |
| | CD-30 positive pleomorphic large T-cell cutaneous |
| 404126000 | lymphoma (disorder) |
| | Primary cutaneous T-cell lymphoma - category |
| 419283005 | (morphologic abnormality) |
| | Primary cutaneous gamma-delta T-cell lymphoma - category |
| 450908002 | (morphologic abnormality) |
| | Primary cutaneous CD8 positive aggressicve epidermotropic |
| 765136002 | cytotoxic T-cell lymphoma (disorder) |
| | Primary cutaneous CD30 antigen positive large T-cell |
| 128875000 | lymphoma (disorder) |
| | Primary cutaneous CD8 positive aggressicve epidermotropic |
| 733895005 | cytotoxic T-cell lymphoma (morphologic abnormality) |
| | Primary cutaneous T-cell lymphoma, large cell, CD30- |
| 419586003 | negative (morphological abnormality) |
| 118611004 | Sezary's disease (disorder) |
| 4950009 | Sezary's disease (morphologic abnormality) |
| 255101006 | Sezary disease of skin (disorder) |
| 95263006 | Sezary's disase of spleen (disorder) |
| 188632001 | Sezary's disase of intra-abdominal lymph nodes (disorder) |
| 188635004 | Sezary's disase of intrapelvic lymph nodes (disorder) |
| 188631008 | Sezary's disase of intrathoracic lymph nodes (disorder) |
| 188637007 | Sezary disease of lymph nodes of multiple sites (disorder) |
| | Sézary's disease of extranodal AND/OR solid organ site |
| 95264000 | (disorder) |
| | Sézary's disease of lymph nodes of axilla and upper limb |
| 188633006 | (disorder) |
| 0500000 | Sézary's disease of lymph nodes of head, face AND/OR neck |
| 95260009 | (disorder) |
| 100624000 | Sézary's disease of lymph nodes of inguinal region and |
| 188634000 | lower limb (disorder) |
| 95261008 | Sézary's disease of lymph nodes of inguinal region AND/OR |
| 419392005 | lower limb (disorder) Primary cutaneous lymphoma (morphologic abnormality) |
| 719392003 | Tumour and germline whole genome sequencing for |
| | anaplastic lymphoma kinase negative anaplastic large cell |
| | lymphoma including primary cutaneous subtypes |
| 82321000000106 | (procedure) |
| | Hypomelanosis surrounding malignant melanoma |
| 403274000 | (disorder) |
| | (************************************** |

| | | Metastatic malignant melanoma with diffuse |
|---|---|---|
| 402563000 | | hypermelanosis (disorder) |
| 276751004 | | Amelanotic malignant melanoma of skin (disorder) |
| 70594002 | | Amelanotic melanoma (morphologic abnormality) |
| 404110001 | | Hypomelanotic mycosis fungoides (disorder) |
| | | Hypomelanosis surrounding melanocytic neoplasm |
| 402623006 | | (disorder) |
| Occupational/drug | induced h | ypomelanoses |
| | Term | |
| Read V2 Code | ID | Description |
| M293. | All | Hypopigmentation |
| | Term | |
| Read CTV3 Code | ID | Description |
| X508z | All | Occupational vitiligo |
| X78VE | All | Chemically-induced hypomelanosis |
| X50Gx | All | Drug-induced hypomelanosis |
| Xa1aV | All | Chemically-induced hypomelanosis |
| M2950 | All | Leucoderma aestivale |
| M295. | All | Acquired hypomelanosis |
| CNOMED Codo | Term | |
| SNOMED Code | ID | Description Occupational vitiliza (disorder) |
| 238713002<br>280962005 | | Occupational vitiligo (disorder) |
| 402622001 | | Chemically-induced hypomelanosis (disorder) |
| 403807001 | | Hypomelanosis due to scarring (disorder) |
| 398656003 | | Phylloid hypomelanosis (disorder) |
| 238999005 | | Acquired hypomelanotic disorder (disorder) |
| 403698000 | | Drug-induced hypomelanosis (disorder) Laser-induced hypopigmentation (disorder) |
| 402622001 | | Hypomelanosis due to scarring (disorder) |
| 280962005 | | Chemically-induced hypomelanosis (disorder) |
| 403692004 | | |
| 403744007 | | Hypomelanosis due to cryotherapy (disorder) |
| 403698000 | | Arsenic-induced "rain-drop" hypomelanosis (disorder) Laser-induced hypopigmentation (disorder) |
| 201290009 | | Leukoderma estivale (disorder) |
| _01230003 | | |
| Para-infectious hyp | opigment | ation |
| Tura iliterativa | Term | |
| Read V2 Code | ID | Description |
| AB10. | All | Pityriasis versicolor |
| | Term | |
| Read CTV3 Code | ID | Description |
| AB10. | All | Pityriasis versicolor |
| | | ., |

| | Term | |
|--------------------|------|---------------------------------------------|
| <b>SNOMED Code</b> | ID | Description |
| 56454009 | | Pityriasis versicolor (disorder) |
| 18097004 | | Malassezia (organism) |
| 721794002 | | Infection caused by Malassezia (disorder) |
| 402133004 | | Malassezia infection of the skin (disorder) |
| 29619007 | | Malassezia furfur (organism) |

Others (including Melasma, Morphoea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, Progressive macular hypomelanosis, Nevus depigmentosus, Cutaneous sarcoidosis)

| 3arcoldosis) | Term | |
|----------------|------|---------------------------------------|
| Read V2 Code | ID | Description |
| M290. | All | <b>Description</b> Melasma |
| M2900 | All | |
| | | Chloasma bronzinum |
| M2901 | All | Chloasma cachecticorum |
| M2902 | All | Chloasma caloricum |
| M2903 | All | Chloasma gravidarum |
| M2903 | All | Chloasma gravidarum |
| M2903 | All | Chloasma gravidarum |
| M290z | All | Chloasma NOS |
| M2103 | All | Morphoea |
| M2104 | All | Linear Morphoea |
| M210. | All | Circumscribed scleroderma |
| M2100 | All | Unspecified circumscribed scleroderma |
| M2101 | All | Localised dermatosclerosis |
| M210z | All | Circumscribed scleroderma NOS |
| PH322 | All | Xeroderma pigmentosum |
| BBE9. | All | [M]Nonpigmented naevus |
| AD530 | All | Lupus Pernio |
| AD53. | All | Sarcoidosis of skin |
| | Term | |
| Read CTV3 Code | ID | Description |
| M290. | All | Melasma |
| Xa1aM | All | Drug-induced melasma |
| M2900 | All | Chloasma bronzinum |
| M2901 | All | Chloasma cachecticorum |
| M2902 | All | Chloasma caloricum |
| M2904 | All | Chloasma hepaticum |
| M2905 | All | Chloasma toxicum |
| M2906 | All | Chloasma traumaticum |
| M290z | All | Chloasma NOS |
| M2903 | All | Melasma of pregnancy |
| Xa1aM | All | Drug-induced melasma |
| | • | |

| M2102 | AII | Marrahaaa |
|-------------|------|-----------------------------------------|
| M2103 | All | Morphoea |
| X7053 | | Generalised morphoea |
| M2101 | All | Localised morphoea |
| M2100 | All | Unspecified circumscribed scleroderma |
| M210z | All | Circumscribed scleroderma NOS |
| X7055 | All | Linear morphoea |
| PH322 | All | Xeroderma pigmentosum |
| X78Cz | All | Xeroderma pigmentosum group A |
| X78D0 | All | Xeroderma pigmentosum group B |
| X78D1 | All | Xeroderma pigmentosum group C |
| X78D2 | All | Xeroderma pigmentosum group D |
| X78D3 | All | Xeroderma pigmentosum group E |
| X78D4 | All | Xeroderma pigmentosum group F |
| X78D5 | All | Xeroderma pigmentosum group G |
| X78D6 | All | Xeroderma pigmentosum XP variant |
| X78D7 | All | De Sanctis-Cacchione syndrome |
| X78D8 | All | Xerodermoid, pigmented |
| X50lw | All | Symmetrical progressive leucopathy |
| X20GW | All | Cutaneous sarcoid |
| X20GX | All | Orofacial sarcoid |
| X20GY | All | Lupus pernio |
| X5089 | All | Acute skin sarcoidosis |
| X508A | All | Sarcoidosis-induced erythema nodosum |
| X508B | All | Lofgrens syndrome |
| X508C | All | Maculopapular sarcoidosis |
| X508D | All | Chronic skin sarcoidosis |
| X508E | All | Sarcoidosis in scar |
| X508F | All | Papular sarcoidosis |
| X508G | All | Lichenoid sarcoidosis |
| X508H | All | Nodular sarcoidosis |
| X508I | All | Angiolupoid sarcoidosis |
| X00YQ | All | Sarcoid skin of eyelid |
| X20G5 | All | Sarcoid dactylitis |
| X50Dy | All | Subacute nodular migratory panniculitis |
| X50Dz | All | Subcutaneous lipogranulomatosis |
| | Term | |
| SNOMED Code | ID | Description |
| 36209000 | | Melasma |
| 201274009 | | Chloasma bronzinum (disorder) |
| 201275005 | | Chloasma cachecticorum (disorder) |
| 201276006 | | Chloasma caloricum (disorder) |
| 201277002 | | Chloasma hepaticum (disorder) |
| 201278007 | | |
| 2012/600/ | | Chloasma toxicum (disorder) |

| 79840007 | Idiopathic chloasma (disorder) |
|------------|--------------------------------------------------------------|
| 111208003 | Melasma gravidarum (disorder) |
| 54397000 | Symptomatic chloasma (disorder) |
| 201279004 | Chloasma traumaticum (disorder) |
| 201049004 | Morphea (disorder) |
| 128458002 | Plaque morphea (disorder) |
| 22784002 | Linear scleroderma (disorder) |
| 403521006 | Guttate morphea (disorder) |
| 201048007 | Localised morphea (disorder) |
| 7513007 | Generalized morphea (disorder) |
| 403522004 | Subcutaneous morphea (disorder) |
| 51156002 | Coup de sabre scleroderma (disorder) |
| 403523009 | Disabling pansclerotic morphea of children (disorder) |
| 128460000 | Diffuse cutaneous scleroderma (disorder) |
| 403524003 | Scleroderma-like secondary cutaneous sclerosis (disorder) |
| 1717003 | Idiopathic guttate hypomelanosis (disorder) |
| | Guttate hypopigmentation and punctate palmoplantar |
| 711154007 | keratoderma with or without ectopic calcification (disorder) |
| 44600005 | Xeroderma pigmentosum (disorder) |
| 56048001 | Xeroderma pigmentosum, group E (disorder) |
| 25784009 | Xeroderma pigmentosum, group C (disorder) |
| 36454001 | Xeroderma pigmentosum, group G (disorder) |
| 1073003 | Xeroderma pigmentosum, group B (disorder) |
| 68637004 | Xeroderma pigmentosum, group D (disorder) |
| 42530008 | Xeroderma pigmentosum, group F (disorder) |
| 43477006 | Xeroderma pigmentosum, group A (disorder) |
| 73663008 | Neurologic xeroderma pigmentosum (disorder) |
| 88877002 | Xeroderma pigmentosum, variant form (disorder) |
| 7806002 | Non-neurologic xeroderma pigmentosum (disorder) |
| 7 00 000 0 | Xeroderma pigmentosum and Cockayne syndrome complex |
| 719819004 | (disorder) |
| 239083007 | Symmetrical progressive leucopathy (disorder) |
| 23303307 | Familial progressive hyper and hypopigmentation of skin |
| 763368004 | (disorder) |
| 403541001 | Nevus depigmentosus |
| 112680001 | Naevus depigmentosus |
| 55941000 | Cutaneous sarcoidosis (disorder) |
| 238680003 | Papular sarcoidosis (disorder) |
| 238679001 | Sarcoidosis in scar (disorder) |
| 402369000 | Atrophic sarcoidosis (disorder) |
| 402369000 | Verrucous sarcoidosis (disorder) |
| 238681004 | Lichenoid sarcoidosis (disorder) |
| 238674006 | Acute skin sarcoidosis (disorder) |
| 402370004 | Ulcerative sarcoidosis (disorder) |
| 58870009 | Sarcoidosis, anular type (disorder) |

| 54515008 | Sarcoidosis, plaque type (disorder) |
|-----------|-------------------------------------------------|
| 80941006 | Subcutaneous sarcoidosis (disorder) |
| 870334009 | Palmoplantar sarcoidosis (disorder) |
| 238678009 | Chronic skin sarcoidosis (disorder) |
| 238677004 | Maculopapular sarcoidosis (disorder) |
| 402368008 | Ichthyosiform sarcoidosis (disorder) |
| 402373002 | Hypomelanotic sarcoidosis (disorder) |
| 9529007 | Sarcoidosis, erythrodermic type (disorder) |
| 72470008 | Sarcoidosis, lupus pernio type (disorder) |
| 402372007 | Subcutaneous nodular sarcoidosis (disorder) |
| 238675007 | Sarcoidosis-induced erythema nodosum (disorder) |
| 238676008 | Lofgrens syndrome (disorder) |
| 31541009 | Lupus pernio of Besnier |
| 231799005 | Sarcoid skin of eyelid (disorder) |

Potential differential diagnoses for vitiligo which will be used as exclusion criteria if they appear as diagnoses in the medical record within six months of the initial diagnosis of vitiligo (six months before or after the vitiligo diagnosis). \*As these conditions are extremely uncommon in the UK they will not be used in the exclusion process. Codes for these conditions are listed in Appendix 1.

| Conditions/causes included |
|-----------------------------------------------|
| Piebaldism |
| Tuberous sclerosis |
| Hypomelanosis of Ito |
| Waardenburg syndrome |
| Hermanski-Pudlak syndrome |
| Griscelli syndrome |
| Menkes syndrome |
| Post-inflammatory leukoderma including after |
| Atopic eczema or Psoriasis |
| Lichen planus |
| Pityriasis alba |
| Lichen sclerosus |
| Post traumatic leukoderma |
| Cutaneous T-cell lymphoma (mycosis fungoides) |
| Melanoma associated depigmentation |
| Occupational vitiligo |
| Other induced hypomelanoses |
| Pityriasis versicolor (or tinea versicolor) |
| Leprosy* |
| Leishmaniasis* |
| Melasma |
| Morphoea |
| Idiopathic guttate hypomelanosis |
| Xeroderma pigmentosum |
| Progressive macular hypomelanosis |
| Nevus depigmentosus |
| Cutaneous sarcoidosis |

Below is a list of the variables to be extracted and utilised for the study

| Variable | Role | Data source(s) | Operational |
|---|---|---|---|
| | | | definition |
| Vitiligo | Case definition | OPCRD | As defined using the |
| | | | codes listed in |
| | | | Appendix 1 |
| Vitiligo exclusion | Case definition | OPCRD | As defined using the |
| conditions | | | codes listed in |
| | | | Appendix 1 and |
| | | | summarised in |
| | | | Appendix 2 |
| Melanoma | Study outcome | OPCRD | Identified using a |
| | | | expert review list of |
| | | | clinical diagnosis codes |
| | | | from the primary care |
| | | | record. Clinical codes |
| | | | listed in Appendix 4. |
| Squamous cell | Study outcome | OPCRD | Identified using a |
| carcinoma (SCC) | | | expert review list of |
| | | | clinical diagnosis codes |
| | | | from the primary care |
| | | | record. Clinical codes |
| | | | listed in Appendix 4. |
| Basal cell carcinoma | Study outcome | OPCRD | Identified using a |
| (BCC) | | | expert review list of |
| | | | clinical diagnosis codes |
| | | | from the primary care |
| | | | record. Clinical codes |
| | | | listed in Appendix 4. |
| Actinic keratoses (AK) | Study outcome | OPCRD | Identified using a |
| | | | expert review list of |
| | | | clinical diagnosis codes |
| | | | from the primary care |
| | | | record. Clinical codes |
| | | | listed in Appendix 4. |
| Age | Baseline characteristic, | OPCRD | Defined as age at the |
| | predictor variable | | start of follow up |
| Gender | Baseline characteristic, | OPCRD | Primary care recorded |
| | predictor variable | | patient gender |

| SES) Predictor variable Index of multiple deprivation quintile | Socioeconomic status | Baseline characteristic, | OPCRD | Defined using patient |
|---|---|---|---|---|
| Ethnicity Baseline characteristic, predictor variable redictor variable substitution predictor variable redictor variable substitution predictor variable substitution substitu | (SES) | predictor variable | | index of multiple |
| predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Body mass index (BMI) Body m | | | | deprivation quintile |
| Smoking status Baseline characteristic, predictor variable Censoring event Death Censoring event OPCRD Deregistration from GP Censoring event OPCRD Deregistration from GP Censoring event OPCRD Deregistration from GP Censoring event OPCRD Deregistration from GP Censoring event OPCRD Deregistration from GP Censoring event OPCRD Identified from coding in the clinical record in | Ethnicity | Baseline characteristic, | OPCRD | Defined using office of |
| Smoking status Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Body mass index (BMI) Body mass index (BMI) Baseline characteristic, predictor variable Body mass index (BMI) Baseline characteristic, predictor variable Censoring event Deregistration from GP Censoring event OPCRD Deregistration from GP Censoring event OPCRD Deregistration from GP Atrial fibrillation Baseline characteristic, predictor variable Angina Baseline characteristic, predictor variable Myocardial infarction Baseline characteristic, oPCRD Identified using clinical codes for the condition Myocardial infarction Baseline characteristic, oPCRD Identified using clinical codes for the condition Myocardial infarction Baseline characteristic, oPCRD Identified using clinical codes for the condition | | predictor variable | | national statistics |
| Smoking status Baseline characteristic, predictor variable Censoring event Death Censoring event Decrop Decrop Defined using most recent clinically recorded BMI information Death Censoring event OPCRD Decrop Identified from coding in the clinical record Atrial fibrillation Baseline characteristic, predictor variable Angina Baseline characteristic, predictor variable Myocardial infarction Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Baseline characteristic, predictor variable Codes for the condition Baseline characteristic, predictor variable | | | | census categories using |
| Smoking status Baseline characteristic, predictor variable Predictor variable Predict | | | | clinically coded |
| Alcohol use Baseline characteristic, predictor variable Baseline characteristic, predictor variable Body mass index (BMI) Body mass index (BMI) Body mass index (BMI) Baseline characteristic, predictor variable Body mass index (BMI) Baseline characteristic, predictor variable Censoring event Defined using most recent clinically recorded BMI information Death Censoring event Deregistration from GP Censoring event OPCRD Identified from coding in the clinical record Identified using clinical record Atrial fibrillation Baseline characteristic, predictor variable Angina Baseline characteristic, oPCRD Identified using clinical codes for the condition Myocardial infarction Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Stroke Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Baseline characteristic, oPCRD Identified using clinical codes for the condition Identified using clinical codes for the condition Baseline characteristic, oPCRD Identified using clinical codes for the condition Baseline characteristic, predictor variable Baseline characteristic, oPCRD Identified using clinical codes for the condition Baseline characteristic, predictor variable Baseline characteristic, oPCRD Identified using clinical codes for the condition Baseline characteristic, predictor variable Baseline characteristic, oPCRD Identified using clinical codes for the condition Baseline characteristic, predictor variable Baseline characteristic, oPCRD Identified using clinical codes for the condition | | | | ethnicity data |
| Alcohol use Baseline characteristic, predictor variable Body mass index (BMI) Death Censoring event Deregistration from GP Atrial fibrillation Baseline characteristic, predictor variable Angina Baseline characteristic, predictor variable Angina Baseline characteristic, predictor variable Myocardial infarction Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, oPCRD Jidentified using clinical codes for the condition Codes for the condition Codes for the condition Diabetes type Baseline characteristic, oPCRD Jidentified using clinical codes for the condition Diabetes type Baseline characteristic, oPCRD Jidentified using clinical codes for the condition Diabetes type Baseline characteristic, oPCRD Jidentified using clinical codes for the condition Diabetes type Baseline characteristic, oPCRD Jidentified using clinical codes for the condition Diabetes type Baseline characteristic, oPCRD Jidentified using clinical codes for the condition Codes for the condition Codes for the condition Decre Didentified using clinical codes for the condition Decre Didentified using clinical codes for the condition Chronic kidney disease Saseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Coper Didentified using clinical codes for the condition | Smoking status | Baseline characteristic, | OPCRD | Using most recent |
| Alcohol use Baseline characteristic, predictor variable Body mass index (BMI) Baseline characteristic, predictor variable Body mass index (BMI) Baseline characteristic, predictor variable Body mass index (BMI) Baseline characteristic, predictor variable Censoring event Death Censoring event Decrop Decrop Identified from coding in the clinical record in the clin | | predictor variable | | clinically recorded |
| Alcohol use Baseline characteristic, predictor variable Body mass index (BMI) Body mass index (Binical) Body massing motar recent (Inical) Body massing motar recent (Inical) Body massing motar recent (Inical) Body massing motar recent (Inical) Body massing motar recent (Inical) Body massi | | | | smoking status |
| Predictor variable Clinically recorded alcohol use status information | | | | information |
| Body mass index (BMI) | Alcohol use | Baseline characteristic, | OPCRD | Using most recent |
| Body mass index (BMI) Body mass index (BMI) Body mass index (BMI) Predictor variable Pred | | predictor variable | | clinically recorded |
| Body mass index (BMI) Baseline characteristic, predictor variable Censoring event OPCRD Identified from coding in the clinical record Deregistration from GP Censoring event OPCRD OPCRD Identified from coding in the clinical record Identified from coding in the clinical record Identified using clinical record Atrial fibrillation Baseline characteristic, predictor variable Angina Baseline characteristic, predictor variable Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Identified using clinical codes for the condition OPCRD Identified using clinical codes for the condition Identified using clinical codes for the condition OPCRD Identified using clinical codes for the condition Diabetes type Baseline characteristic, predictor variable Hyperlipidaemia Baseline characteristic, predictor variable | | | | alcohol use status |
| predictor variable Precent clinically recorded BMI information | | | | information |
| Death Censoring event OPCRD Identified from coding in the clinical record Deregistration from GP Censoring event OPCRD Identified from coding in the clinical record Atrial fibrillation Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Angina Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Myocardial infarction Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Congestive heart failure Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Stroke Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Diabetes type Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Hyperlipidaemia Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Hypertension Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition | Body mass index (BMI) | Baseline characteristic, | OPCRD | Defined using most |
| Death Censoring event OPCRD Identified from coding in the clinical record Deregistration from GP Censoring event OPCRD Identified from coding in the clinical record Atrial fibrillation Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Angina Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Myocardial infarction Baseline characteristic, predictor variable Codes for the condition Congestive heart failure Baseline characteristic, predictor variable Codes for the condition Stroke Baseline characteristic, predictor variable Codes for the condition Diabetes type Baseline characteristic, predictor variable Codes for the condition Hyperlipidaemia Baseline characteristic, predictor variable Codes for the condition Baseline characteristic, OPCRD Identified using clinical codes for the condition Hypertension Baseline characteristic, predictor variable Codes for the condition Chronic kidney disease stages 3-5 | | predictor variable | | recent clinically |
| Death Censoring event OPCRD Identified from coding in the clinical record Deregistration from GP Censoring event OPCRD Identified from coding in the clinical record Atrial fibrillation Baseline characteristic, predictor variable Angina Baseline characteristic, predictor variable Myocardial infarction Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Stroke Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Hyperlipidaemia Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 DPCRD Identified using clinical codes for the condition Identified using clinical codes for the condition | | | | recorded BMI |
| Deregistration from GP Censoring event OPCRD Identified from coding in the clinical record Atrial fibrillation Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Angina Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Myocardial infarction Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Congestive heart failure Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Stroke Baseline characteristic, oPCRD Identified using clinical codes for the condition Diabetes type Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Hyperlipidaemia Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Hypertension OPCRD Identified using clinical codes for the condition Chronic kidney disease stages 3-5 Baseline characteristic, oPCRD Identified using clinical codes for the condition | | | | information |
| Deregistration from GP Censoring event OPCRD Identified from coding in the clinical record Atrial fibrillation Baseline characteristic, predictor variable OPCRD Identified using clinical codes for the condition Angina Baseline characteristic, predictor variable Codes for the condition Myocardial infarction Baseline characteristic, predictor variable Codes for the condition Congestive heart failure Baseline characteristic, predictor variable Codes for the condition Stroke Baseline characteristic, predictor variable Codes for the condition Diabetes type Baseline characteristic, predictor variable Codes for the condition Hyperlipidaemia Baseline characteristic, predictor variable Codes for the condition Baseline characteristic, OPCRD Identified using clinical codes for the condition Hypertension Baseline characteristic, predictor variable Codes for the condition Chronic kidney disease stages 3-5 | Death | Censoring event | OPCRD | Identified from coding |
| Atrial fibrillation Baseline characteristic, predictor variable Angina Baseline characteristic, predictor variable Myocardial infarction Baseline characteristic, predictor variable Myocardial infarction Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Stroke Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Baseline characteristic, predictor variable Hyperlipidaemia Baseline characteristic, predictor variable Baseline characteristic, predictor variable Codes for the condition Hypertension Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 Identified using clinical codes for the condition Identified using clinical codes for the condition Identified using clinical codes for the condition Identified using clinical codes for the condition Identified using clinical codes for the condition | | | | in the clinical record |
| Atrial fibrillation Baseline characteristic, predictor variable Angina Baseline characteristic, predictor variable Baseline characteristic, predictor variable Myocardial infarction Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Stroke Baseline characteristic, predictor variable Codes for the condition Diabetes type Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Baseline characteristic, predictor variable Codes for the condition Hyperlipidaemia Baseline characteristic, predictor variable Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 Identified using clinical codes for the condition Identified using clinical codes for the condition | Deregistration from GP | Censoring event | OPCRD | Identified from coding |
| Angina Baseline characteristic, predictor variable Codes for the condition Myocardial infarction Baseline characteristic, predictor variable Codes for the condition Myocardial infarction Baseline characteristic, predictor variable Codes for the condition Congestive heart failure Baseline characteristic, predictor variable Codes for the condition Stroke Baseline characteristic, predictor variable Codes for the condition Diabetes type Baseline characteristic, predictor variable Codes for the condition Hyperlipidaemia Baseline characteristic, predictor variable Codes for the condition Hyperlipidaemia Baseline characteristic, predictor variable Codes for the condition Hypertension Baseline characteristic, predictor variable Codes for the condition Chronic kidney disease stages 3-5 | | | | in the clinical record |
| Angina Baseline characteristic, predictor variable Myocardial infarction Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Stroke Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Hyperlipidaemia Baseline characteristic, predictor variable Baseline characteristic, predictor variable Codes for the condition Hypertension Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 Baseline characteristic, predictor variable Baseline characteristic, predictor variable COPCRD Identified using clinical codes for the condition Identified using clinical codes for the condition | Atrial fibrillation | Baseline characteristic, | OPCRD | Identified using clinical |
| myocardial infarction Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Congestive heart failure Baseline characteristic, predictor variable Stroke Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Hyperlipidaemia Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 Baseline characteristic, predictor variable Baseline characteristic, predictor variable COPCRD Identified using clinical codes for the condition Identified using clinical codes for the condition Identified using clinical codes for the condition | | predictor variable | | codes for the condition |
| Myocardial infarctionBaseline characteristic,<br>predictor variableOPCRDIdentified using clinical<br>codes for the conditionCongestive heart failureBaseline characteristic,<br>predictor variableOPCRDIdentified using clinical<br>codes for the conditionStrokeBaseline characteristic,<br>predictor variableOPCRDIdentified using clinical<br>codes for the conditionDiabetes typeBaseline characteristic,<br>predictor variableOPCRDIdentified using clinical<br>codes for the conditionHyperlipidaemiaBaseline characteristic,<br>predictor variableOPCRDIdentified using clinical<br>codes for the conditionHypertensionBaseline characteristic,<br>predictor variableOPCRDIdentified using clinical<br>codes for the conditionChronic kidney disease<br>stages 3-5Baseline characteristic,<br>predictor variableOPCRDIdentified using clinical<br>codes for the condition | Angina | Baseline characteristic, | OPCRD | Identified using clinical |
| predictor variable codes for the condition Congestive heart failure Baseline characteristic, predictor variable codes for the condition Stroke Baseline characteristic, predictor variable codes for the condition Diabetes type Baseline characteristic, predictor variable codes for the condition Hyperlipidaemia Baseline characteristic, predictor variable codes for the condition Hyperlipidaemia Baseline characteristic, predictor variable codes for the condition Hypertension Baseline characteristic, predictor variable codes for the condition Chronic kidney disease stages 3-5 Baseline characteristic, predictor variable codes for the condition Codes for the condition Identified using clinical codes for the condition Identified using clinical codes for the condition Codes for the condition | | predictor variable | | codes for the condition |
| Congestive heart failure Baseline characteristic, predictor variable Stroke Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Baseline characteristic, OPCRD Diabetes type Baseline characteristic, predictor variable Hyperlipidaemia Baseline characteristic, oPCRD Hyperlipidaemia Baseline characteristic, oPCRD Hypertension Baseline characteristic, oPCRD Baseline characteristic, oPCRD Baseline characteristic, oPCRD Baseline characteristic, oPCRD Identified using clinical codes for the condition Codes for the condition Codes for the condition Identified using clinical codes for the condition Identified using clinical codes for the condition Codes for the condition Codes for the condition | Myocardial infarction | Baseline characteristic, | OPCRD | Identified using clinical |
| Stroke Baseline characteristic, OPCRD Identified using clinical codes for the condition Diabetes type Baseline characteristic, OPCRD Identified using clinical predictor variable codes for the condition Hyperlipidaemia Baseline characteristic, OPCRD Identified using clinical codes for the condition Hyperlipidaemia Baseline characteristic, OPCRD Identified using clinical codes for the condition Hypertension OPCRD Identified using clinical codes for the condition Baseline characteristic, OPCRD Identified using clinical codes for the condition Chronic kidney disease stages 3-5 | | predictor variable | | codes for the condition |
| Stroke Baseline characteristic, predictor variable Diabetes type Baseline characteristic, predictor variable Baseline characteristic, predictor variable Hyperlipidaemia Baseline characteristic, predictor variable | Congestive heart failure | Baseline characteristic, | OPCRD | Identified using clinical |
| predictor variable Diabetes type Baseline characteristic, OPCRD predictor variable Hyperlipidaemia Baseline characteristic, OPCRD predictor variable Baseline characteristic, OPCRD predictor variable Hypertension Baseline characteristic, OPCRD predictor variable Baseline characteristic, OPCRD predictor variable Chronic kidney disease stages 3-5 DPCRD Identified using clinical codes for the condition Identified using clinical codes for the condition | | predictor variable | | codes for the condition |
| Diabetes type Baseline characteristic, predictor variable Hyperlipidaemia Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 Baseline characteristic, predictor variable Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable | Stroke | Baseline characteristic, | OPCRD | Identified using clinical |
| predictor variable codes for the condition Hyperlipidaemia Baseline characteristic, predictor variable codes for the condition Hypertension Decemble Decemble Chronic kidney disease stages 3-5 predictor variable codes for the condition Codes for the condition dentified using clinical codes for the condition Codes for the condition dentified using clinical codes for the condition | | predictor variable | | codes for the condition |
| Hyperlipidaemia Baseline characteristic, predictor variable Baseline characteristic, predictor variable Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 Baseline characteristic, predictor variable Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 | Diabetes type | Baseline characteristic, | OPCRD | Identified using clinical |
| predictor variable codes for the condition Hypertension Baseline characteristic, predictor variable codes for the condition Chronic kidney disease stages 3-5 Codes for the condition codes for the condition OPCRD Identified using clinical codes for the condition | | predictor variable | | codes for the condition |
| Hypertension Baseline characteristic, predictor variable Chronic kidney disease stages 3-5 Baseline characteristic, oPCRD ocdes for the condition CPCRD Identified using clinical codes for the condition | Hyperlipidaemia | Baseline characteristic, | OPCRD | Identified using clinical |
| Hypertension predictor variable codes for the condition Chronic kidney disease stages 3-5 Baseline characteristic, OPCRD Identified using clinical codes for the condition | | predictor variable | | codes for the condition |
| predictor variable codes for the condition Chronic kidney disease stages 3-5 Baseline characteristic, OPCRD Identified using clinical codes for the condition | Hypertension | Baseline characteristic, | OPCRD | Identified using clinical |
| Chronic kidney disease predictor variable codes for the condition | Try per terision | predictor variable | | codes for the condition |
| stages 3-5 predictor variable codes for the condition | Chronic kidney disease | Baseline characteristic, | OPCRD | Identified using clinical |
| and lab test results | - | predictor variable | | codes for the condition |
| | Janges 5 5 | | | and lab test results |

| Chronic obstructive pulmonary disease, | Baseline characteristic, predictor variable | | |
|---|---|---|---|
| Asthma | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Chronic liver disease | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| dementia | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| immunotherapy use | Potential predictor | OPCRD | Identified using |
| | variable | | prescription records for |
| | | | immunotherapy |
| Phototherapy | Potential predictor OPCRD Identified usin | | Identified using |
| treatment | variable | | prescription records |
| | | | and clinical codes for |
| | | | phototherapy |

Read codes and SNOMED codes to be used to identify skin cancers

| Melanoma skin cancer | | | |
|---|---|---|--|
| Read V2 Code | Term<br>ID | Description | |
| BBE1. | All | [M] Melanoma NOS | |
| BBE10 | All | [M] Malignant melanoma, regressing | |
| BBE11 | All | [M] Desmoplastic melanoma, malignant | |
| 7G03J | All | Excision of melanoma | |
| BBE4. | All | [M] Balloon cell melanoma | |
| BBEA. | All | [M] Amelanotic melanoma | |
| BBEC. | All | [M] Malignant melanoma in junctional naevus | |
| BBED. | All | [M] Precancerous melanosis NOS | |
| BBEE. | All | [M] Malignant melanoma in precancerous melanosis | |
| BBEF. | All | [M] Hutchinson's melanotic freckle | |
| BBEG. | All | [M] Malignant melanoma in Hutchinson's melanotic freckle | |
| BBEG0 | All | [M]Acral lentingous melanoma, malignant | |
| ВВЕН. | All | [M] Superficial spreading melanoma | |
| ВВЕМ. | All | [M] Malignant melanoma in giant pigmented naevus | |
| BBEP. | All | [M] Epitheliod cell melanoma | |
| BBEQ. | All | [M] Spindle cell melanoma, NOS | |
| BBER. | All | [M] Spindle cell melanoma, type A | |
| BBES. | All | [M] Spindle cell melanoma, type B | |
| ВВЕТ. | All | [M] Mixed epitheliod and spindle melanoma | |
| BBEX. | All | [M] Melanoma in situ | |
| BBEz. | All | [M] Naevi or melanoma, NOS | |
| 14250 | All | H/O Malignant Melanoma | |
| B828. | All | Melanoma in situ of skin | |
| B8280 | All | Melanoma in situ of lip | |
| B8281 | All | Melanoma in situ of eyelid, including canthus | |
| B8282 | All | Melanoma in situ of ear and external auricular canal | |
| B8283 | All | Melanoma in situ of scalp and neck | |
| B8284 | All | Melanoma in situ of trunk | |
| B8285 | All | Melanoma in situ of upper limb, including shoulder | |
| B8286 | All | Melanoma in situ of lower limb, including hip |
|-------|-----|-----------------------------------------------------------|
| B8287 | All | Melanoma in situ of scalp |
| B8288 | All | Melanoma in situ of back of hand |
| B8289 | All | Melanoma in situ of back |
| B828W | All | Melanoma in situ, unspecified |
| B828X | All | Melanoma in situ of other and unspecified parts of face |
| B509. | All | Malignant melanoma of eye |
| B32 | All | Malignant melanoma of skin |
| B321. | All | Malignant melanoma of eyelid, including canthus |
| B322. | All | Malignant melanoma of ear and external auricular canal |
| B320. | All | Malignant melanoma of lip |
| B3220 | All | Malignant melanoma of auricle (ear) |
| B3221 | All | Malignant melanoma of external auditory meatus |
| | | Malignant melanoma of ear and external auricular canal |
| B322z | All | NOS |
| B323. | All | Malignant melanoma of other and unspecified parts of face |
| B3230 | All | Malignant melanoma of external surface of cheek |
| B3231 | All | Malignant melanoma of chin |
| B3232 | All | Malignant melanoma of eyebrow |
| B3233 | All | Malignant melanoma of forehead |
| B3234 | All | Malignant melanoma of external surface of nose |
| B3235 | All | Malignant melanoma of temple |
| B323z | All | Malignant melanoma of face NOS |
| B324. | All | Malignant melanoma of scalp and neck |
| B3240 | All | Malignant melanoma of scalp |
| B3241 | All | Malignant melanoma of neck |
| B324z | All | Malignant melanoma of scalp and neck NOS |
| B325. | All | Malignant melanoma of trunk excluding scrotum |
| B3250 | All | Malignant melanoma of axilla |
| B3251 | All | Malignant melanoma of breast |
| B3252 | All | Malignant melanoma of buttock |
| B3253 | All | Malignant melanoma of groin |
| B3254 | All | Malignant melanoma of perianal skin |
| B3255 | All | Malignant melanoma of perineum |

| B3256 | All | Malignant melanoma of umbilicus |
|-------|-----|---------------------------------------------------|
| B3257 | All | Malignant melanoma of back |
| B3258 | All | Malignant melanoma of chest wall |
| B325z | All | Malignant melanoma of trunk excluding scrotum NOS |
| B326. | All | Malignant melanoma of upper limb and shoulder |
| B3260 | All | Malignant melanoma of shoulder |
| B3261 | All | Malignant melanoma of upper arm |
| B3262 | All | Malignant melanoma of forearm |
| B3263 | All | Malignant melanoma of hand |
| B3264 | All | Malignant melanoma of finger |
| B3265 | All | Malignant melanoma of thumb |
| B326z | All | Malignant melanoma of upper limb and shoulder NOS |
| B327. | All | Malignant melanoma of lower limb and hip |
| B3270 | All | Malignant melanoma of hip |
| B3271 | All | Malignant melanoma of thigh |
| B3272 | All | Malignant melanoma of knee |
| B3273 | All | Malignant melanoma of popliteal fossa area |
| B3274 | All | Malignant melanoma of lower leg |
| B3275 | All | Malignant melanoma of ankle |
| B3276 | All | Malignant melanoma of heel |
| B3277 | All | Malignant melanoma of foot |
| B3278 | All | Malignant melanoma of toe |
| B3279 | All | Malignant melanoma of great toe |
| B327z | All | Malignant melanoma of lower limb and hip NOS |
| B328. | All | Malignant melanoma stage IA |
| B329. | All | Malignant melanoma stage IB |
| B32A. | All | Malignant melanoma stage IIA |
| B32B. | All | Malignant melanoma stage IIB |
| B32C. | All | Malignant melanoma stage IIC |
| B32D. | All | Malignant melanoma stage IIIA |
| B32E. | All | Malignant melanoma stage IIIB |
| B32F. | All | Malignant melanoma stage IIIC |
| B32G. | All | Malignant melanoma stage IV M1a |
| В32Н. | All | Malignant melanoma stage IV M1b |

| В32Ј. | All | Malignant melanoma stage IV M1c |
|---|---|---|
| В32у. | All | Malignant melanoma of other specified skin site |
| B32y0 | All | Overlapping malignant melanoma of skin |
| B32z. | All | Malignant melanoma of skin NOS |
| 4M3 | All | Breslow depth for staging for melanoma |
| D. LOWYO C. L | Term | B |
| Read CTV3 Code | ID<br>All | Description Excision of melanoma |
| XSHw6 | All | Clark melanoma level 3 |
| XSHw7 | All | Clark melanoma level 4 |
| XSHw8 | All | Clark melanoma level 5 |
| 14250 | All | H/O Malignant melanoma |
| XSHw4 | All | Clark melanoma level 1 |
| XSHw5 | All | Clark melanoma level 2 |
| B8280 | All | Melanoma in situ of lip |
| X78TH | All | In situ melanoma of skin |
| B8281 | All | Melanoma in situ of eyelid, including canthus |
| B8282 | All | Melanoma in situ of ear and external auricular canal |
| B8283 | All | Melanoma in situ of scalp and neck |
| B8284 | All | Melanoma in situ of trunk |
| B8285 | All | Melanoma in situ of upper limb, including shoulder |
| B8286 | All | Melanoma in situ of lower limb, including hip |
| XaFsS | All | Melanoma in situ of scalp |
| XaFsU | All | Melanoma in situ of back of hand |
| XaFw7 | All | Melanoma in situ of back |
| XaFsT | All | Melanoma in situ of neck |
| ByuF5 | All | [X] Melanoma in situ of other and unspecified parts of face |
| Xa99Y | All | Lentingo maligna melanoma |
| X78TD | All | Nodular melanoma of skin |
| B3270 | All | Malignant melanoma of hip |
| B3278 | All | Malignant melanoma of toe |
| XM0ps | All | Malignant melanoma of eye |
| B320. | All | Malignant melaoma of lip |
| B3263 | All | Malignant melaoma of hand |
| B3276 | All | Malignant melanoma of heel |

| X78bc | All | Malignant melanoma of iris |
|-------|-----|-----------------------------------------------------------|
| B3272 | All | Malignant melanoma of knee |
| B3241 | All | Malignant melanoma of neck |
| B32 | All | Malignant melanoma of skin |
| XaclU | All | Malignant melanoma stage IA |
| XaclV | All | Malignant melanoma stage IB |
| XaclW | All | Malignant melanoma stage IIA |
| XaclX | All | Malignant melanoma stage IIB |
| XaclY | All | Malignant melanoma stage IIC |
| XaclZ | All | Malignant melanoma stage IIIA |
| Xacla | All | Malignant melanoma stage IIIB |
| Xaclb | All | Malignant melanoma stage IIIC |
| Xacld | All | Malignant melanoma stage IV M1a |
| Xacle | All | Malignant melanoma stage IV M1b |
| Xaclf | All | Malignant melanoma stage IV M1c |
| XaFrT | All | Local recurrence of malignant melanoma of skin |
| X78TC | All | Superficial spreading malignant melanoma of skin |
| X78TD | All | Nodular malignant melanoma of skin |
| Xa0CE | All | Amelanotic malignant melanoma of skin |
| X78TE | All | Acral lentiginous melanoma of skin |
| XaBAw | All | Malignant blue naevus of skin |
| X78TF | All | Malignant melanoma arising in intradermal naevus |
| X78TG | All | Malignant melanoma arising in congenital naevus |
| XM0ps | All | Malignant melanoma of eye |
| B32 | All | Malignant melanoma of skin |
| B321. | All | Malignant melanoma of eyelid, including canthus |
| B322. | All | Malignant melanoma of ear and external auricular canal |
| B320. | All | Malignant melanoma of lip |
| B3220 | All | Malignant melanoma of auricle (ear) |
| B3221 | All | Malignant melanoma of external auditory meatus |
| | | Malignant melanoma of ear and external auricular canal |
| B322z | All | NOS |
| B323. | All | Malignant melanoma of other and unspecified parts of face |
| B3230 | All | Malignant melanoma of external surface of cheek |

| B3231 | All | Malignant melanoma of chin |
|-------|-----|---------------------------------------------------|
| B3232 | All | Malignant melanoma of eyebrow |
| B3233 | All | Malignant melanoma of forehead |
| B3234 | All | Malignant melanoma of external surface of nose |
| B3235 | All | Malignant melanoma of temple |
| B323z | All | Malignant melanoma of face NOS |
| B324. | All | Malignant melanoma of scalp and neck |
| B3240 | All | Malignant melanoma of scalp |
| B3241 | All | Malignant melanoma of neck |
| B324z | All | Malignant melanoma of scalp and neck NOS |
| B325. | All | Malignant melanoma of trunk excluding scrotum |
| B3250 | All | Malignant melanoma of axilla |
| B3251 | All | Malignant melanoma of breast |
| B3252 | All | Malignant melanoma of buttock |
| B3253 | All | Malignant melanoma of groin |
| B3254 | All | Malignant melanoma of perianal skin |
| B3255 | All | Malignant melanoma of perineum |
| B3256 | All | Malignant melanoma of umbilicus |
| XaClv | All | Malignant melanoma of back |
| XaEGU | All | Malignant melanoma of chest wall |
| B325z | All | Malignant melanoma of trunk excluding scrotum NOS |
| B326. | All | Malignant melanoma of upper limb and shoulder |
| B3260 | All | Malignant melanoma of shoulder |
| B3261 | All | Malignant melanoma of upper arm |
| B3262 | All | Malignant melanoma of forearm |
| B3263 | All | Malignant melanoma of hand |
| B3264 | All | Malignant melanoma of finger |
| B3265 | All | Malignant melanoma of thumb |
| B326z | All | Malignant melanoma of upper limb and shoulder NOS |
| B327. | All | Malignant melanoma of lower limb and hip |
| B3270 | All | Malignant melanoma of hip |
| B3271 | All | Malignant melanoma of thigh |
| B3272 | All | Malignant melanoma of knee |
| B3273 | All | Malignant melanoma of popliteal fossa area |

| B3274 | All | Malignant melanoma of lower leg |
|-------|-----|----------------------------------------------------|
| B3275 | All | Malignant melanoma of ankle |
| B3276 | All | Malignant melanoma of heel |
| B3277 | All | Malignant melanoma of foot |
| B3278 | All | Malignant melanoma of toe |
| B3279 | All | Malignant melanoma of great toe |
| B327z | All | Malignant melanoma of lower limb and hip NOS |
| В32у. | All | Malignant melanoma of other specified skin site |
| B32y0 | All | Overlapping malignant melanoma of skin |
| B32z. | All | Malignant melanoma of skin NOS |
| Byu41 | All | [X] Malignant melanoma of skin unspecified |
| XE1yl | All | Malignant melanoma of head and neck |
| XE1yn | All | Malignant melanoma of trunk |
| X78bV | All | Malignant melanoma of cornea |
| XE1yp | All | Malignant melanoma of upper limb |
| XE1yr | All | Malignant melanoma of lower limb |
| Xa0Di | All | Malignant melanoma of anus |
| X78Xx | All | Malignant melanoma of vulva |
| X78bw | All | Malignant melanoma of choriod |
| XM0ps | All | Malignant melanoma of eye |
| Xa0RU | All | Malignant melanoma of meninges |
| XaE6A | All | Melanoma associated retinopathy |
| ByuF6 | All | [X] Melanoma in situ of other sites |
| XSNL7 | All | Breslow depth for staging of melanoma |
| X78Fn | All | TNM Malignant melanoma of skin staging |
| X78G8 | All | TNM Malignant melanoma of uvea staging |
| X78G9 | All | TNM Malignant melanoma of iris staging |
| X78GA | All | TNM Malignant melanoma of ciliary body staging |
| X78GB | All | TNM Malignant melanoma of choriod staging |
| X78G5 | All | TNM Malignant melanoma of eyelid staging |
| XaFrd | All | Metastasis from malignant melanoma of skin |
| X78G7 | All | TNM Malignant melanoma of conjunctiva staging |
| Byu4. | All | [X] Melanoma and other malignant neoplasms of skin |

| | Term | |
|-------------|------|---------------------------------------------------------|
| SNOMED Code | ID | Description |
| SNOWLD Code | 1D | • |
| | | Malignant melanoma, no International Classification of |
| | | Diseases for Oncology subtype (morphologic abnormality) |
| 2092003 | | |
| 255012009 | | Malignant melanoma of iris (disorder) |
| 399475009 | | Minimal deviation melanoma (morphologic abnormality) |
| 77986002 | | Melanoma in situ (morphologic abnormality) |
| 2142002 | | Nodular melanoma (morphologic abnormality) |
| 399521000 | | Necrotic melanoma (morphologic abnormality) |
| 423673009 | | Malignant melanoma of retina (disorder) |
| 372244006 | | Malignant melanoma (disorder) |
| 726420002 | | Meningeal melanoma (morphologic abnormality) |
| 276751004 | | Amelanotic malignant melanoma of skin (disorder) |
| 70594002 | | Amelanotic melanoma (morphologic abnormality) |
| 276821000 | | Malignant melanoma of anus (disorder) |
| 103419001 | | Clark's melanoma level (observable entity) |
| 177281002 | | Excision of melanoma (procedure) |
| 68827007 | | Spindle cell melanoma (morphologic abnormality) |
| 115223002 | | Nevus AND/OR melanoma (morphologic abnormality) |
| 255015006 | | Malignant melanoma of ciliary body (disorder) |
| 39274007 | | Balloon cell melanoma (morphologic abnormality) |
| 21165006 | | Clark melanoma level 3 (finding) |
| 83284001 | | Clark melanoma level 1 (finding) |
| 276822007 | | Malignant melanoma of rectum (disorder) |
| 50542000 | | Clark melanoma level 2 (finding) |
| 161432005 | | History of malignant melanoma (situation) |
| 16034002 | | Clark melanoma level 5 (finding) |
| 1556006 | | Clark melanoma level 4 (finding) |
| 109272006 | | Melanoma in situ of lip (disorder) |
| 109278005 | | Melanoma in situ of ear (disorder) |
| 128731008 | | Meningeal melanomatosis (morphologic abnormality) |
| 109296001 | | Melanoma in situ of hip (disorder) |
| 315230006 | | Melanoma in situ of back (disorder) |
| 109266006 | | Melanoma in situ of skin (disorder) |
| 302837001 | | Lentigo maligna melanoma (disorder) |
| 109282007 | | Melanoma in situ of neck (disorder) |
| 254731001 | | Nodular malignant melanoma of skin (disorder) |
| | | Malignant melanoma in Hutchinson's melanotic freckle |
| 44474009 | | (morphologic abnormality) |
| 109270003 | | Melanoma in situ of face (disorder) |
| 816204007 | | Nodular melanoma of mucous membrane (disorder) |
| 109266006 | | Melanoma in situ of skin (disorder) |
| 274087000 | | Malignant melanoma of eye (disorder) |
| 37138001 | | Epithelioid cell melanoma (morphologic abnormality) |
| 707361004 | | Malignant melanoma of frontal sinus (disorder) |
| 109276009 | | Melanoma in situ of scalp (disorder) |
| 188030005 | | Malignant melanoma of lip (disorder) |
| 109284008 | | Melanoma in situ of trunk (disorder) |

| 188068007 | Malignant melanoma of hip (disorder) |
|---|---|
| 698287002 | Malignant melanoma of gum (disorder) |
| 188076009 | Malignant melanoma of toe (disorder) |
| 396368008 | Skin melanoma TNM finding (finding) |
| 310498001 | Malignant melanoma of back (disorder) |
| 276821000 | Malignant melanoma of anus (disorder) |
| 255012009 | Malignant melanoma of iris (disorder) |
| 188063003 | Malignant melanoma of hand (disorder) |
| 188075008 | Malignant melanoma of foot (disorder) |
| 188070003 | Malignant melanoma of knee (disorder) |
| 93655004 | Malignant melanoma of skin (disorder) |
| 399705007 | Uveal melanoma TNM finding (finding) |
| 188038003 | Malignant melanoma of chin (disorder) |
| 399475009 | Minimal deviation melanoma (morphologic abnormality) |
| 188074007 | Malignant melanoma of heel (disorder) |
| 188046002 | Malignant melanoma of neck (disorder) |
| 698285005 | Malignant melanoma of ethmoid sinus (disorder) |
| 188052001 | Malignant melanoma of groin (disorder) |
| 866072004 | Malignant melanoma of orbit (disorder) |
| 403923002 | Spindle cell malignant melanoma (disorder) |
| 956331000000107 | Malignant melanoma stage IA (finding) |
| 956351000000107 | |
| 188045003 | Malignant melanoma stage IB (finding) Malignant melanoma of scalp (disorder) |
| 269579005 | Malignant melanoma of trunk (disorder) |
| 188069004 | |
| | Malignant melanoma of thigh (disorder) Malignant melanoma of accessory sinus (disorder) |
| 707350007 | |
| 698288007 | Malignant melanoma of maxillary sinus (disorder) |
| 68827007 | Spindle cell melanoma (morphologic abnormality) |
| 399634005<br>188073001 | Choroidal melanoma, diffuse (morphologic abnormality) |
| | Malignant melanoma of ankle (disorder) |
| 254896002 | Malignant melanoma of vulva (disorder) |
| 188065005 | Malignant melanoma of thumb (disorder) |
| 188049009 | Malignant melanoma of axilla (disorder) |
| 188050009<br>707362006 | Malignant melanoma of breast (disorder) |
| | Malignant melanoma of sphenoidal sinus (disorder) |
| 956411000000108 | Malignant melanoma stage IIC (finding |
| 128732001 | Mucosal lentiginous melanoma (morphologic abnormality) |
| 403927001 | Malignant melanoma of nail apparatus (disorder) |
| 231834005 | Malignant melanoma of eyelid (disorder) |
| 423673009 | Malignant melanoma of retina (disorder) |
| 698042007 | Malignant melanoma of tongue (disorder) |
| 385347004 | Clark melanoma level finding (finding) |
| 188042000 | Malignant melanoma of temple (disorder) |
| 698286006 | Malignant melanoma of palate (disorder) |
| 956371000000109 | Malignant melanoma stage IIA (finding) |
| 109292004 | Melanoma in situ of shoulder (disorder) |
| 188064009 | Malignant melanoma of finger (disorder) |
| 956391000000108 | Malignant melanoma stage IIB (finding) |
| 188051008 | Malignant melanoma of buttock (disorder) |

| 05647400000400 | |
|---|---|
| 956471000000103 | Malignant melanoma stage IIIC (finding) |
| 956431000000100 | Malignant melanoma stage IIIA (finding) |
| 255021005 | Malignant melanoma of choroid (disorder) |
| 403921000 | Borderline malignant melanoma (disorder) |
| 402559007 | Congenital malignant melanoma (disorder) |
| 372156000 | Malignant melanoma - category (morphologic abnormality) |
| 24653009 | Spindle cell melanoma, type A (morphologic abnormality) |
| 127330008 | Melanoma in situ by body site (disorder) |
| 443493003 | Metastatic malignant melanoma (disorder) |
| 188062008 | Malignant melanoma of forearm (disorder) |
| 40244008 | Spindle cell melanoma, type B (morphologic abnormality) |
| 93223008 | Malignant melanoma of skin of eyebrow (disorder) |
| 399660006 | Ring melanoma of ciliary body (disorder) |
| 698287002 | Malignant melanoma of gum (disorder) |
| 385371006 | International Federation of Gynecology and Obstetrics stage for vulvar melanoma (observable entity) |
| 51757004 | Desmoplastic melanoma, malignant (morphologic abnormality) |
| 109290007 | Melanoma in situ of upper limb (disorder) |
| 274087000 | Malignant melanoma of eye (disorder) |
| 109294003 | Melanoma in situ of lower limb (disorder) |
| 109266006 | Melanoma in situ of skin (disorder) |
| 188060000 | Malignant melanoma of shoulder (disorder) |
| 403925009 | Neurotropic malignant melanoma (disorder) |
| 55320002 | Superficial spreading melanoma (morphologic abnormality) |
| 188054000 | Malignant melanoma of perineum (disorder) |
| 402562005 | Malignant melanoma animal-type (disorder) |
| 402302003 | Malignant melanoma, metastatic (morphologic |
| 372158004 | abnormality) |
| | Neurotropic melanoma, malignant (morphologic |
| 399644007 | abnormality) |
| 277530005 | Malignant melanoma of meninges (disorder) |
| 302837001 | Lentigo maligna melanoma (disorder) |
| 188040008 | Malignant melanoma of forehead (disorder) |
| | Malignant melanoma, regressing (morphologic |
| 39896009 | abnormality) |
| 403922007 | Balloon cell malignant melanoma (disorder) |
| 188061001 | Malignant melanoma of upper arm (disorder) |
| 721627007 | Malignant melanoma of esophagus (disorder) |
| 2 231 | International Federation of Gynecology and Obstetrics |
| 106246001 | staging system for vulvar melanoma (tumor staging) |
| 188072006 | Malignant melanoma of lower leg (disorder) |
| 403924008 | Desmoplastic malignant melanoma (disorder) |
| 188055004 | Malignant melanoma of umbilicus (disorder) |
| 956551000000106 | Malignant melanoma stage IV M1c (finding) |
| | Desmoplastic melanoma, malignant (morphologic |
| 51757004 | abnormality) |
| 722689005 | Melanoma in situ of conjunctiva (disorder) |
| 956531000000104 | Malignant melanoma stage IV M1b (finding) |
| 188077000 | Malignant melanoma of great toe (disorder) |

| | Malignant melanoma in precancerous melanosis |
|------------------|---------------------------------------------------------|
| 18450009 | (morphologic abnormality) |
| 312941005 | Melanoma-associated retinopathy (disorder) |
| 956511000000107 | Malignant melanoma stage IV M1a (finding) |
| 1556006 | Clark melanoma level 4 (finding) |
| 315036008 | Melanoma in situ of back of hand (disorder) |
| 16034002 | Clark melanoma level 5 (finding) |
| 307603002 | Malignant blue nevus of skin (disorder) |
| 313248004 | Malignant melanoma of chest wall (disorder) |
| 93640008 | Malignant melanoma of skin of lip (disorder) |
| 93637008 | Malignant melanoma of skin of hip (disorder) |
| 93650009 | Malignant melanoma of skin of toe (disorder) |
| 255004001 | Malignant melanoma of conjuctiva (disorder) |
| 109268007 | Melanoma in situ of non-skin site (disorder) |
| 271944004 | Clear cell sarcoma (morphologic abnormality) |
| 93220006 | Malignant melanoma of skin of ear (disorder) |
| 385345007 | Clark system for melanoma staging (tumor staging) |
| 109288006 | Melanoma in situ of perianal skin (disorder) |
| 403926005 | Malignant melanoma of oral cavity (disorder) |
| 93214005 | Malignant melanoma of skin of back (disorder) |
| 93638003 | Malignant melanoma of skin of knee (disorder) |
| 109266006 | Melanoma in situ of skin (disorder) |
| 109286005 | Melanoma in situ of skin of breast (disorder) |
| 93642000 | Malignant melanoma of skin of neck (disorder) |
| 93636004 | Malignant melanoma in skin of hand (disorder) |
| 93227009 | Malignant melanoma of skin of foot (disorder) |
| 33227003 | Clear cell sarcoma (except of Kidney M-89643) |
| 12622007 | (morphologic abnormality) |
| 385348009 | Breslow depth finding for melanoma (finding) |
| 93225001 | Malignant melanoma of skin of face (disorder) |
| 93643005 | Malignant melanoma of skin of nose (disorder) |
| 723281005 | Primary malignant melanoma of anus (disorder) |
| 698040004 | Malignant melanoma of nasal cavity (disorder) |
| 106243009 | Breslow depth staging for melanoma (observable entity) |
| 1080941000119109 | Malignant melanoma of left choroid (disorder) |
| 93219000 | Malignant melanoma of skin of chin (disorder) |
| 109296001 | Melanoma in situ of hip (disorder) |
| 402561003 | Malignant melanoma of soft tissues (disorder) |
| 254732008 | Acral lentiginous malignant melanoma of skin (disorder) |
| 447712006 | Malignant melanoma of skin of anus (disorder) |
| 385346008 | Breslow system for melanoma staging (tumor staging) |
| 269578002 | Malignant melanoma of head and neck (disorder) |
| 448298007 | Malignant melanoma of skin of penis (disorder) |
| 448300007 | Malignant melanoma of skin of vulva (disorder) |
| 1080981000119100 | Malignant melanoma of right choroid (disorder) |
| 698044008 | Malignant melanoma of palatine arch (disorder) |
| 698045009 | Malignant melanoma of buccal mucosa (disorder) |
| 1251000119106 | History of melanoma in situ of skin (situation) |
| 396368008 | Skin melanoma TNM finding (finding) |
| 33030000 | JAMI Inclandina Hawi iniding (iniding) |

| 93209006 Malignant melanoma of perianal skin (disorder) 93211002 Malignant melanoma of skin of ankle (disorder) 932117003 Malignant melanoma of skin of cheek (disorder) 93218008 Malignant melanoma of skin of cheek (disorder) 93218005 Malignant melanoma of skin of cheek (disorder) 93212005 Malignant melanoma of skin of cheek (disorder) 93212006 Melanoma in situ of back (disorder) 188033007 Malignant melanoma of savin of leow (disorder) 93654000 Malignant melanoma of skin of wrist (disorder) 93654000 Malignant melanoma of skin of wrist (disorder) 93664000 Malignant melanoma of skin of trunk (disorder) 93230002 Malignant melanoma of skin of triph (disorder) 93230002 Malignant melanoma of skin of scalp (disorder) 93230002 Malignant melanoma of skin of scalp (disorder) 93230000 Malignant melanoma of skin of scalp (disorder) 9324000 Minimal deviation malignant melanoma (disorder) 93226000 Malignant melanoma of unknown origin (disorder) 9322600 Malignant melanoma of skin of finger (disorder) 93224002 Malignant melanoma of skin of finger (disorder) 93224002 Malignant melanoma of skin of scalp (disorder) 93224002 Malignant melanoma of skin of scalp (disorder) 93221000119100 Melanoma in situ of right upper limb (disorder) 10927609 Melanoma in situ of right lower limb (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of scalp (disorder) 93213004 Malignant melanoma of skin of swalla (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 93213007 Malignant melanoma of skin of forenem (disorder) 93213008 Malignant melanoma of skin of forerem (disorder) 93223008 Malign | 726019003 | Familial malignant melanoma of skin (disorder) |
|---|---|---|
| Malignant melanoma of skin of ankle (disorder) 93217003 Malignant melanoma of skin of cheek (disorder) 93218008 Malignant melanoma of skin of cheek (disorder) 93218008 Malignant melanoma of skin of chest (disorder) 93221005 Malignant melanoma of skin of chest (disorder) 93221006 Melanoma in situ of back (disorder) 93653000 Malignant melanoma of auricle (ear) (disorder) 93654000 Malignant melanoma of skin of wrist (disorder) 93654000 Malignant melanoma of skin of trunk (disorder) 93654000 Malignant melanoma of skin of trunk (disorder) 93649009 Malignant melanoma of skin of scalp (disorder) 93230002 Malignant melanoma of skin of scalp (disorder) 93230002 Malignant melanoma of skin of scalp (disorder) 93246002 Malignant melanoma of skin of scalp (disorder) 93290004 Malignant melanoma of skin of scalp (disorder) 93226000 Malignant melanoma of unknown origin (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 93224002 Malignant melanoma of skin of eyelid (disorder) 93224002 Malignant melanoma of skin of eyelid (disorder) 93224002 Malignant melanoma of skin of scalp (disorder) 93221000119100 Melanoma in situ of right lower limb (disorder) 9322100019107 Melanoma in situ of right lower limb (disorder) 93213000 Malignant melanoma of skin of scalp (disorder) 93213000 Primary malignant melanoma of skin (disorder) 93213000 Primary malignant melanoma of skin (disorder) 93213000 Malignant melanoma of skin of buttock (disorder) 93223000 Malignant melanoma of skin of buttock (disorder) 93223000 Malignant melanoma of skin of scrotum (disorder) 93223000 Malignant melanoma of skin of scrotum (disorder) 93223000 Malignant melanoma | | |
| Malignant melanoma of skin of cheek (disorder) 93218008 Malignant melanoma of skin of cheek (disorder) 93218008 Malignant melanoma of skin of clibow (disorder) 315230006 Melanoma in situ of back (disorder) 188033007 Malignant melanoma of skin of wrist (disorder) 93654000 Malignant melanoma of skin of trunk (disorder) 93654000 Malignant melanoma of skin of trunk (disorder) 93654009 Malignant melanoma of skin of trunk (disorder) 93649009 Malignant melanoma of skin of trunk (disorder) 93230002 Malignant melanoma of skin of scalp (disorder) 93290002 Malignant melanoma of skin of scalp (disorder) 9399705007 Uveal melanoma TNM finding (finding) 403920004 Minimal deviation malignant melanoma (disorder) 424190005 Malignant melanoma of skin of finger (disorder) 424190005 Malignant melanoma of skin of finger (disorder) 115561000119102 History of malignant melanoma of eye (situation) 93224002 Malignant melanoma of skin of eyelid (disorder) 1352161000119100 Melanoma in situ of right upper limb (disorder) 109276009 Melanoma in situ of right upper limb (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of preast (disorder) 93213006 Malignant melanoma of skin of preast (disorder) 93213007 Malignant melanoma of skin of scalp (disorder) 93213008 Malignant melanoma of skin of scalp (disorder) 93213009 Malignant melanoma of skin of scalp (disorder) 93213000 Malignant melanoma of skin of scalp (disorder) 93223000 Malignant melanoma of skin of scalp (disorder) 93223000 Malignant melanom | | |
| Malignant melanoma of skin of chest (disorder) 33221005 Malignant melanoma of skin of elbow (disorder) 315230006 Melanoma in situ of back (disorder) 188033007 Malignant melanoma of auricle (ear) (disorder) 93654000 Malignant melanoma of skin of wrist (disorder) 93654000 Malignant melanoma of skin of trunk (disorder) 93664000 Malignant melanoma of skin of trunk (disorder) 93664000 Malignant melanoma of skin of trunk (disorder) 93230002 Malignant melanoma of skin of groin (disorder) 93230002 Malignant melanoma of skin of groin (disorder) 939705007 Uveal melanoma TNM finding (finding) 403920004 Minimal deviation malignant melanoma (disorder) 93226000 Malignant melanoma of unknown origin (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 115561000119102 History of malignant melanoma of eye (situation) 93224002 Malignant melanoma of skin of eyelid (disorder) 932216000 Melanoma in situ of right upper limb (disorder) 932216000 Melanoma in situ of right upper limb (disorder) 932216000 Melanoma in situ of skin of scalp (disorder) 93211000119107 Melanoma in situ of skin of scalp (disorder) 93215006 Malignant melanoma of skin of breast (disorder) 93215006 Malignant melanoma of skin of breast (disorder) 93215006 Malignant melanoma of skin of situla (disorder) 93215006 Malignant melanoma of skin of situla (disorder) 93215006 Malignant melanoma of skin of breast (disorder) 93215006 Malignant melanoma of skin of breast (disorder) 93215000 Primary malignant melanoma of vagina (disorder) 93215000 Primary malignant melanoma of skin | | |
| Malignant melanoma of skin of elbow (disorder) 315230006 Melanoma in situ of back (disorder) 93654000 Malignant melanoma of auricle (ear) (disorder) 93654000 Malignant melanoma of skin of virist (disorder) 93654008 Malignant melanoma of skin of trunk (disorder) 93654009 Malignant melanoma of skin of trunk (disorder) 93649009 Malignant melanoma of skin of skin of lostorder) 93230002 Malignant melanoma of skin of scalp (disorder) 93230002 Malignant melanoma of skin of scalp (disorder) 939705007 Uveal melanoma TNM finding (finding) 403920004 Minimal deviation malignant melanoma (disorder) 424190005 Malignant melanoma of unknown origin (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 93226000 Malignant melanoma of skin of scalp (disorder) 93224002 Malignant melanoma of skin of seyelid (disorder) 93224002 Malignant melanoma of skin of seyelid (disorder) 93224002 Malignant melanoma of skin of scalp (disorder) 93224000 Melanoma in situ of right lower limb (disorder) 932161000119100 Melanoma in situ of right lower limb (disorder) 932161000119107 Melanoma in situ of skin of scalp (disorder) 93215000 Superficial spreading melanoma (morphologic abnormality) 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 921565003 Primary malignant melanoma of cornea (disorder) 9216751004 Amelanotic malignant melanoma of skin (disorder) 926765003 Primary malignant melanoma of skin (disorder) 93213000 Malignant melanoma of skin of scrotum (disorder) 93213000 Malignant melanoma of skin of skin of scrotum (disorder) 93216007 Malignant melanoma of skin of skin of scrotum (disorder) 93216007 Malignant melanoma of skin of skin of scrotum (disorder) 93228004 Malignant melanoma of skin of scrotum (disorder) 93228004 Malignant melanoma of skin of scrotum (disorder) 93228004 Malignant melanoma of skin of scrotum (disorder) 93228004 Malignant melanoma of skin of scrotum (disorder) 93228007 Malignant melanoma o | | |
| Melanoma in situ of back (disorder) 188033007 Malignant melanoma of auricle (ear) (disorder) 93654000 Malignant melanoma of skin of wrist (disorder) 93651008 Malignant melanoma of skin of trunk (disorder) 93649009 Malignant melanoma of skin of trunk (disorder) 93230002 Malignant melanoma of skin of groin (disorder) 9324002 Malignant melanoma of skin of groin (disorder) 939464002 Malignant melanoma of skin of scalp (disorder) 9399705007 Uveal melanoma TNM finding (finding) 403920004 Malignant melanoma of skin of scalp (disorder) 93226000 Malignant melanoma of skin of signer (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 93224002 Malignant melanoma of skin of finger (disorder) 93224002 Malignant melanoma of skin of finger (disorder) 93224002 Malignant melanoma of skin of eyelid (disorder) 93221000 Melanoma in situ of right upper limb (disorder) 93221000 Melanoma in situ of right lower limb (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 93213000 Malignant melanoma of skin of breast (disorder) 93213000 Malignant melanoma of skin of breast (disorder) 93213000 Malignant melanoma of skin of breast (disorder) 93213000 Malignant melanoma of skin of breast (disorder) 93213000 Malignant melanoma of skin of breast (disorder) 93213000 Malignant melanoma of skin of swill (disorder) 93213000 Malignant melanoma of skin of swill (disorder) 721563000 Primary malignant melanoma of scorea (disorder) 72265003 Primary malignant melanoma of skin of swill (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) 83736003 Malignant melanoma of skin of breatm (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) Malignant melanoma of skin of foretra (disorder) Malignant melanoma of skin of foretra (disorder) Malignant melanoma of skin of foretra (disorder) Malignant melanoma of skin of foretra (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of foretra (disorder) Malignant melanoma of skin of foretra (disorder) Malignant m | | |
| Malignant melanoma of auricle (ear) (disorder) 93654000 Malignant melanoma of skin of wrist (disorder) 93651008 Malignant melanoma of skin of trunk (disorder) 93649009 Malignant melanoma of skin of trunk (disorder) 93230002 Malignant melanoma of skin of trunk (disorder) 93230002 Malignant melanoma of skin of groin (disorder) 9324000 Malignant melanoma of skin of scalp (disorder) 9325000 Malignant melanoma of skin of scalp (disorder) 9322600 Malignant melanoma of unknown origin (disorder) 9322600 Malignant melanoma of skin of finger (disorder) 93224002 Malignant melanoma of skin of finger (disorder) 93224002 Malignant melanoma of skin of eyelid (disorder) 93224002 Malignant melanoma of skin of eyelid (disorder) 93221000 Melanoma in situ of right lower limb (disorder) 93221000 Melanoma in situ of skin of scalp (disorder) 932215000 Melanoma in situ of skin of scalp (disorder) 93215000 Melanoma in situ of skin of scalp (disorder) 93215000 Melanoma in situ of skin of scalp (disorder) 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 9321506 Malignant melanoma of skin of breast (disorder) 93215006 Malignant melanoma of skin of breast (disorder) 93215006 Malignant melanoma of skin of breast (disorder) 93215006 Malignant melanoma of skin of breast (disorder) 93215000 Primary malignant melanoma of skin of worth (disorder) 93216000 Primary malignant melanoma of skin of scalp (disorder) 93216000 Malignant melanoma of skin of scalp (disorder) 93216000 Malignant melanoma of skin of scalp (disorder) 93216000 Malignant melanoma of skin of breatm (disorder) 93216000 Malignant melanoma of skin of scalp (disorder) 93216000 Malignant melanoma of skin of scalp (disorder) 93216000 Malignant melanoma of skin of scalp (disorder) 93216000 Malignant melanoma of skin of scalp (disorder) 93216007 Malignant melanoma of skin of scalp (disorder) 93216007 Malignant melanoma of skin of scalp (disorder) 93216007 Malignant me | | |
| 93654000 Malignant melanoma of skin of wrist (disorder) 93651008 Malignant melanoma of skin of trunk (disorder) 93649009 Malignant melanoma of skin of trunk (disorder) 93230002 Malignant melanoma of skin of proin (disorder) 93230002 Malignant melanoma of skin of scalp (disorder) 93970507 Uveal melanoma TNM finding (finding) 403920004 Minimal deviation malignant melanoma (disorder) 424190005 Malignant melanoma of unknown origin (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 93226000 Malignant melanoma of skin of scalp (disorder) 93226000 Malignant melanoma of skin of spelid (disorder) 93226000 Malignant melanoma of skin of spelid (disorder) 93226000 Malignant melanoma of skin of spelid (disorder) 93226000 Malignant melanoma of skin of scalp (disorder) 932161000119100 Melanoma in situ of right lower limb (disorder) 932191000119107 Melanoma in situ of skin of scalp (disorder) 932190002 Superficial spreading melanoma (morphologic abnormality) 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of svalila (disorder) 93213004 Malignant melanoma of skin of svalila (disorder) 93213004 Malignant melanoma of skin of svalila (disorder) 93213004 Malignant melanoma of skin of svalila (disorder) 93213004 Malignant melanoma of skin of svalida (disorder) 93213004 Malignant melanoma of skin of svalida (disorder) 93213000 Primary malignant melanoma of skin (disorder) 93213000 Malignant melanoma of skin of breast (disorder) 93213000 Malignant melanoma of skin of svalida (disorder) 93213000 Malignant melanoma of skin of svalida (disorder) 93213000 Malignant melanoma of skin of svalida (morphologic abnormality) 9321300 Malignant melanoma of skin of svalida (morphologic abnormality) 9321300 Malignant melanoma of skin of svalida (morphologic abnormality) 9321300 Malignant melanoma of skin of svalida (morphologic abnormality) 9321300 Malignant melanoma of skin o | | |
| 93651008 Malignant melanoma of skin of trunk (disorder) 93649009 Malignant melanoma of skin of thigh (disorder) 93230002 Malignant melanoma of skin of groin (disorder) 93646002 Malignant melanoma of skin of scalp (disorder) 399705007 Uveal melanoma TNM finding (finding) 403920004 Minimal deviation malignant melanoma (disorder) 424190005 Malignant melanoma of unknown origin (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 115561000119102 History of malignant melanoma of eye (situation) 93224002 Malignant melanoma of skin of eyelid (disorder) 93221000 Melanoma in situ of right upper limb (disorder) 93221000 Melanoma in situ of right lower limb (disorder) 9322100019100 Melanoma in situ of skin of scalp (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 1092100019100 Malignant melanoma of skin of scalp (disorder) 10921000 Melanoma in situ of skin of scalp (disorder) 10921000 Malignant melanoma of skin of breast (disorder) 10921000 Malignant melanoma of skin of breast (disorder) 10921000 Malignant melanoma of skin of breast (disorder) 1092100 Primary malignant melanoma of vagina (disorder) 1092100 Primary malignant melanoma of vagina (disorder) 109265003 Primary malignant melanoma of skin (disorder) 109266008 Malignant melanoma of skin of skin (disorder) 109276751004 Amelanotic malignant melanoma of skin (disorder) 109276006 Multiple primary malignant melanoma (disorder) 109276006 Malignant melanoma of skin of buttock (disorder) 109283000 Malignant melanoma of skin of buttock (disorder) 109283000 Malignant melanoma of skin of buttock (disorder) 109267000 Malignant melanoma of skin of scrotum (disorder) 109267001 Malignant melanoma of skin of forearm (disorder) 109267002 Malignant melanoma of skin of forearm (disorder) 109267002 Malignant melanoma of skin of forearm (disorder) 109267002 Malignant melanoma of skin of forehead (disorder) 109267002 Malignant melanoma of skin of forehead (disorder) 109269007 Malignant melanoma of ski | | |
| 93649009 Malignant melanoma of skin of thigh (disorder) 93230002 Malignant melanoma of skin of groin (disorder) 93646002 Malignant melanoma of skin of groin (disorder) 399705007 Uveal melanoma TMM finding (finding) 403920004 Minimal deviation malignant melanoma (disorder) 424190005 Malignant melanoma of unknown origin (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 115561000119102 History of malignant melanoma of sey (situation) 93224002 Malignant melanoma of skin of eyel (disorder) 93221000 Melanoma in situ of right upper limb (disorder) 93221000 Melanoma in situ of right upper limb (disorder) 93211000119107 Melanoma in situ of skin of scalp (disorder) 93215000 Superficial spreading melanoma (morphologic abnormality) 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of floor of mouth (disorder) 93213000 Primary malignant melanoma of vagina (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 722665003 Primary malignant melanoma of skin (disorder) 72665004 Amelanotic malignant melanoma of skin (disorder) 72665005 Malignant melanoma of skin of scrotum (disorder) 72665001 Multiple primary malignant melanoma (disorder) 727671004 Amelanotic malignant melanoma of skin (disorder) 72873600 Malignant melanoma of skin of forearm (disorder) 72873700 Malignant melanoma of skin of buttock (disorder) 72873700 Malignant melanoma of skin of buttock (disorder) 72873700 Malignant melanoma of skin of forearm (disorder) 72873700 Malignant melanoma of skin of scrotum (disorder) 72873700 Malignant melanoma of skin of forearm (disorder) 72873700 Malignant melanoma o | | |
| 93230002 Malignant melanoma of skin of groin (disorder) 93646002 Malignant melanoma of skin of scalp (disorder) 399705007 Uveal melanoma TNM finding (finding) 403920004 Minimal deviation malignant melanoma (disorder) 424190005 Malignant melanoma of unknown origin (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 115561000119102 History of malignant melanoma of eye (situation) 93224002 Malignant melanoma of skin of eyelid (disorder) 93224002 Malignant melanoma of skin of eyelid (disorder) 932191000119100 Melanoma in situ of right upper limb (disorder) 932191000119107 Melanoma in situ of right upper limb (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 93213000 Primary malignant melanoma of cornea (disorder) 93215000 Primary malignant melanoma of oragina (disorder) 721563000 Primary malignant melanoma of cornea (disorder) 721665003 Primary malignant melanoma of skin of skin (disorder) Amelanotic malignant melanoma of skin (disorder) 402564006 Multiple primary malignant melanoma (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) 783736003 Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of foream (disorder) 188069004 Malignant melanoma of skin of foream (disorder) 188069004 Malignant melanoma of of skin of foream (disorder) 188069004 Malignant melanoma of of skin of foream (disorder) 188069004 Malignant melanoma of skin of foream (disorder) 188069004 Malignant melanoma of skin of foream (disorder) 188069004 Malignant melanoma of skin of foream (disorder) 188069004 Malignant melanoma of skin of foream (disorder) 188069004 Malignant melanoma of skin of foream (disorder) 19227907 Malignant melanoma of skin of forehead (disorder) 109267002 Overlapping malignant | | |
| Malignant melanoma of skin of scalp (disorder) 399705007 Uveal melanoma TMM finding (finding) 403920004 Minimal deviation malignant melanoma (disorder) 424190005 Malignant melanoma of unknown origin (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 115561000119102 History of malignant melanoma of skin of eyelid (disorder) 352161000119100 Melanoma in situ of right lower limb (disorder) 352191000119107 Melanoma in situ of right lower limb (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 109215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 408043002 Malignant melanoma of floor of mouth (disorder) 721563000 Primary malignant melanoma of vagina (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 722655003 Primary malignant melanoma of skin (disorder) Malignant melanoma of lacrimal gland (disorder) Multiple primary malignant melanoma (skin (disorder) Multiple primary malignant melanoma (skin (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of foream (disorder) Malignant melanoma of skin of foream (disorder) Malignant melanoma of skin of foream (disorder) Malignant melanoma of skin of foream (disorder) Malignant melanoma of skin of foream (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of foream (disorder) Malignant melanoma of skin of foream (disorder) Malignant melanoma of skin of foream (disorder) Malignant melanoma of skin of foream (disorder) Malignant melanoma of skin of foream (disorder) Malignant melanoma of skin of forehead (disorder) Malignant melanoma of orbit (disorder) Malignant melanoma of orbit (disorder) Malignant melanoma of skin of forehead (disorder) | | |
| Uveal melanoma TNM finding (finding) | | |
| Minimal deviation malignant melanoma (disorder) 424190005 Malignant melanoma of unknown origin (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 115561000119102 History of malignant melanoma of eye (situation) 93224002 Malignant melanoma of skin of eyelid (disorder) 352161000119100 Melanoma in situ of right upper limb (disorder) 352191000119107 Melanoma in situ of right lower limb (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 109210002 Superficial spreading melanoma (morphologic abnormality) 93215006 Malignant melanoma of skin of breast (disorder) 93215006 Malignant melanoma of skin of or a mouth (disorder) 109276009 Malignant melanoma of floor of mouth (disorder) 1092763000 Primary malignant melanoma of rornea (disorder) 109265003 Primary malignant melanoma of cornea (disorder) 109265003 Malignant melanoma of lacrimal gland (disorder) 109267004 Maleanotic malignant melanoma of skin (disorder) 1092674005 Malignant melanoma of mucous membrane (disorder) 10974005 Malignant melanoma of mucous membrane (disorder) 10974005 Malignant melanoma of skin of buttock (disorder) 109223008 Malignant melanoma of skin of scrotum (disorder) 109223008 Malignant melanoma of skin of forearm (disorder) 109223008 Malignant melanoma of skin of forearm (disorder) 109267002 Malignant melanoma of skin of forearm (disorder) 109267002 Malignant melanoma of skin of forearm (disorder) 109267002 Maligna | | |
| Malignant melanoma of unknown origin (disorder) 93226000 Malignant melanoma of skin of finger (disorder) 115561000119102 History of malignant melanoma of eyelid (disorder) 93224002 Malignant melanoma of skin of eyelid (disorder) 932161000119100 Melanoma in situ of right upper limb (disorder) 932191000119107 Melanoma in situ of skin of scalp (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 109275000 Superficial spreading melanoma (morphologic abnormality) 93213004 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 93213004 Malignant melanoma of floor of mouth (disorder) 721563000 Primary malignant melanoma of vagina (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 866079008 Malignant melanoma of lacrimal gland (disorder) 866079008 Malignant melanoma of lacrimal gland (disorder) Amelanotic malignant melanoma of skin (disorder) Acral lentiginous melanoma of skin (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) 783736003 Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of of syncology and Obstetrics stage finding for vulvar melanoma of skin (disorder) Malignant melanoma of orbit (disorder) Malignant melanoma of orbit (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of skin | | |
| Malignant melanoma of skin of finger (disorder) 115561000119102 History of malignant melanoma of eye (situation) 93224002 Malignant melanoma of skin of eyelid (disorder) 352161000119100 Melanoma in situ of right upper limb (disorder) 352191000119107 Melanoma in situ of right lower limb (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 109275000 Malignant melanoma of skin of breast (disorder) 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 93213000 Primary malignant melanoma of vagina (disorder) 721563000 Primary malignant melanoma of vagina (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 866079008 Malignant melanoma of lacrimal gland (disorder) 866079008 Malignant melanoma of skin (disorder) 402564006 Multiple primary malignant melanomata (disorder) 402564006 Multiple primary malignant melanoma (disorder) 402564006 Malignant melanoma of mucous membrane (disorder) 402564006 Malignant melanoma of skin of buttock (disorder) 402564006 Malignant melanoma of skin of buttock (disorder) 402564006 Malignant melanoma of skin of prearm (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564006 Malignant melanoma of skin of forearm (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564007 Malignant melanoma of skin of scrotum (disorder) 402564008 Malignant melanoma of skin of scrotum (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564006 Mali | | |
| History of malignant melanoma of eye (situation) 93224002 Malignant melanoma of skin of eyelid (disorder) 352161000119100 Melanoma in situ of right upper limb (disorder) 352191000119107 Melanoma in situ of right lower limb (disorder) 352191000119107 Melanoma in situ of skin of scalp (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 55320002 Superficial spreading melanoma (morphologic abnormality) 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 698043002 Malignant melanoma of floor of mouth (disorder) 721563000 Primary malignant melanoma of vagina (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 866079008 Malignant melanoma of lacrimal gland (disorder) 402564006 Multiple primary malignant melanoma of skin (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) Malignant melanoma of mucous membrane (disorder) 448273006 Malignant melanoma of skin of buttock (disorder) 448273006 Malignant melanoma of skin of scrotum (disorder) 93223008 Malignant melanoma of skin of scrotum (disorder) 188069004 Malignant melanoma of skin of | | |
| Malignant melanoma of skin of eyelid (disorder) 352161000119100 Melanoma in situ of right upper limb (disorder) 352191000119107 Melanoma in situ of right lower limb (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 55320002 Superficial spreading melanoma (morphologic abnormality) 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 698043002 Malignant melanoma of floor of mouth (disorder) 698043002 Primary malignant melanoma of vagina (disorder) 721563000 Primary malignant melanoma of vagina (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 866079008 Malignant melanoma of lacrimal gland (disorder) 402564006 Multiple primary malignant melanoma of skin (disorder) 402564006 Multiple primary malignant melanomata (disorder) 402564006 Multiple primary malignant melanomata (disorder) 402564006 Multiple primary malignant melanomata (disorder) 402564006 Malignant melanoma of mucous membrane (disorder) 402564006 Malignant melanoma of skin of buttock (disorder) 402564006 Malignant melanoma of skin of buttock (disorder) 402564006 Malignant melanoma of skin of forearm (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564006 Malignant melanoma of skin of scrotum (disorder) 402564006 Malignant melanoma of skin of forearm (disorder) 402564006 Malignant melanoma of skin of forearm (disorder) 402564007 Malignant melanoma of skin of forearm (disorder) 402564009 Malignant melanoma of skin of forearm (disorder) 402564000 Malignant melanoma of skin of forearm (disorder) 402564000 Malignant melanoma of skin of forearm (disorder) 402564000 Malignant melanoma of skin of forearm (disorder) 402564000 Malignant melanoma of skin of forearm (disorder) 402564000 Malignant melanoma of skin of forehead (disorder) 402564000 Malignant melanoma of skin of forehead (disorder) 402564000 Malignant melanoma of skin of forehead (disorder) 402564000 Malignant melanoma of skin of forehead (disorder) | | |
| 352161000119100 Melanoma in situ of right upper limb (disorder) 352191000119107 Melanoma in situ of right lower limb (disorder) 109276009 Melanoma in situ of skin of scalp (disorder) 55320002 Superficial spreading melanoma (morphologic abnormality) 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 698043002 Malignant melanoma of floor of mouth (disorder) 721563000 Primary malignant melanoma of vagina (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 72665003 Primary malignant melanoma of skin (disorder) 866079008 Malignant melanoma of lacrimal gland (disorder) 876751004 Amelanotic malignant melanoma of skin (disorder) 876751004 Amelanotic malignant melanoma of skin (disorder) 8776751004 Amelanotic malignant melanoma of skin (disorder) 878736003 Malignant melanoma of mucous membrane (disorder) 8783736003 Malignant melanoma of skin of buttock (disorder) 8783736003 Malignant melanoma of skin of buttock (disorder) 878373006 Malignant melanoma of skin of scrotum (disorder) 8793223008 Malignant melanoma of skin of eyebrow (disorder) 8793228004 Malignant melanoma of skin of eyebrow (disorder) 8793228004 Malignant melanoma of thigh (disorder) 8793228004 Malignant melanoma of thigh (disorder) 8793228004 Malignant melanoma of thigh (disorder) 8793228004 Malignant melanoma of skin of forearm (disorder) 8793228004 Malignant melanoma of skin of scrotum (disorder) 8793228004 Malignant melanoma of skin of scrotum (disorder) 8793228004 Malignant melanoma of skin of scrotum (disorder) 8793228004 Malignant melanoma of skin of scrotum (disorder) 8793228004 Malignant melanoma of skin of forehead (disorder) 8793228007 Malignant melanoma of skin of forehead (disorder) | | |
| Melanoma in situ of right lower limb (disorder) | | |
| Melanoma in situ of skin of scalp (disorder) Superficial spreading melanoma (morphologic abnormality) Malignant melanoma of skin of breast (disorder) Malignant melanoma of skin of axilla (disorder) Malignant melanoma of skin of axilla (disorder) Malignant melanoma of skin of axilla (disorder) Malignant melanoma of floor of mouth (disorder) Primary malignant melanoma of vagina (disorder) Primary malignant melanoma of cornea (disorder) Malignant melanoma of lacrimal gland (disorder) Malignant melanoma of lacrimal gland (disorder) Multiple primary malignant melanoma of skin (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) Malignant melanoma of mucous membrane (disorder) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of bottock (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of of opechology and Obstetrics stage finding for vulvar melanoma of skin (disorder) Malignant melanoma of orbit (disorder) Malignant melanoma of orbit (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | |
| Superficial spreading melanoma (morphologic abnormality) 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 698043002 Malignant melanoma of floor of mouth (disorder) 721563000 Primary malignant melanoma of vagina (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 866079008 Malignant melanoma of lacrimal gland (disorder) 276751004 Amelanotic malignant melanoma of skin (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) 783736003 Malignant melanoma of mucous membrane (disorder) 93216007 Malignant melanoma of skin of buttock (disorder) 93223008 Malignant melanoma of skin of scrotum (disorder) 93228004 Malignant melanoma of skin of forearm (disorder) 188069004 Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | |
| 93215006 Malignant melanoma of skin of breast (disorder) 93213004 Malignant melanoma of skin of axilla (disorder) 698043002 Malignant melanoma of floor of mouth (disorder) 721563000 Primary malignant melanoma of vagina (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 866079008 Malignant melanoma of lacrimal gland (disorder) 276751004 Amelanotic malignant melanoma of skin (disorder) 402564006 Multiple primary malignant melanomata (disorder) 402564006 Acral lentiginous melanoma, malignant (morphologic abnormality) 783736003 Malignant melanoma of mucous membrane (disorder) 93216007 Malignant melanoma of skin of buttock (disorder) 448273006 Malignant melanoma of skin of scrotum (disorder) 93223008 Malignant melanoma of skin of eyebrow (disorder) 93223004 Malignant melanoma of skin of forearm (disorder) 188069004 Malignant melanoma of thigh (disorder) 186072004 Malignant melanoma of thigh (disorder) 109267002 Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) 7 Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) 7 Tumor-node-metastasis (TNM) malignant melanoma of iris | 109276009 | Melanoma in situ of skin of scalp (disorder) |
| 93213004Malignant melanoma of skin of axilla (disorder)698043002Malignant melanoma of floor of mouth (disorder)721563000Primary malignant melanoma of vagina (disorder)722665003Primary malignant melanoma of cornea (disorder)866079008Malignant melanoma of lacrimal gland (disorder)276751004Amelanotic malignant melanoma of skin (disorder)402564006Multiple primary malignant melanomata (disorder)402564006Multiple primary malignant melanomata (disorder)46974005Acral lentiginous melanoma, malignant (morphologic abnormality)783736003Malignant melanoma of mucous membrane (disorder)93216007Malignant melanoma of skin of buttock (disorder)93223008Malignant melanoma of skin of scrotum (disorder)93223008Malignant melanoma of skin of forearm (disorder)93228004Malignant melanoma of thigh (disorder)188069004Malignant melanoma of thigh (disorder)1nternational Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding)866072004Malignant melanoma of orbit (disorder)109267002Overlapping malignant melanoma of skin (disorder)915007Malignant melanoma in junctional nevus (morphologic abnormality)109267002Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging)93229007Malignant melanoma of skin of forehead (disorder)109267002Tumor-node-metastasis (TNM) malignant melanoma of iris | 55320002 | Superficial spreading melanoma (morphologic abnormality) |
| Malignant melanoma of floor of mouth (disorder) 721563000 Primary malignant melanoma of vagina (disorder) 722665003 Primary malignant melanoma of cornea (disorder) 866079008 Malignant melanoma of lacrimal gland (disorder) 276751004 Amelanotic malignant melanoma of skin (disorder) 402564006 Multiple primary malignant melanomata (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) 783736003 Malignant melanoma of mucous membrane (disorder) 93216007 Malignant melanoma of skin of buttock (disorder) 448273006 Malignant melanoma of skin of scrotum (disorder) 93223008 Malignant melanoma of skin of eyebrow (disorder) 188069004 Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma of skin (disorder) 109267002 Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 93215006 | Malignant melanoma of skin of breast (disorder) |
| Primary malignant melanoma of vagina (disorder) Primary malignant melanoma of cornea (disorder) Malignant melanoma of lacrimal gland (disorder) Malignant melanoma of lacrimal gland (disorder) Amelanotic malignant melanoma of skin (disorder) Multiple primary malignant melanomata (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) Malignant melanoma of mucous membrane (disorder) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of eyebrow (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma of skin (disorder) Malignant melanoma of orbit (disorder) Malignant melanoma of orbit (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) Malignant melanoma of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 93213004 | Malignant melanoma of skin of axilla (disorder) |
| Primary malignant melanoma of cornea (disorder) Malignant melanoma of lacrimal gland (disorder) Amelanotic malignant melanoma of skin (disorder) Multiple primary malignant melanomata (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) Malignant melanoma of mucous membrane (disorder) Malignant melanoma of mucous membrane (disorder) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) Malignant melanoma of orbit (disorder) Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 698043002 | Malignant melanoma of floor of mouth (disorder) |
| Malignant melanoma of lacrimal gland (disorder) Amelanotic malignant melanoma of skin (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of eyebrow (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) Malignant melanoma of orbit (disorder) Malignant melanoma of orbit (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 721563000 | Primary malignant melanoma of vagina (disorder) |
| Amelanotic malignant melanoma of skin (disorder) 402564006 | 722665003 | Primary malignant melanoma of cornea (disorder) |
| Multiple primary malignant melanomata (disorder) Acral lentiginous melanoma, malignant (morphologic abnormality) 783736003 Malignant melanoma of mucous membrane (disorder) 93216007 Malignant melanoma of skin of buttock (disorder) 448273006 Malignant melanoma of skin of scrotum (disorder) 93223008 Malignant melanoma of skin of eyebrow (disorder) 93228004 Malignant melanoma of skin of forearm (disorder) 188069004 Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) 866072004 Malignant melanoma of orbit (disorder) 109267002 Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 866079008 | Malignant melanoma of lacrimal gland (disorder) |
| Acral lentiginous melanoma, malignant (morphologic abnormality) 783736003 Malignant melanoma of mucous membrane (disorder) 93216007 Malignant melanoma of skin of buttock (disorder) 448273006 Malignant melanoma of skin of scrotum (disorder) 93223008 Malignant melanoma of skin of eyebrow (disorder) 93228004 Malignant melanoma of skin of forearm (disorder) 188069004 Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) 866072004 Malignant melanoma of orbit (disorder) 109267002 Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 276751004 | Amelanotic malignant melanoma of skin (disorder) |
| abnormality) 783736003 Malignant melanoma of mucous membrane (disorder) 93216007 Malignant melanoma of skin of buttock (disorder) 448273006 Malignant melanoma of skin of scrotum (disorder) 93223008 Malignant melanoma of skin of eyebrow (disorder) 93228004 Malignant melanoma of skin of forearm (disorder) 188069004 Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) 866072004 Malignant melanoma of orbit (disorder) 109267002 Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 402564006 | Multiple primary malignant melanomata (disorder) |
| Malignant melanoma of mucous membrane (disorder) Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of eyebrow (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) Malignant melanoma of orbit (disorder) Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | |
| Malignant melanoma of skin of buttock (disorder) Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of eyebrow (disorder) Malignant melanoma of skin of eyebrow (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) Malignant melanoma of orbit (disorder) Malignant melanoma of orbit (disorder) Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | |
| Malignant melanoma of skin of scrotum (disorder) Malignant melanoma of skin of eyebrow (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of skin of forearm (disorder) Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) Malignant melanoma of orbit (disorder) Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | |
| 93223008 Malignant melanoma of skin of eyebrow (disorder) 93228004 Malignant melanoma of skin of forearm (disorder) 188069004 Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) 866072004 Malignant melanoma of orbit (disorder) 109267002 Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | |
| 93228004 Malignant melanoma of skin of forearm (disorder) 188069004 Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) 866072004 Malignant melanoma of orbit (disorder) 109267002 Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | |
| 188069004 Malignant melanoma of thigh (disorder) International Federation of Gynecology and Obstetrics stage finding for vulvar melanoma (finding) 866072004 Malignant melanoma of orbit (disorder) 109267002 Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | |
| International Federation of Gynecology and Obstetrics stage 385372004 finding for vulvar melanoma (finding) 866072004 Malignant melanoma of orbit (disorder) 109267002 Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) 109267002 Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 93228004 | |
| finding for vulvar melanoma (finding) Malignant melanoma of orbit (disorder) Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 188069004 | |
| Malignant melanoma of orbit (disorder) Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | , |
| Overlapping malignant melanoma of skin (disorder) Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 385372004 | 1 2 |
| Malignant melanoma in junctional nevus (morphologic abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 866072004 | |
| 915007 abnormality) Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 109267002 | |
| Tumor-node-metastasis (TNM) malignant melanoma of skin staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | |
| 254325002 staging (tumor staging) 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | 915007 | - · |
| 93229007 Malignant melanoma of skin of forehead (disorder) Tumor-node-metastasis (TNM) malignant melanoma of iris | | , , , |
| Tumor-node-metastasis (TNM) malignant melanoma of iris | 254325002 | |
| | 93229007 | |
| 254347002 staging (tumor staging) | | Tumor-node-metastasis (TNM) malignant melanoma of iris |
| | 254347002 | staging (tumor staging) |

| 9364004 | Malignant melanoma of skin of perineum (disorder) |
|------------------|----------------------------------------------------------|
| 188044004 | Malignant melanoma of scalp and/or neck (disorder) |
| 93652001 | Malignant melanoma of skin of umbilicus (disorder) |
| 449636007 | Malignant melanoma of skin of lower leg (disorder) |
| 449637003 | Malignant melanoma of skin of upper arm (disorder) |
| 424487008 | Malignant melanoma of skin of upper lip (disorder) |
| 424302003 | Malignant melanoma of skin of lower lip (disorder) |
| 12.00200 | Malignant melanoma in junctional nevus (morphologic |
| 915007 | abnormality) |
| 956451000000107 | Malignant melanoma stage IIIB (finding) |
| 351961000119109 | Malignant melanoma of skin of right arm (disorder) |
| 399660006 | Ring melanoma of ciliary body (disorder) |
| | Tumor-node-metastasis (TNM) malignant melanoma of |
| 254343003 | eyelid staging (tumor staging) |
| 698041000 | Malignant melanoma of vestibule of mouth (disorder) |
| 722543005 | Primary malignant melanoma of anal canal (disorder) |
| 402556000 | Malignant melanoma (radial growth phase) (disorder) |
| | Tumor-node-metastasis (TNM) malignant melanoma of |
| 254349004 | choroid staging (tumor staging) |
| 188071004 | Malignant melanoma of popliteal fossa area (disorder) |
| 423447006 | Malignant melanoma of skin of lower eyelid |
| 423494003 | Malignant melanoma of skin of upper eyelid (disorder) |
| | Psoralen and long-wave ultraviolet radiation therapy- |
| 403714009 | associated malignant melanoma (disorder) |
| 314987003 | Metastasis from malignant melanoma of skin (disorder) |
| 402558004 | Malignant melanoma (vertical growth phase) (disorder) |
| 103419001 | Clark's melanoma level (observable entity) |
| | Malignant melanoma of giant pigmented nevus |
| 75931002 | (morphologic abnormality) |
| | Mixed epithelioid and spindle cell melanoma (morphologic |
| 50813003 | abnormality) |
| 109280004 | Melanoma in situ of external auditory canal (disorder |
| 399521000 | Necrotic melanoma (morphologic abnormality) |
| | Malignant melanoma with B-Raf proto-oncogene, |
| | serine/threonine kinase V600E mutation (morphologic |
| 830195005 | abnormality) |
| | Malignant melanoma with B-Raf proto-oncogene, |
| 830150003 | serine/threonine kinase V600E mutation (disorder) |
| 402560002 | Materno-fetal metastatic malignant melanoma |
| | Malignant melanoma in precancerous melanosis |
| 18450009 | (morphologic abnormality) |
| 423280002 | Malignant melanoma of skin of canthus of eye (disorder) |
| 109288006 | Melanoma in situ of perianal skin (disorder) |
| 402557009 | In situ acral lentiginous malignant melanoma (disorder) |
| 109286005 | Melanoma in situ of skin of breast (disorder) |
| 352201000119105 | Malignant melanoma of skin of left upper limb (disorder) |
| 396369000 | pTis: Melanoma in situ (melanoma of the skin) (finding) |
| 1081021000119100 | Malignant melanoma of skin of left lower limb (disorder) |
| 93648001 | Malignant melanoma of skin of temporal region (disorder) |
| 109274007 | Melanoma in situ of eyelid, including canthus (disorder) |

| 188034001 | Malignant melanoma of external auditory meatus (disorder) |
|---|---|
| 352001000119100 | Malignant melanoma of skin of right lower limb (disorder) |
| 254734009 | Malignant melanoma arising in congenital nevus (disorder) |
| 866082003 | Malignant melanoma of lacrimal drainage system (disorder) |
| 314976006 | Local recurrence of malignant melanoma of skin (disorder) |
| 396391007 | pM1b: Metastasis to lung (melanoma of the skin) (finding) |
| 0000000 | Distance of malignant melanoma from deep margin |
| 396518001 | (observable entity) |
| 33333333 | Malignant melanoma arising in intradermal nevus |
| 254733003 | (disorder) |
| | Malignant melanoma of trunk (excluding scrotum) |
| 188048001 | (navigational concept) |
| 93210001 | Malignant melanoma of skin of abdomen (disorder) |
| 402564006 | Multiple primary malignant melanomata (disorder) |
| 115561000119102 | History of malignant melanoma of eye (situation) |
| 93647006 | Malignant melanoma of skin of shoulder (disorder) |
| 95047000 | Malignant melanoma in Hutchinson's melanotic freckle |
| 44474009 | (morphologic abnormality) |
| 44474009 | , |
| 75931002 | Malignant melanoma in giant pigmented nevus |
| 75951002 | (morphologic abnormality) |
| 200517000 | Surgical deep margin involved by malignant melanoma |
| 396517006 | (finding) |
| 200400002 | Surgical lateral margin involved by in situ melanoma |
| 396400002 | (finding) |
| 399634005 | Choroidal melanoma, diffuse (morphologic abnormality) |
| 200540002 | Surgical deep margin uninvolved by malignant melanoma |
| 396516002 | (finding) |
| 206200000 | Surgical lateral margin uninvolved by in situ melanoma |
| 396399009 | (finding) |
| 200501001 | pT1: Tumor limited to the iris (iris) (uveal melanoma) |
| 399501001 | (finding) |
| 200512005 | Surgical lateral margin involved by malignant melanoma |
| 396513005 | (finding) |
| 402274000 | Hypomelanosis surrounding malignant melanoma |
| 403274000 | (disorder) Surgical lateral margin uninvolved by malignant melanoma |
| 396512000 | , , |
| 390312000 | (finding) |
| 20806000 | Malignant melanoma, regressing (morphologic |
| 39896009 | abnormality) |
| 206511007 | Distance of in situ melanoma from closest lateral margin |
| 396511007 | (observable entity) |
| 396391007 | pM1b: Metastasis to lung (melanoma of the skin) (finding) |
| 403563000 | Metastatic malignant melanoma with diffuse |
| 402563000 | hypermelanosis (disorder) |
| 000073000 | Malignant melanoma of overlapping lesion of eye and |
| 866073009 | adnexa (disorder) |
| 200545002 | Distance of malignant melanoma from closest lateral |
| 396515003 | margin (observable entity) |
| 200670000 | pT4: Tumor with extraocular extension (iris) (uveal |
| 399679009 | melanoma) (finding) |

| | Surgical deep margin involved by malignant melanoma |
|-------------|------------------------------------------------------------|
| 396517006 | (finding) |
| 330317000 | Surgical lateral margin involved by in situ melanoma |
| 396400002 | (finding) |
| 330100002 | Tumor-node-metastasis (TNM) malignant melanoma of |
| 254346006 | uvea staging (tumor staging) |
| 23 13 10000 | Surgical deep margin involvement by melanoma cannot be |
| 399717009 | assessed (finding) |
| 333717003 | pN1: Metastasis in one regional lymph node (melanoma of |
| 396382008 | the skin) (finding) |
| 189324006 | Melanoma in situ of skin of scalp and/or neck (disorder) |
| 103324000 | Surgical lateral margin involvement by melanoma cannot be |
| 399385006 | assessed (finding) |
| 333383000 | Malignant melanoma of ear and/or external auditory canal |
| 188032002 | (disorder) |
| 188032002 | Metastatic malignant melanoma with diffuse |
| 402563000 | hypermelanosis (disorder) |
| 402303000 | Location of malignant melanoma in specimen with involved |
| 425133002 | deep margin (observable entity) |
| 423133002 | Tumor-node-metastasis (TNM) malignant melanoma of |
| 254345005 | conjunctiva staging (tumor staging) |
| 234343003 | Location of melanoma in situ in specimen with involved |
| 424082007 | lateral margin (observable entity) |
| 424082007 | Tumor-node-metastasis (TNM) malignant melanoma of |
| 254348007 | ciliary body staging (tumor staging) |
| 234348007 | Location of malignant melanoma in specimen with |
| 424949006 | uninvolved deep margin (observable entity) |
| 424343000 | Malignant melanoma in precancerous melanosis |
| 18450009 | (morphologic abnormality) |
| 10430003 | pN2a: Clinically occult (microscopic) metastasis (melanoma |
| 396386006 | of the skin) (finding) |
| 33030000 | pN1a: Clinically occult (microscopic) metastasis (melanoma |
| 396383003 | of the skin) (finding) |
| 33030300 | pT4: Tumor with extraocular extension (iris) (uveal |
| 399679009 | melanoma) (finding) |
| | Surgical deep margin involvement by melanoma cannot be |
| 399717009 | assessed (finding) |
| | pN1b: Clinically apparent (macroscopic) metastasis |
| 396384009 | (melanoma of the skin) (finding) |
| | pN2b: Clinically apparent (macroscopic) metastasis |
| 396387002 | (melanoma of the skin) (finding) |
| | College of American Pathologists Cancer Checklist; Uveal |
| 406039001 | Melanoma: Resection (record artifact) |
| | International Federation of Gynecology and Obstetrics |
| 70046009 | vulvar melanoma stage I (finding) |
| | International Federation of Gynecology and Obstetrics |
| 73055006 | vulvar melanoma stage V (finding) |
| | International Federation of Gynecology and Obstetrics |
| 65306007 | vulvar melanoma stage II (finding) |
| | International Federation of Gynecology and Obstetrics |
| 80588003 | vulvar melanoma stage IV (finding) |

| CEE2CO04 | International Federation of Gynecology and Obstetrics |
|---|---|
| 65536004 | vulvar melanoma stage III (finding) |
| 206277001 | pT3a: Melanoma 2.01 to 4.0 mm in thickness, no ulceration |
| 396377001 | (melanoma of the skin) (finding) |
| 200274000 | pT2a: Melanoma 1.01 to 2.0 mm in thickness, no ulceration |
| 396374008 | (melanoma of the skin) (finding) |
| 206206006 | pN2a: Clinically occult (microscopic) metastasis (melanoma |
| 396386006 | of the skin) (finding) |
| 200202002 | pN1a: Clinically occult (microscopic) metastasis (melanoma |
| 396383003 | of the skin) (finding) |
| 206270006 | pT3b: Melanoma 2.01 to 4.0 mm in thickness, with |
| 396378006 | ulceration (melanoma of the skin) (finding) |
| 206275000 | pT2b: Melanoma 1.01 to 2.0 mm in thickness, with |
| 396375009 | ulceration (melanoma of the skin) (finding) |
| 200602001 | pT1c: Tumor limited to the iris with melanomalytic |
| 399602001 | glaucoma (iris) (uveal melanoma) (finding) |
| 206297002 | pN2b: Clinically apparent (macroscopic) metastasis |
| 396387002 | (melanoma of the skin) (finding) |
| 20.620.4000 | pN1b: Clinically apparent (macroscopic) metastasis |
| 396384009 | (melanoma of the skin) (finding) |
| 200602004 | pT1c: Tumor limited to the iris with melanomalytic |
| 399602001 | glaucoma (iris) (uveal melanoma) (finding) |
| 20.5200000 | pT4a: Melanoma greater than 4.0 mm in thickness, no |
| 396380000 | ulceration (melanoma of the skin) (finding) |
| 206204004 | pT4b: Melanoma greater than 4.0 mm in thickness, with |
| 396381001 | ulceration (melanoma of the skin) (finding) |
| 206200007 | pN2c: Satellite or in-transit metastasis without nodal |
| 396388007 | metastasis (melanoma of the skin) (finding) |
| 200511000 | pT1b: Tumor limited to the iris (more than 3 clock hours in |
| 399511008 | size) (iris) (uveal melanoma) (finding) |
| 422706005 | Location of melanoma in situ in specimen with uninvolved |
| 422796005 | lateral margin (observable entity) |
| 206272002 | pT2: Melanoma 1.01 to 2.0 mm in thickness, with or |
| 396373002 | without ulceration (melanoma of the skin) (finding) |
| 200270005 | pT3: Melanoma 2.01 to 4.0 mm in thickness, with or |
| 396376005 | without ulceration (melanoma of the skin) (finding) pT1: Melanoma 1.0 mm or less in thickness, with or without |
| 396370004 | ulceration (melanoma of the skin) (finding) |
| 390370004 | |
| 206200000 | pM1a: Metastasis to skin, subcutaneous tissues, or distant |
| 396390008 | lymph nodes (melanoma of the skin) (finding |
| 200507000 | pT1a: Tumor limited to the iris (not more than 3 clock hours in size) (iris) (uvoal malanema) (finding) |
| 399597008 | in size) (iris) (uveal melanoma) (finding) |
| 406058005 | College of American Pathologists Cancer Checklist; |
| +00030003 | Melanoma of the Skin: Excision; Re-Excision (record artifact) pT4: Melanoma greater than 4.0 mm in thickness, with or |
| 396379003 | |
| 330373003 | without ulceration (melanoma of the skin) (finding) |
| 206291001 | pT4b: Melanoma greater than 4.0 mm in thickness, with |
| 396381001 | ulceration (melanoma of the skin) (finding) |
| 200615005 | pT2: Tumor confluent with or extending into the ciliary body |
| 399615005 | and/or choroid (iris) (uveal melanoma) (finding) |

| | .T4. Mala |
|---|---|
| 206274000 | pT1a: Melanoma 1.0 mm or less in thickness and level II or |
| 396371000 | III, no ulceration (melanoma of the skin) (finding |
| 200645005 | pT2: Tumor confluent with or extending into the ciliary body |
| 399615005 | and/or choroid (iris) (uveal melanoma) (finding) |
| 20.627.6005 | pT3: Melanoma 2.01 to 4.0 mm in thickness, with or |
| 396376005 | without ulceration (melanoma of the skin) (finding) |
| 206272007 | pT1b: Melanoma 1.0 mm or less in thickness and level IV or |
| 396372007 | V or with ulceration (melanoma of the skin) (finding) |
| | pT1: Tumor 2 cm or less in greatest dimension (carcinoma |
| 396493009 | of skin excluding eyelid, vulva, penis, and melanomas) |
| 390493009 | (finding) |
| | pT3: Tumor more than 5 cm in greatest dimension |
| 396501000 | (carcinoma of skin excluding eyelid, vulva, penis, and |
| 390301000 | melanomas) (finding) |
| | pT3: Tumor confluent with or extending into the ciliary body |
| 200557005 | and/or choroid with scleral extension (iris) (uveal |
| 399557005 | melanoma) (finding) pT3: Tumor more than 5 cm in greatest dimension |
| | (carcinoma of skin excluding eyelid, vulva, penis, and |
| 396501000 | melanomas) (finding) |
| 390301000 | , , <u>u</u> , |
| | pN2: Metastasis in 2 to 3 regional nodes or intralymphatic regional metastasis without nodal metastasis (melanoma of |
| 396385005 | the skin) (finding) |
| 330363003 | pT1: Tumor 10 mm or less in greatest diameter and 2.5 mm |
| | or less in greatest height (thickness) (ciliary body and |
| 399448002 | choroid) (uveal melanoma) (finding) |
| 333440002 | pM1c: Metastasis to visceral site other than lung or distant |
| | metastasis at any site associated with an elevated serum |
| 396392000 | lactic dehydrogenase (melanoma of the skin) (finding) |
| 330332000 | pT4: Tumor invades deep extradermal structures (i.e. |
| | cartilage, skeletal muscle, or bone) (carcinoma of skin |
| 396506005 | excluding eyelid, vulva, penis, and melanomas) (finding) |
| 33030000 | pT3a: Tumor more than 5 cm in greatest dimension, limited |
| | to dermis or not more than 2 mm in thickness (carcinoma |
| | of skin excluding eyelid, vulva, penis, and melanomas) |
| 396502007 | (finding) |
| | pT1c: Tumor 2 cm or less in greatest dimension, invading the |
| | subcutis and/or greater than 6 mm in thickness (carcinoma |
| | of skin excluding eyelid, vulva, penis, and melanomas) |
| 396496001 | (finding) |
| | pT4: Tumor more than 16 mm in greatest diameter and/or |
| | greater than 10 mm in maximum height (thickness) with |
| | extraocular extension (ciliary body and choroid) (uveal |
| 399729000 | melanoma) (finding) |
| | pN3: Metastasis in four or more regional nodes, or matted |
| | metastatic nodes, or in-transit metastasis or satellite(s) with |
| | metastasis in regional node(s) (melanoma of the skin) |
| 396389004 | (finding) |
| | pT3c: Tumor more than 5 cm in greatest dimension, |
| | invading the subcutis and/or greater than 6 mm in thickness |
| | (carcinoma of skin excluding eyelid, vulva, penis, and |
| 396504008 | melanomas) (finding) |

| | | nT2. Tumor more than 16 mm in greatest diameter and/or |
|---|---|---|
| | | pT3: Tumor more than 16 mm in greatest diameter and/or |
| | | greater than 10 mm in maximum height (thickness) without |
| 200610000 | | extraocular extension (ciliary body and choroid) (uveal |
| 399610000 | | melanoma) (finding) |
| | | pT1c: Tumor 10 mm or less in greatest diameter and 2.5 mm |
| | | or less in greatest height (thickness) with macroscopic |
| 399493005 | | extraocular extension (ciliary body and choroid) (uveal melanoma) (finding) |
| 399493003 | | pT1b: Tumor 10 mm or less in greatest diameter and 2.5 mm |
| | | or less in greatest height (thickness) with microscopic |
| | | extraocular extension (ciliary body and choroid) (uveal |
| 399461002 | | melanoma) (finding) |
| 333401002 | | pT1a: Tumor 10 mm or less in greatest diameter and 2.5 mm |
| | | or less in greatest height (thickness) without microscopic |
| | | extraocular extension (ciliary body and choroid) (uveal |
| 399516003 | | melanoma) (finding) |
| | | pT4b: Tumor invades deep extradermal structures (i.e. |
| | | cartilage, skeletal muscle, or bone) greater than 6mm in |
| | | thickness (carcinoma of skin excluding eyelid, vulva, penis, |
| 396507001 | | and melanomas) (finding) |
| | | pT4a: Tumor invades deep extradermal structures (i.e. |
| | | cartilage, skeletal muscle, or bone) not more than 6mm in |
| | | thickness (carcinoma of skin excluding eyelid, vulva, penis, |
| 396508006 | | and melanomas) (finding) |
| | | pT2b: Tumor 10 mm to 16 mm in greatest basal diameter |
| | | and between 2.5 and 10 mm in maximum height (thickness) |
| | | with microscopic extraocular extension (ciliary body and |
| 399616006 | | choroid) (uveal melanoma) (finding) |
| | | pT2c: Tumor 10 mm to 16 mm in greatest basal diameter |
| | | and between 2.5 and 10 mm in maximum height (thickness) |
| 399543008 | | with macroscopic extraocular extension (ciliary body and choroid) (uveal melanoma) (finding) |
| 399343006 | | pT2a: Tumor more than 2 cm, but not more than 5 cm, in |
| | | greatest dimension, limited to dermis or greater than 2 mm |
| | | in thickness (carcinoma of skin excluding eyelid, vulva, |
| 396498000 | | penis, and melanomas) (finding) |
| Nonmelanoma skin c | ancers | |
| | Term | |
| Read V2 Code | ID | Description |
| B338. | All | Squamous cell carcinoma of skin |
| B33z. | All | Squamous cell carcinoma of skin NOS |
| BB24. | All | [M] Verrucous carcinoma NOS |
| B8 | All | Bowen's disease |
| BB2L. | All | [M] Bowen's disease |
| BB3 | All | Basal cell neoplasms |
| BB30. | All | [M]Basal cell tumour |
| BB31. | All | [M]Basal cell carcinoma NOS |
| Bb32. | All | [M]Multicentric basal cell carcinoma |
| BB33. | All | [M]Basal cell carcinoma, morhoea type |
| BB34. | All | [M]Basal cell carcinoma, fibroepithelial type |
| BB35. | All | [M]Basosquamous carcinoma |

| BB36. | All | [M]Metatypical carcinoma |
|---|---|---|
| BB37. | All | [M]Intraepidermal epithelioma of Jadassohn |
| BB3C. | All | [M]Superficial basal cell carcinoma |
| BB3D. | All | [M]Basal cell carcinoma, nodular |
| BB3E. | All | [M]Basal cell carcinoma, micronodular |
| BB3F. | All | [M]Basal cell carcinoma, infiltrative |
| BB3G. | All | [M]Pigmented basal cell carcinoma |
| BB3z. | All | [M]Basal cell neoplasm NOS |
| BB5y0 | All | [M]Basal cell adenocarcinoma |
| 7G05D | All | Excision biopsy of basal cell carcinoma |
| B33z0 | All | Kaposi sarcoma of the skin |
| BB5RA | All | [M]Merkel cell carcinoma |
| B621. | All | Mycosis fungoides |
| B6210 | All | Mycosis fungoides of unspecified site |
| B6211 | All | Mycosis fungoides of lymph nodes of head, face and neck |
| B6212 | All | Mycosis fungoides of intrathoracic lymph nodes |
| B6213 | All | Mycosis fungoides of intractionate lymph nodes |
| B6214 | All | Mycosis fungoides of lymph nodes of axilla and upper limb |
| B6215 | All | Mycosis fungoides of lymph nodes of inguinal region and leg |
| B6216 | All | Mycosis fungoides of hymph nodes Mycosis fungoides of intrapelvic lymph nodes |
| B6217 | All | Mycosis fungoides of intrapervic lymph flodes Mycosis fungoides of spleen |
| B6217 | All | Mycosis fungoides of lymph nodes of multiple sites |
| B621z | All | Mycosis fungoides NOS |
| BBI | All | [M]Mycosis fungoides |
| BBIO. | All | [M]Mycosis fungoides |
| BBI1. | | [M]Sezary's disease |
| BBIz. | All | [M]Mycosis fungoides NOS |
| B62xX | All | Oth and unspecif peripheral & cutaneous T-cell lymphomas |
| B62E7 | All | Subcutaneous panniculitis like T-cell lymphoma |
| BBmD. | All | [M]Cutaneous lymphoma |
| B622. | All | Sezary's disease |
| B6220 | All | Sezary's disease of unspecified site |
| B6221 | All | Sezary's disease of lymph nodes of head, face and neck |
| B6222 | All | Sezary's disease of intrathoracic lymph nodes |
| B6223 | All | Sezary's disease of intra-abdominal lymph nodes |
| B6224 | All | Sezary's disease of lymph nodes of axilla and upper limb |
| B6225 | All | Sezary's disease of lymph nodes of inguinal region and leg |
| B6226 | All | Sezary's disease of intrapelvic lymph nodes |
| B6227 | All | Sezary's disease of spleen |
| B6228 | All | Sezary's disease of lymph nodes of multiple sites |
| B622z | All | Sezary's disease NOS |
| Read CTV3 Code | Term ID | Description |
| X78el | All | Squamous cell carcinoma of lip |
| 1 1/201 11 | | |
| X78bU | All | Squamous cell carcinoma of cornea |
| X00Z8 | All | Squamous cell carcinoma of eyelid |
| X00Z8<br>X78RR | All | Squamous cell carcinoma of eyelid Squamous cell carcinoma of skin |
| X00Z8<br>X78RR<br>Xa34C | All<br>All | Squamous cell carcinoma of eyelid Squamous cell carcinoma of skin Squamous cell carcinoma of skin of upper lip |
| X00Z8<br>X78RR | All | Squamous cell carcinoma of eyelid Squamous cell carcinoma of skin |

| X78RS | All | Clear cell squamous cell carcinoma of skin |
|---|---|---|
| X78RT | All | Spindle cell carcinoma of skin |
| X78RU | All | Acantholytic squamous cell carcinoma of skin |
| X78RV | All | Plantar verrucous squamous cell carcinoma of skin |
| Xa0EY | All | Squamous cell carcinoma of scrotum |
| X78Xw | All | - |
| | | Squamous cell carcinoma of vulva |
| B33z.<br>X78bM | All | Squamous cell carcinoma of skin NOS |
| | All | Squamous cell carcinoma of conjunctiva |
| X78gS | All | Squamous cell carcinoma of anal margin |
| X78RW | All | Squamous cell carcinoma in situ of skin |
| X78il | All | Queryat's erythroplasia |
| X0027 | All | Bowen's disease of eyelid |
| XaEJc | All | Bowen's disease of vulva |
| X78VL | All | Basal cell naevus syndrome |
| X78SS | All | Basal cell carcinoma of skin |
| X78ST | All | Basosquamous carcinomaof skin |
| X78VL | All | Naevoid basal cell carcinoma syndrome |
| X78SU | All | Fibroepithelioma of Pinkus |
| X78VK | All | Follicularatrophoderma and basal cell epitheliomata |
| X00Z9 | All | Basal cell carcinoma of eyelid |
| Xa7OT | All | Excision of basal cell carcinoma |
| 7G056 | All | Excision biopsy of basal cell carcinoma |
| Xa7OU | All | Cryotherapy of basal cell carcinoma |
| X78ST | All | Metatypical basal cell carcinoma of skin |
| X78Sg | All | Basal cell carcinoma with eccrine differentiation |
| XM1ML | All | Epithelioma basal cell |
| X77nR | All | Merkel cell carcinoma |
| X78ha | All | Kaposi's sarcoma of skin |
| X78Ut | All | Epitheliod sarcoma of skin |
| B621. | All | Mycosis fungoides |
| XaQbT | All | Poikiloderma vasculare atrophicans |
| X78hm | All | Mycosis fungoides of skin |
| B6210 | All | Mycosis fungoides of unspecified site |
| B6211 | All | Mycosis fungoides of lymph nodes of head, face and neck |
| B6212 | All | Mycosis fungoides of intrathoracic lymph nodes |
| B6213 | All | Mycosis fungoides of intra-abdominal lymph nodes |
| B6214 | All | Mycosis fungoides of lymph nodes of axilla and upper limb |
| B6215 | All | Mycosis fungoides of lymph nodes of inguinal region and leg |
| B6216 | All | Mycosis fungoides of intrapelvic lymph nodes |
| B6217 | All | Mycosis fungoides of spleen |
| B6218 | All | Mycosis fungoides of lymph nodes of multiple sites |
| B621z | All | Mycosis fungoides NOS |
| B622. | All | Sezary's disease |
| B6220 | All | Sezary's disease of unspecified site |
| B6220 | All | Sezary's disease of unspectified site Sezary's disease of lymph nodes of head, face and neck |
| B6221 | All | Sezary's disease of intrathoracic lymph nodes |
| B6223 | All | Sezary's disease of intra-abdominal lymph nodes |
| B6224 | All | Sezary's disease of lymph nodes of axilla and upper limb |
| B6225 | All | Sezary's disease of lymph nodes of inguinal region and leg |

| B6227 All Sezary's disease of spieen B6228 All Sezary's disease of lymph nodes of multiple sites B6222 All Sezary's disease of lymph nodes of multiple sites B6222 All Sezary's disease NOS X78hn All Cutaneous lymphoma XAVin All Cutaneous lymphoma XAVin All Cutaneous lymphoma XAVin All Cutaneous panniculitis like T-cell lymphoma XAVIf All Subcutaneous panniculitis like T-cell lymphoma XAVIf All Subcutaneous panniculitis like T-cell lymphoma XAVIf All Subcutaneous panniculitis like T-cell lymphoma XAVII All lymphomas Primary cutaneous CD30 antigen positive large T-cell lymphoma All lymphomas Primary cutaneous CD30 antigen positive large T-cell lymphoma XAVII All lymphoma Squamous cell carcinoma (disorder) Squamous cell carcinoma (disorder) Squamous cell carcinoma of anal margin (disorder) Squamous cell carcinoma of anal margin (disorder) Squamous cell carcinoma of penis (disorder) Squamous cell carcinoma of penis (disorder) Squamous cell carcinoma of penis (disorder) Squamous cell carcinoma of penis (disorder) Squamous cell carcinoma of back (disorder) Squamous cell carcinoma of foot (disorder) Squamous cell carcinoma of chin (disorder) Squamous cell carcinoma of chin (disorder) Squamous cell carcinoma of chin (disorder) Squamous cell carcinoma of chin (disorder) Squamous cell carcinoma of nose (disorder) Squamous cell carcinoma of scalp (disorder) Squamous cell carcinoma of of cornea (disorder) Squamous cell carcinoma of cornea (disorder) Squamous cell carcinoma of evelid (disorder) Papillary squamous cell carcinoma (morphologic abnormality) S | B6226 | All | Sezary's disease of intrapelvic lymph nodes |
|---|---|---|---|
| B6228 | | | |
| B622z All Sezary's disease NOS | | | , |
| X78hn All Sezary's disease of skin X78hl All Cutaneous lymphoma XaYin All Cutaneous lymphoma XaYin All Cutaneous follicle centre lymphoma XaOSZ All Cutaneous follicle centre lymphoma XaYif All Subcutaneous panniculitis like T-cell lymphoma XaYif All Subcutaneous panniculitis like T-cell lymphoma XaYif All Subcutaneous panniculitis like T-cell lymphoma XaYil Yindhama Primary cutaneous CD30 antigen positive large T-cell lymphoma Yindhama Primary cutaneous CD30 antigen positive large T-cell lymphoma Yindhama | | | |
| X78hl All Cutaneous lymphoma XaVin All Cutaneous follicle centre lymphoma XaVin All Cutaneous follicle centre lymphoma XaVif All Subcutaneous panniculitis like T-cell lymphoma XaVif All Subcutaneous panniculitis like T-cell lymphoma XaVif All Subcutaneous panniculitis like T-cell lymphoma Xi)Oth and unspecif peripheral & cutaneous T-cell lymphomas Primary cutaneous CD30 antigen positive large T-cell lymphoma SNOMED Code Term ID Description Squamous cell carcinoma (disorder) Squamous cell carcinoma, no International Classification of Diseases for Oncology subtype (morphologic abnormality) 255084004 Squamous cell carcinoma of anal margin (disorder) 403468003 Squamous cell carcinoma of anal margin (disorder) 403468003 Squamous cell carcinoma of penis (disorder) 403468003 Squamous cell carcinoma of penis (disorder) 403468003 Squamous cell carcinoma of penis (disorder) 403468003 Squamous cell carcinoma of penis (disorder) 403896005 Squamous cell carcinoma of lip (disorder) 403896003 Squamous cell carcinoma of hand (disorder) 403896003 Squamous cell carcinoma of hand (disorder) 403895004 Squamous cell carcinoma of note (disorder) 403895004 Squamous cell carcinoma of note (disorder) 403895004 Squamous cell carcinoma of note (disorder) 403895004 Squamous cell carcinoma of note (disorder) 403895004 Squamous cell carcinoma of note (disorder) 59529006 Squamous cell carcinoma of note (disorder) 59529006 Squamous cell carcinoma of note (disorder) 5962900 Squamous cell carcinoma of note (disorder) 5929006 Squamous cell carcinoma of cornea (disorder) 5929006 Squamous cell carcinoma of cornea (disorder) 5929006 Squamous cell carcinoma of mouth (disorder) 5929006 Squamous cell carcinoma of mouth (disorder) 5929006 Squamous cell carcinoma of mouth (disorder) 5929009 Spindle cell carcinoma of mouth (disorder) 5929009 Squamous cell carcinoma of cornea (disorder) 5929000 Squamous cell carcinoma of cornea (disorder) 5929000 Squamous cell carcinoma of cornea (disorder) 5929000 Squamous cell carcinoma of cornea (disorder) 5929000 Squa | | | |
| XaVin All Cutaneous follicle centre lymphoma XaOS2 All Cutaneous/peripheral T-cell lymphoma XaViff All Subcutaneous panniculitis like T-cell lymphoma [XIOth and unspecif peripheral & cutaneous T-cell lymphomas Primary cutaneous CD30 antigen positive large T-cell lymphomas Primary cutaneous CD30 antigen positive large T-cell lymphoma SNOMED Code Term ID Description Squamous cell carcinoma, no International Classification of Diseases for Oncology subtype (morphologic abnormality) 255084004 Squamous cell carcinoma of anal margin (disorder) 255084004 Squamous cell carcinoma of anal margin (disorder) 255084004 Squamous cell carcinoma of gem (disorder) 276953005 Squamous cell carcinoma of gem (disorder) 276953005 Squamous cell carcinoma of gem (disorder) 276953005 Squamous cell carcinoma of gem (disorder) 276953005 Squamous cell carcinoma of back (disorder) 276953005 Squamous cell carcinoma of foot (disorder) 276953005 Squamous cell carcinoma of hack (disorder) 276953006 Squamous cell carcinoma of hose (disorder) 276953006 Squamous cell carcinoma of hose (disorder) 276953007 Squamous cell carcinoma of nose (disorder) 276953008 Squamous cell carcinoma of nose (disorder) 276953009 Squamous cell carcinoma of nose (disorder) 276953000 Squamous cell carcinoma of nose (disorder) 2776953000 Squamous cell carcinoma of nose (disorder) 2776953000 Squamous cell carcinoma of nose (disorder) 2776953000 Squamous cell carcinoma of nose (disorder) 27776000 Squamous cell carcinoma of nose (disorder) 27776000 Squamous cell carcinoma of nose (disorder) 277776000 Squamous cell carcinoma of nose (disorder) 2777777777777777777777777777777777777 | | + | , |
| Xa0Sz All Cutaneous/peripheral T-cell lymphoma Xavjf All Subcutaneous panniculitis like T-cell lymphoma [X]Oth and unspecif peripheral & cutaneous T-cell lymphoma Navjl All lymphoma Navjl All lymphoma Navjl All lymphoma Navjl All lymphoma Navjl NOMED Code Navjl NOMED Code Navjl Nome Nome | | | · · |
| XaYjf | | + | |
| [X]0th and unspecif peripheral & cutaneous T-cell lymphomas | | - | |
| ByuDD | XaYjt | All | |
| Primary cutaneous CD30 antigen positive large T-cell lymphoma | | | |
| XaYji | ByuDD | All | |
| SNOMED Code Term ID Description 402815007 Squamous cell carcinoma, no International Classification of Diseases for Oncology subtype (morphologic abnormality) 28899001 Squamous cell carcinoma, no International Classification of Diseases for Oncology subtype (morphologic abnormality) 255084004 Squamous cell carcinoma of anal margin (disorder) 425303004 Squamous cell carcinoma of penis (disorder) 276953005 Squamous cell carcinoma of gum (disorder) 255071008 Squamous cell carcinoma of gip (disorder) 422599000 Squamous cell carcinoma of back (disorder) 403896003 Squamous cell carcinoma of hand (disorder) 403895004 Squamous cell carcinoma of foot (disorder) 422572002 Squamous cell carcinoma of foot (disorder) 448930008 Squamous cell carcinoma of nose (disorder) Squamous cell carcinoma of nose (disorder) Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) 859529006 Adenoid squamous cell carcinoma (morphologic abnormality) 85956000 Squamous cell carcinoma in situ (disorder) 85956000 Squamous cell carcinoma of mouth (disorder) 86692009 Spindle | | | |
| Squamous cell carcinoma (disorder) | • | | |
| Squamous cell carcinoma, no International Classification of Diseases for Oncology subtype (morphologic abnormality) 255084004 Squamous cell carcinoma of anal margin (disorder) 425303004 Squamous cell carcinomatosis (disorder) 425303005 Squamous cell carcinoma of penis (disorder) 276953005 Squamous cell carcinoma of gum (disorder) 255071008 Squamous cell carcinoma of lip (disorder) 422599000 Squamous cell carcinoma of back (disorder) 403896003 Squamous cell carcinoma of hand (disorder) 403895004 Squamous cell carcinoma of hand (disorder) 403895004 Squamous cell carcinoma of host (disorder) 422572002 Squamous cell carcinoma of nose (disorder) 448930008 Squamous cell carcinoma of nose (disorder) 59529006 (morphologic abnormality) 59529006 (morphologic abnormality) 426000 Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) 189565007 Squamous cell carcinoma in situ (disorder) 5952909 Squamous cell carcinoma in situ (disorder) 5952009 Squamous cell carcinoma of mouth (disorder) 5952009 Spindle cell carcinoma (morphologic abnormality) 8836100 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 403891008 Squamous cell carcinoma of vulva (disorder) 5050000 Squamous cell carcinoma of scalp (disorder) 5050000 Squamous cell carcinoma of cornea (disorder) 5050000 Squamous cell carcinoma of cornea (disorder) 5050000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 82906000 Verrucous carcinoma of temple (disorder) 82906000 Squamous cell carcinoma of temple (disorder) 82906008 Squamous cell carcinoma of eyelid (disorder) 82056008 Squamous cell carcinoma of eyelid (disorder) 82056008 Squamous cell carcinoma, metastatic (morphologic | | Term ID | • |
| Diseases for Oncology subtype (morphologic abnormality) 255084004 Squamous cell carcinoma of anal margin (disorder) 425303004 Squamous cell carcinomatosis (disorder) 403468003 Squamous cell carcinoma of penis (disorder) 276953005 Squamous cell carcinoma of penis (disorder) 255071008 Squamous cell carcinoma of gum (disorder) 422599000 Squamous cell carcinoma of back (disorder) 403896003 Squamous cell carcinoma of hand (disorder) 403895004 Squamous cell carcinoma of chin (disorder) 422572002 Squamous cell carcinoma of nose (disorder) 44893008 Squamous cell carcinoma of nose (disorder) Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) Adenoid squamous cell carcinoma (morphologic abnormality) Adenoid squamous cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 823700001 Squamous cell carcinoma of scalp (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 525008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 89906000 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) Papillary squamous cell carcinoma (morphologic abnormality) 8006008 Squamous cell carcinoma of eyelid (disorder) Papillary squamous cell carcinoma (morphologic abnormality) Papillary squamous cell carcinoma (morphologic abnormality) Papillary squamous cell carcinoma (morphologic abnormality) Papillary squamous cell carcinoma (morphologic abnormality) Papillary squamous cell carcinoma (morphologic abnormality) | 402815007 | | . , |
| Squamous cell carcinoma of anal margin (disorder) | | | |
| 425303004 Squamous cell carcinomatosis (disorder) 403468003 Squamous cell carcinoma of penis (disorder) 276953005 Squamous cell carcinoma of gum (disorder) 255071008 Squamous cell carcinoma of gum (disorder) 422599000 Squamous cell carcinoma of back (disorder) 422599000 Squamous cell carcinoma of back (disorder) 403895004 Squamous cell carcinoma of hand (disorder) 422572002 Squamous cell carcinoma of coti (disorder) 422572002 Squamous cell carcinoma of nose (disorder) 422572002 Squamous cell carcinoma of nose (disorder) 4295008 Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) 403895600 abnormality) 403895600 Squamous cell carcinoma (morphologic abnormality) 40408000 Squamous cell carcinoma of mouth (disorder) 40592009 Spindle cell carcinoma (morphologic abnormality) 403891008 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 403891008 Squamous cell carcinoma of vulva (disorder) 403891008 Squamous cell carcinoma of vulva (disorder) 403891008 Squamous cell carcinoma of vulva (disorder) 403891008 Squamous cell carcinoma of vulva (disorder) 403891008 Squamous cell carcinoma of vulva (disorder) 4254895003 Squamous cell carcinoma of vulva (disorder) 4254895000 Squamous cell carcinoma of vulva (disorder) 425480500 Squamous cell carcinoma of vulva (disorder) 42548008 Squamous cell carcinoma of vulva (disorder) 42548008 Squamous cell carcinoma (morphologic abnormality) 42548008 Squamous cell carcinoma (morphologic abnormality) 4266008 Squamous cell carcinoma of temple (disorder) 42548008 Squamous cell carcinoma ( | | | |
| 403468003 Squamous cell carcinoma of penis (disorder) 276953005 Squamous cell carcinoma of gum (disorder) 255071008 Squamous cell carcinoma of lip (disorder) 422599000 Squamous cell carcinoma of back (disorder) 403896003 Squamous cell carcinoma of hand (disorder) 403895004 Squamous cell carcinoma of foot (disorder) 422572002 Squamous cell carcinoma of chin (disorder) 448930008 Squamous cell carcinoma of chin (disorder) 448930008 Squamous cell carcinoma of nose (disorder) 59529006 Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) 4297600 Adenoid squamous cell carcinoma (morphologic abnormality) 8595600 Squamous cell carcinoma in situ (disorder) 8707502000 Squamous cell carcinoma of mouth (disorder) 8707502000 Squamous cell carcinoma of mouth (disorder) 8707502000 Spindle cell carcinoma (morphologic abnormality) 8707502000 Squamous cell carcinoma of mouth (disorder) 8707502000 Squamous cell carcinoma of mouth (disorder) 8707502000 Squamous cell carcinoma of mouth (disorder) 8707502000 Squamous cell carcinoma of mouth (disorder) 8707502000 Squamous cell carcinoma of auricle of ear (disorder) 8707502000 Squamous cell carcinoma of scalp (disorder) 8707502000 Squamous cell carcinoma of scalp (disorder) 8707502000 Squamous cell carcinoma of scalp (disorder) 8707502000 Squamous cell carcinoma of cornea (disorder) 8707502000 Squamous cell carcinoma of cornea (disorder) 8707502000 Squamous cell carcinoma (morphologic abnormality) 8719052000 Squamous cell carcinoma of temple (disorder) 8707502000 Squamous cell carcinoma of temple (disorder) 870752000 Squamous cell carcinoma of temple (disorder) 870752000 Squamous cell carcinoma of temple (disorder) 870752000 Squamous cell carcinoma of temple (disorder) 870752000 Squamous cell carcinoma of temple (disorder) 870752000 Squamous cell carcinoma (morphologic abnormality) 870752000 Squamous cell carcinoma (morphologic abnormality) 870752000 Squamous cell carcinoma (morphologic abnormality) 870752000 Squamo | 255084004 | | |
| 276953005 Squamous cell carcinoma of gum (disorder) 255071008 Squamous cell carcinoma of lip (disorder) 422599000 Squamous cell carcinoma of back (disorder) 403896003 Squamous cell carcinoma of hand (disorder) 403895004 Squamous cell carcinoma of foot (disorder) 422572002 Squamous cell carcinoma of chin (disorder) 448930008 Squamous cell carcinoma of nose (disorder) 5quamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) 859529006 (morphologic abnormality) 85956000 Squamous cell carcinoma in situ (disorder) 870000 Squamous cell carcinoma of mouth (disorder) 8700000 Squamous cell carcinoma (morphologic abnormality) 88365007 Squamous cell carcinoma (morphologic abnormality) 88365007 Squamous cell carcinoma of mouth (disorder) 890000 Spindle cell carcinoma (morphologic abnormality) 8838101 Squamous cell carcinoma of auricle of ear (disorder) 89381008 Squamous cell carcinoma of scalp (disorder) 89390000 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 89906000 Squamous cell carcinoma of temple (disorder) 89911 Papillary squamous cell carcinoma (morphologic abnormality) 8231831002 Squamous cell carcinoma of eyelid (disorder) 8905000 History of squamous cell carcinoma (situation) 8005000 Squamous cell carcinoma (morphologic abnormality) 8005000 Squamous cell carcinoma of eyelid (disorder) 8005000 Squamous cell carcinoma of eyelid (disorder) | 425303004 | | Squamous cell carcinomatosis (disorder) |
| Squamous cell carcinoma of lip (disorder) | 403468003 | | Squamous cell carcinoma of penis (disorder) |
| 422599000 Squamous cell carcinoma of back (disorder) 403896003 Squamous cell carcinoma of hand (disorder) 403895004 Squamous cell carcinoma of foot (disorder) 422572002 Squamous cell carcinoma of chin (disorder) 42893008 Squamous cell carcinoma of nose (disorder) Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) Adenoid squamous cell carcinoma (morphologic abnormality) 189565007 Squamous cell carcinoma in situ (disorder) 307502000 Squamous cell carcinoma of mouth (disorder) 65692009 Spindle cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 25508003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 89906000 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 276953005 | | Squamous cell carcinoma of gum (disorder) |
| 403896003 Squamous cell carcinoma of hand (disorder) 403895004 Squamous cell carcinoma of foot (disorder) 422572002 Squamous cell carcinoma of chin (disorder) 448930008 Squamous cell carcinoma of nose (disorder) Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) Adenoid squamous cell carcinoma (morphologic abnormality) 189565007 Squamous cell carcinoma in situ (disorder) 307502000 Squamous cell carcinoma of mouth (disorder) 55952909 Spindle cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 128634009 Basaloid squamous cell carcinoma (morphologic abnormality) 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of vulva (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 255071008 | | Squamous cell carcinoma of lip (disorder) |
| 403895004 Squamous cell carcinoma of foot (disorder) 422572002 Squamous cell carcinoma of chin (disorder) 448930008 Squamous cell carcinoma of nose (disorder) Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) Adenoid squamous cell carcinoma (morphologic abnormality) 189565007 Squamous cell carcinoma in situ (disorder) 307502000 Squamous cell carcinoma of mouth (disorder) 55692009 Spindle cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 128634009 Aguamous cell carcinoma of auricle of ear (disorder) 423700001 Squamous cell carcinoma of scalp (disorder) 403891008 Squamous cell carcinoma of svulva (disorder) 254895003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 719052006 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) Papillary squamous cell carcinoma (morphologic abnormality) Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) | 422599000 | | Squamous cell carcinoma of back (disorder) |
| 422572002Squamous cell carcinoma of chin (disorder)448930008Squamous cell carcinoma of nose (disorder)Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality)44893000Adenoid squamous cell carcinoma (morphologic abnormality)85956000Squamous cell carcinoma in situ (disorder)307502000Squamous cell carcinoma of mouth (disorder)65692009Spindle cell carcinoma (morphologic abnormality)8asaloid squamous cell carcinoma (morphologic abnormality)423700001Squamous cell carcinoma of auricle of ear (disorder)403891008Squamous cell carcinoma of scalp (disorder)254895003Squamous cell carcinoma of vulva (disorder)255008003Squamous cell carcinoma of cornea (disorder)89906000Verrucous carcinoma (morphologic abnormality)719052006Recurrent squamous cell carcinoma (disorder)425148008Squamous cell carcinoma of temple (disorder)Papillary squamous cell carcinoma (morphologic abnormality)231831002Squamous cell carcinoma of eyelid (disorder)69551000119109History of squamous cell carcinoma (situation)Squamous cell carcinoma, metastatic (morphologic | 403896003 | | Squamous cell carcinoma of hand (disorder) |
| Squamous cell carcinoma of nose (disorder) Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) Adenoid squamous cell carcinoma (morphologic abnormality) 189565007 Squamous cell carcinoma in situ (disorder) 307502000 Squamous cell carcinoma of mouth (disorder) 556692009 Spindle cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 403895004 | | Squamous cell carcinoma of foot (disorder) |
| Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) Adenoid squamous cell carcinoma (morphologic abnormality) 189565007 Squamous cell carcinoma in situ (disorder) 307502000 Squamous cell carcinoma of mouth (disorder) 65692009 Spindle cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 422572002 | | Squamous cell carcinoma of chin (disorder) |
| Squamous cell carcinoma in situ, no International Classification of Diseases for Oncology subtype (morphologic abnormality) Adenoid squamous cell carcinoma (morphologic abnormality) 189565007 Squamous cell carcinoma in situ (disorder) 307502000 Squamous cell carcinoma of mouth (disorder) 65692009 Spindle cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 448930008 | | Squamous cell carcinoma of nose (disorder) |
| S9529006 | | | Squamous cell carcinoma in situ, no International |
| S9529006 | | | Classification of Diseases for Oncology subtype |
| abnormality) 189565007 Squamous cell carcinoma in situ (disorder) 307502000 Squamous cell carcinoma of mouth (disorder) 65692009 Spindle cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 39056008 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 59529006 | | |
| 189565007 Squamous cell carcinoma in situ (disorder) 307502000 Squamous cell carcinoma of mouth (disorder) 65692009 Spindle cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | | | Adenoid squamous cell carcinoma (morphologic |
| Squamous cell carcinoma of mouth (disorder) Spindle cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 85956000 | | abnormality) |
| Spindle cell carcinoma (morphologic abnormality) Basaloid squamous cell carcinoma (morphologic abnormality) 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 189565007 | | Squamous cell carcinoma in situ (disorder) |
| Basaloid squamous cell carcinoma (morphologic abnormality) 423700001 | 307502000 | | Squamous cell carcinoma of mouth (disorder) |
| abnormality) 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 65692009 | | Spindle cell carcinoma (morphologic abnormality) |
| 423700001 Squamous cell carcinoma of auricle of ear (disorder) 403891008 Squamous cell carcinoma of scalp (disorder) 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | | | Basaloid squamous cell carcinoma (morphologic |
| 403891008 Squamous cell carcinoma of scalp (disorder) Squamous cell carcinoma of vulva (disorder) Squamous cell carcinoma of cornea (disorder) Squamous cell carcinoma of cornea (disorder) Verrucous carcinoma (morphologic abnormality) Recurrent squamous cell carcinoma (disorder) Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 128634009 | | abnormality) |
| 254895003 Squamous cell carcinoma of vulva (disorder) 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 423700001 | | Squamous cell carcinoma of auricle of ear (disorder) |
| 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 403891008 | | Squamous cell carcinoma of scalp (disorder) |
| 255008003 Squamous cell carcinoma of cornea (disorder) 89906000 Verrucous carcinoma (morphologic abnormality) 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 254895003 | | Squamous cell carcinoma of vulva (disorder) |
| 89906000 Verrucous carcinoma (morphologic abnormality) Recurrent squamous cell carcinoma (disorder) Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 255008003 | | |
| 719052006 Recurrent squamous cell carcinoma (disorder) 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 89906000 | | · |
| 425148008 Squamous cell carcinoma of temple (disorder) Papillary squamous cell carcinoma (morphologic abnormality) Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 719052006 | | |
| Papillary squamous cell carcinoma (morphologic abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | | | |
| 39056008 abnormality) 231831002 Squamous cell carcinoma of eyelid (disorder) 69551000119109 History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | | | |
| 231831002 Squamous cell carcinoma of eyelid (disorder) 69551000119109 History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | 39056008 | | . , |
| 69551000119109 History of squamous cell carcinoma (situation) Squamous cell carcinoma, metastatic (morphologic | | | |
| Squamous cell carcinoma, metastatic (morphologic | | | |
| , , , , , | | | |
| | 64204000 | | , |

| 423700001 | Squamous cell carcinoma of auricle of ear (disorder) |
|-----------|--------------------------------------------------------|
| 276860003 | Squamous cell carcinoma of scrotum (disorder) |
| 403905005 | Multiple squamous cell carcinomata (disorder) |
| 403903003 | Signet ring squamous cell carcinoma (disorder) |
| 403893006 | Squamous cell carcinoma of forehead (disorder) |
| | Metaplastic squamous cell carcinoma (morphologic |
| 399739006 | abnormality) |
| 448931007 | Squamous cell carcinoma of shoulder (disorder) |
| 450434000 | Excision of squamous cell carcinoma (procedure) |
| 37304002 | Basosquamous carcinoma (morphologic abnormality) |
| 422676009 | Squamous cell carcinoma of ala nasi (disorder) |
| 403901001 | Acantholytic squamous cell carcinoma (disorder) |
| | Squamous cell carcinoma, spindle cell (morphologic |
| 10288008 | abnormality) |
| | Disseminated squamous cell carcinoma (morphologic |
| 300987004 | abnormality) |
| 403900000 | Spindle cell squamous cell carcinoma (disorder) |
| | Squamous cell carcinoma, keratinizing (morphologic |
| 18048008 | abnormality) |
| | Squamous cell carcinoma, microinvasive (morphologic |
| 12478003 | abnormality) |
| 733344004 | Primary squamous cell carcinoma of lip (disorder |
| 403894000 | Squamous cell carcinoma of skin of ear (disorder) |
| 722112006 | Primary squamous cell carcinoma of ear (disorder) |
| | Pseudovascular squamous cell carcinoma (morphologic |
| 733897002 | abnormality) |
| 255003007 | Squamous cell carcinoma of conjunctiva (disorder) |
| 423896007 | Squamous cell carcinoma of tip of nose (disorder) |
| 89906000 | Verrucous carcinoma (morphologic abnormality) |
| 423284006 | Squamous cell carcinoma of skin of neck (disorder) |
| 400066006 | Intraepithelial squamous cell carcinoma (disorder) |
| 254656002 | Squamous cell carcinoma in situ of skin (disorder) |
| 723265000 | Primary squamous cell carcinoma of anus (disorder) |
| 403892001 | Squamous cell carcinoma of skin of face (disorder) |
| 716659002 | Squamous cell carcinoma of head and neck (disorder) |
| 440527006 | Primary squamous cell carcinoma of naris (disorder) |
| | Squamous cell carcinoma, clear cell type (morphologic |
| 128635005 | abnormality) |
| | Squamous cell carcinoma, large cell, nonkeratinizing |
| 45490001 | (morphologic abnormality) |
| 403899005 | Squamous cell carcinoma of skin of trunk (disorder) |
| 402817004 | Squamous cell carcinoma of nail apparatus (disorder) |
| 422378004 | Squamous cell carcinoma of bridge of nose (disorder) |
| | Papillary squamous cell carcinoma, non-invasive |
| 128647004 | (morphologic abnormality) |
| 429024007 | History of squamous cell carcinoma of skin (situation) |
| 254652000 | Clear cell squamous cell carcinoma of skin (disorder) |
| 424260006 | Squamous cell carcinoma of nasolabial fold (disorder) |
| 403897007 | Squamous cell carcinoma of upper extremity (disorder) |
| 402816008 | Squamous cell carcinoma of anogenital area (disorder) |

| 403896003 | Squamous cell carcinoma of hand (disorder) |
|---|---|
| 254895003 | Squamous cell carcinoma of vulva (disorder) |
| 1082071000119102 | Primary squamous cell carcinoma of left ear (disorder) |
| | Squamous cell carcinoma with horn formation |
| 128633003 | (morphologic abnormality) |
| 403891008 | Squamous cell carcinoma of scalp (disorder) |
| 1082191000119100 | Primary squamous cell carcinoma of right ear (disorder) |
| 285308002 | Squamous cell carcinoma of skin of lower lip (disorder) |
| 285307007 | Squamous cell carcinoma of skin of upper lip (disorder) |
| 91151000119103 | Primary squamous cell carcinoma of chest wall (disorder) |
| | Squamous cell carcinoma in situ of skin caused by sunlight |
| 789051005 | (disorder) |
| | Psoralen and long-wave ultraviolet radiation therapy- |
| 403713003 | associated squamous cell carcinoma (disorder) |
| 448165009 | Squamous cell carcinoma arising in chronic ulcer (disorder) |
| | Squamous cell carcinoma of external auditory canal |
| 423506005 | (disorder) |
| | Squamous cell carcinoma of skin of lower extremity |
| 403898002 | (disorder) |
| 285309005 | Squamous cell carcinoma of skin of cheek (disorder) |
| 422378004 | Squamous cell carcinoma of bridge of nose (disorder) |
| 84999002 | Bowen's disease (morphologic abnormality) |
| 0.00000 | Squamous cell carcinoma, large cell, nonkeratinizing |
| 45490001 | (morphologic abnormality) |
| | Squamous cell carcinoma, small cell, nonkeratinizing |
| 35718007 | (morphologic abnormality) |
| | Human papillomavirus positive squamous cell carcinoma |
| 783212001 | (morphologic abnormality) |
| | Metastasis to lymph node from squamous cell carcinoma |
| 1671000119100 | (disorder) |
| | Squamous cell carcinoma in post-traumatic skin lesion |
| 399494004 | (morphologic abnormality) |
| | Human papillomavirus negative squamous cell carcinoma |
| 783213006 | (morphologic abnormality) |
| | Primary squamous cell carcinoma of lacrimal apparatus |
| 722666002 | (disorder) |
| | Squamous cell carcinoma of mucous membrane of lower lip |
| 418372008 | (disorder) |
| | Squamous cell carcinoma, nonkeratinizing, differentiated |
| 399582005 | (morphologic abnormality) |
| | Undifferentiated nonkeratinizing squamous cell carcinoma |
| 449778005 | (morphologic abnormality) |
| 24111000119105 | Primary squamous cell carcinoma of upper limb (disorder) |
| | Squamous cell carcinoma of vulva due to lichen sclerosus |
| 403890009 | (disorder) |
| 91151000119103 | Primary squamous cell carcinoma of chest wall (disorder) |
| | Primary squamous cell carcinoma of skin of left lower limb |
| 1082101000119106 | (disorder) |
| | Primary squamous cell carcinoma of vermilion border of lip |
| 242951000119108 | (disorder) |

| | Squamous cell carcinoma in situ of skin caused by sunlight |
|---|---|
| 789051005 | (disorder) |
| 703031003 | Primary squamous cell carcinoma of skin of right lower limb |
| 1082221000119106 | (disorder) |
| 1002221000113100 | Squamous cell carcinoma - category (morphologic |
| 400155002 | abnormality) |
| | Intraepithelial squamous cell carcinoma of anogenital |
| 767544007 | region (disorder) |
| | Squamous cell carcinoma of mucous membrane of upper lip |
| 419240004 | (disorder) |
| | Squamous cell carcinoma in situ with questionable stromal |
| 5688000 | invasion (morphologic abnormality) |
| | Undifferentiated nonkeratinizing squamous cell carcinoma |
| 449778005 | (morphologic abnormality) |
| | Squamous cell carcinoma, nonkeratinizing, mixed |
| | differentiated and undifferentiated (morphologic |
| 399694008 | abnormality) |
| 724504004 | Primary squamous cell carcinoma of overlapping lesion of |
| 721604004 | male genital organ (disorder) |
| | Grade III squamous intraepithelial neoplasia with |
| 449406000 | microinvasive squamous cell carcinoma (morphologic |
| 448406002 | abnormality) |
| 1338007 | Basal cell carcinoma (morphologic abnormality) |
| 402521004 | Basal cell carcinoma of upper extremity (disorder) |
| 403912001<br>402820007 | Cystic basal cell carcinoma (disorder) |
| 402820007 | Basal cell carcinoma of ear (disorder) |
| 402519009 | Basal cell carcinoma of hand (disorder) Basal cell carcinoma of face (disorder) |
| 402319009 | Basal cell carcinoma of nose (disorder) |
| 402010009 | Basal cell carcinoma with eccrine differentiation |
| 399470004 | (morphologic abnormality) |
| 423463003 | Basal cell carcinoma of back (disorder) |
| 402509003 | Basal cell carcinoma of neck (disorder) |
| 80071000119103 | Basal cell carcinoma of skin in situ (disorder) |
| 403915004 | Basal cell carcinoma of scalp (disorder) |
| 717731002 | Basal cell carcinoma of vulva (disorder) |
| 402507001 | Basal cell carcinoma of cheek (disorder) |
| 128636006 | Basal cell carcinoma, nodular (morphologic abnormality) |
| 61471000119100 | Basal cell carcinoma of naris (disorder) |
| 424666005 | Basal cell carcinoma of auricle of ear (disorder) |
| 402513005 | Basal cell carcinoma of tragus (disorder) |
| 402536001 | Basal cell carcinoma - primary (disorder) |
| 402525008 | Basal cell carcinoma - adenoid (disorder) |
| 399585007 | Pigmented basal cell carcinoma (morphologic abnormality) |
| 403909004 | Pigmented basal cell carcinoma (disorder) |
| 402538000 | Recurrent basal cell carcinoma (disorder) |
| 231832009 | Basal cell carcinoma of eyelid (disorder) |
| 403917007 | Basal cell carcinoma of temple (disorder) |
| 56665009 | Infiltrating basal cell carcinoma (morphologic abnormality) |
| 399547009 | Keratotic basal cell carcinoma (morphologic abnormality) |
| | the state of the s |

| 403914000 | Superficial basal cell carcinoma (disorder) |
|----------------|-------------------------------------------------------------|
| 402537005 | Metastatic basal cell carcinoma (disorder) |
| 402516002 | Basal cell carcinoma of abdomen (disorder) |
| 102310002 | Basal cell carcinoma with follicular differentiation |
| 399746002 | (morphologic abnormality) |
| 399954008 | Basal cell carcinoma of earlobe (disorder) |
| 134152008 | Basal cell carcinoma - morpheic (morphologic abnormality) |
| 400137006 | Basal cell carcinoma - category (morphologic abnormality) |
| 403918002 | Basal cell carcinoma of glabella (disorder) |
| 402500004 | Basal cell carcinoma of ala nasi (disorder) |
| 403916003 | Basal cell carcinoma of forehead (disorder) |
| 403913006 | Morpheic basal cell carcinoma (disorder) |
| 403913006 | |
| 120624000 | , , , |
| 128634009 | abnormality) |
| 300025007 | Excision of basal cell carcinoma (procedure) |
| 402528005 | Basal cell carcinoma - keratotic (disorder) |
| 402506005 | Basal cell carcinoma of lower lip (disorder) |
| 64.000004 | Multifocal superficial basal cell carcinoma (morphologic |
| 61098004 | abnormality) |
| 402526009 | Basal cell carcinoma - follicular (disorder) |
| 402505009 | Basal cell carcinoma of upper lip (disorder) |
| 56665009 | Infiltrating basal cell carcinoma (morphologic abnormality) |
| | Basal cell carcinoma, micronodular (morphologic |
| 400071004 | abnormality) |
| 254701007 | Basal cell carcinoma of skin (disorder) |
| 402512000 | Basal cell carcinoma of antitragus (disorder) |
| 402517006 | Basal cell carcinoma of upper back (disorder) |
| 402518001 | Basal cell carcinoma of lower back (disorder) |
| 423535002 | Basal cell carcinoma of chest wall (disorder) |
| 402527000 | Basal cell carcinoma - infiltrative (disorder) |
| 402502007 | Basal cell carcinoma of tip of nose (disorder) |
| 402529002 | Basal cell carcinoma - micronodular (disorder) |
| 37304002 | Basosquamous carcinoma (morphologic abnormality) |
| 300026008 | Cryotherapy of basal cell carcinoma (procedure) |
| 402819001 | Basal cell carcinoma of skin of lip (disorder) |
| 402524007 | Basal cell carcinoma - adamantinoid (disorder) |
| 402497005 | Basal cell carcinoma of root of nose (disorder) |
| 716274007 | Nodular basal cell carcinoma of skin (disorder) |
| 402494003 | Basal cell carcinoma of lower eyelid (disorder) |
| 402523001 | Basal cell carcinoma of truncal skin (disorder) |
| 80071000119103 | Basal cell carcinoma of skin in situ (disorder) |
| 403919005 | Basal cell carcinoma of upper eyelid (disorder) |
| | Basal cell carcinoma, fibroepithelial (morphologic |
| 43369006 | abnormality) |
| 402510008 | Basal cell carcinoma of helix of ear (disorder) |
| 400057007 | Basal cell carcinoma of pinnal sulcus (disorder) |
| | Basal cell carcinoma - sclerosing type (morphologic |
| 302821007 | abnormality) |
| 403911008 | Nodulo-ulcerative basal cell carcinoma (disorder) |
| 402495002 | Basal cell carcinoma of medial canthus (disorder) |

| 402515003 | Basal cell carcinoma of anterior chest (disorder) |
|---|---|
| 402313003 | Basal cell carcinoma with follicular differentiation |
| 399746002 | (morphologic abnormality) |
| | Basal cell carcinoma - sclerosing type (morphologic |
| 302821007 | abnormality) |
| 402498000 | Basal cell carcinoma of dorsum of nose (disorder) |
| 402508006 | Basal cell carcinoma of chin (disorder) |
| 402546004 | Basal cell carcinoma - third recurrence (disorder) |
| 402532004 | Basal cell carcinoma with monster cells (disorder) |
| 428796002 | Excisional biopsy of basal cell carcinoma (procedure) |
| 402503002 | Basal cell carcinoma of nasal columella (disorder |
| 402519009 | Basal cell carcinoma of face (disorder) |
| 402544001 | Basal cell carcinoma - first recurrence (disorder) |
| 402496001 | Basal cell carcinoma of lateral canthus (disorder) |
| 402521004 | Basal cell carcinoma of upper extremity (disorder) |
| 402522006 | Basal cell carcinoma of lower extremity (disorder) |
| 403910009 | Circumscribed solid basal cell carcinoma (disorder) |
| 1079101000119100 | Primary basal cell carcinoma of left ear (disorder) |
| 402501000 | Basal cell carcinoma of supratip of nose (disorder) |
| 400174005 | Basal cell carcinoma of antihelix of ear (disorder) |
| 402514004 | Basal cell carcinoma of obverse of pinna (disorder) |
| 403913006 | Morpheic basal cell carcinoma (disorder) |
| 254702000 | Basosquamous carcinoma (disorder) |
| 69411000119107 | History of basal cell carcinoma of eyelid (situation) |
| 1079161000119100 | Primary basal cell carcinoma of right ear (disorder) |
| 402504008 | Basal cell carcinoma of naolabial groove (disorder) |
| 428796002 | Excisional biopsy of basal cell carcinoma (procedure) |
| 403909004 | Pigmented basal cell carcinoma (disorder) |
| 399934007 | Basal cell carcinoma of preauricular skin (disorder) |
| 403916003 | Basal cell carcinoma of forehead (disorder) |
| 399897004 | Basal cell carcinoma of postauricular skin (disorder) |
| 1079111000119100 | Primary basal cell carcinoma of left eyelid (disorder) |
| 402511007 | Basal cell carcinoma of conchal bowl of ear (disorder) |
| 402500004 | Basal cell carcinoma of ala nasi (disorder) |
| 300025007 | Excision of basal cell carcinoma (procedure) |
| 1079171000119100 | Primary basal cell carcinoma of right eyelid (disorder) |
| 402534003 | Basal cell carcinoma with signet ring change (disorder) |
| | Psoralen and long-wave ultraviolet radiation therapy- |
| 403712008 | associated basal cell carcinoma (disorder) |
| 402531006 | Basal cell carcinoma with granular cell change (disorder) |
| 80071000119103 | Basal cell carcinoma of skin in situ (disorder) |
| 402497005 | Basal cell carcinoma of root of nose (disorder) |
| 1079091000119100 | Primary basal cell carcinoma of left upper limb |
| 423325007 | Basal cell carcinoma of external auditory canal (disorder) |
| 1079131000119100 | Primary basal cell carcinoma of left lower limb (disorder) |
| 1079151000119100 | Primary basal cell carcinoma of right upper limb (disorder) |
| 1079191000119100 | Primary basal cell carcinoma of right lower limb (disorder) |
| | Basal cell carcinoma with eccrine differentiation |
| 399470004 | (morphologic abnormality) |

| Basal cell carcinoma, fibroepithelial (morphologic abnormality) | | Basal cell carcinoma in basal cell nevus syndrome |
|---|---|---|
| Basal cell carcinoma, fibroepithelial (morphologic abnormality) Basal cell carcinoma with eccrine differentiation (disorder) Basal cell carcinoma with adnexal differentiation (morphologic abnormality) Basal cell carcinoma of lateral side wall of nose (disorder) Basal cell carcinoma of a lateral side wall of nose (disorder) Basal cell carcinoma of dorsum of nose (disorder) Basal cell carcinoma recurrent following excision (disorder) Basal cell carcinoma recurrent following excision (disorder) Basal cell carcinoma recurrent following curettage (disorder) Basal cell carcinoma recurrent following curettage (disorder) Basal cell carcinoma recurrent following curettage (disorder) Basal cell carcinoma recurrent following curettage (disorder) Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma of obverse of pinna (disorder) Basal cell carcinoma of obverse of pinna (disorder) Basal cell carcinoma of obverse of pinna (disorder) Basal cell carcinoma with sarcomatoid differentiation (morphologic abnormality) Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Dasal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel cell carcinoma of oper limb (disorder) Merkel cell carcinoma of face (disorder) 13381000119103 Merkel cell carcinoma of lower limb (disorder) Merkel cell carcinoma of skin (disorder) Primary malignant sarcoma of skin (disorder) Primary malignant sarcoma of skin ( | 399569002 | · |
| abnormality) 254710004 Basal cell carcinoma with eccrine differentiation (disorder) Basal cell carcinoma with adnexal differentiation (morphologic abnormality) Basal cell carcinoma of lateral side wall of nose (disorder) 402499008 Basal cell carcinoma of lateral side wall of nose (disorder) 402498000 Basal cell carcinoma of dorsum of nose (disorder) Basal cell carcinoma recurrent following excision (disorder) Basal cell carcinoma with matrical differentiation (morphologic abnormality) Basal cell carcinoma recurrent following curettage (disorder) Basal cell carcinoma with sebaceous differentiation (morphologic abnormality) Basal cell carcinoma - second recurrence (disorder) Basal cell carcinoma - second recurrence (disorder) Basal cell carcinoma of obverse of pinna (disorder) Basal cell carcinoma of obverse of pinna (disorder) Basal cell carcinoma with sarcomatoid differentiation (morphologic abnormality) Basal cell carcinoma with sarcomatoid differentiation (morphologic abnormality) Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel cell carcinoma of select (disorder) Merkel cell carcinoma of face (disorder) 13881000119105 Merkel cell carcinoma of lower limb (disorder) Merkel cell carcinoma of lower limb (disorder) Merkel cell carcinoma of skin (disorder) Primary malignant sarcoma of skin (disorder) Primary malignant sarcoma of skin (disorder) 1013860008 Saposi's sarcoma of skin (disorder) Prima | | |
| Basal cell carcinoma with adnexal differentiation (disorder) Basal cell carcinoma with adnexal differentiation (morphologic abnormality) 402499008 Basal cell carcinoma of lateral side wall of nose (disorder) 402498000 Basal cell carcinoma of dorsum of nose (disorder) 402498000 Basal cell carcinoma of dorsum of nose (disorder) 402539008 Basal cell carcinoma recurrent following excision (disorder) Basal cell carcinoma with matrical differentiation (morphologic abnormality) Basal cell carcinoma recurrent following curettage (disorder) Basal cell carcinoma with sebaceous differentiation (morphologic abnormality) Basal cell carcinoma second recurrence (disorder) Basal cell carcinoma - second recurrence (disorder) Basal cell carcinoma of obverse of pinna (disorder) Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel cell carcinoma (disorder) Basal tell carcinoma of fower limb (disorder) Merkel cell carcinoma of fower limb (disorder) Merkel cell carcinoma of fower limb (disorder) Merkel cell carcinoma of fisht lower limb (disorder) Merkel cell carcinoma of fisht lower limb (disorder) Primary malignant sarcoma of skin (disorder) Merkel cell carcinoma of skin (disorder) Despensal fell carcinoma of skin (disorder) Merkel cell carcinoma of skin (disorder) Merkel cell carcinoma of skin (disorder) Merkel | 43369006 | |
| 399487002 (morphologic abnormality) | 254710004 | |
| Basal cell carcinoma of lateral side wall of nose (disorder) | | Basal cell carcinoma with adnexal differentiation |
| Basal cell carcinoma of lateral side wall of nose (disorder) | 399487002 | (morphologic abnormality) |
| Basal cell carcinoma recurrent following excision (disorder) | 402499008 | Basal cell carcinoma of lateral side wall of nose (disorder) |
| Basal cell carcinoma with matrical differentiation (morphologic abnormality) Basal cell carcinoma recurrent following curettage (disorder) Basal cell carcinoma with sebaceous differentiation (morphologic abnormality) 402545000 Basal cell carcinoma - second recurrence (disorder) Basal cell carcinoma of obverse of pinna (disorder) Basal cell carcinoma of obverse of pinna (disorder) Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel cell carcinoma (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel cell carcinoma (disorder) 10149001 Merkel cell carcinoma (disorder) 33841000119105 Merkel cell carcinoma of face (disorder) 133841000119105 Merkel cell carcinoma of face (disorder) 133841000119106 Merkel cell carcinoma of lower limb (disorder) 352071000119105 Merkel cell carcinoma of lower limb (disorder) 72154109 Primary malignant sarcoma of skin (disorder) 72154109 Primary malignant sarcoma of skin (disorder) 72154109 Primary malignant sarcoma of skin (disorder) 72154109 Primary malignants arcoma of skin (disorder) 72154109 Primary malignants arcoma of skin (disorder) 72154109 Primary malignants arcoma of skin (disorder) 72154109 Primary malignantsarcoma of skin (disorder) 72154109 Primary malignants arcoma of skin (disorder) 72154109 | 402498000 | Basal cell carcinoma of dorsum of nose (disorder) |
| 39958006 | 402539008 | Basal cell carcinoma recurrent following excision (disorder) |
| Basal cell carcinoma recurrent following curettage (disorder) Basal cell carcinoma with sebaceous differentiation (morphologic abnormality) 402545000 Basal cell carcinoma - second recurrence (disorder) Basal cell carcinoma of obverse of pinna (disorder) Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma with sarcomatoid differentiation (morphologic abnormality) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel cell carcinoma (disorder) Merkel cell carcinoma (disorder) Merkel cell carcinoma of face (disorder) 133841000119105 Merkel cell carcinoma of face (disorder) 133841000119100 Merkel cell carcinoma of lower limb (disorder) Merkel cell carcinoma of right lower limb (disorder) Merkel cell carcinoma of skin (disorder) Merkel cell carcinoma of skin (disorder) Primary malignant sarcoma of skin (disorder) Mersel cell carcinoma of skin (disorder) Mersel cell carcinoma of skin (disorder) Mersel cell carcinoma of skin (disorder) Merkel cell carcinoma of skin (disorder) Mersel cell carcinoma of skin (disorder) | | Basal cell carcinoma with matrical differentiation |
| A02541009 Basal cell carcinoma with sebaceous differentiation (morphologic abnormality) | 399958006 | (morphologic abnormality) |
| Basal cell carcinoma with sebaceous differentiation (morphologic abnormality) 402545000 Basal cell carcinoma - second recurrence (disorder) Basal cell carcinoma of obverse of pinna (disorder) Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma with sarcomatoid differentiation (morphologic abnormality) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel's cell (cell) 253001006 Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) 33841000119105 Merkel cell carcinoma of lower limb (disorder) 133871000119100 Merkel cell carcinoma of lower limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 352071000119105 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 721541009 Primary malignant sarcoma of skin (disorder) A04093001 Sarcomatous metastasis in skin (disorder) Mycosis fungoides (morphologic abnormality) | | Basal cell carcinoma recurrent following curettage |
| 40087001 (morphologic abnormality) 402545000 Basal cell carcinoma - second recurrence (disorder) 402514004 Basal cell carcinoma of obverse of pinna (disorder) 402542002 (disorder) Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma with sarcomatoid differentiation (morphologic abnormality) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma recurrent following radiotherapy (disorder) Basal cell carcinoma of eyelid (situation) 402543007 Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) Merkel cell carcinoma of face (disorder) 13841000119108 History of merkel cell carcinoma (situation) 133881000119100 Merkel cell carcinoma of lower limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 352071000119105 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of fecting skin (disorder) 40403001 Sarcomatous metastasis in skin (disorder) 40403001 Mycosis fungoides (morphologic abnormality) | 402541009 | (disorder) |
| Basal cell carcinoma - second recurrence (disorder) | | Basal cell carcinoma with sebaceous differentiation |
| Basal cell carcinoma of obverse of pinna (disorder) | 400087001 | (morphologic abnormality) |
| Basal cell carcinoma recurrent following cryotherapy (disorder) Basal cell carcinoma with sarcomatoid differentiation (morphologic abnormality) Basal cell carcinoma recurrent following radiotherapy (disorder) 69411000119107 History of basal cell carcinoma of eyelid (situation) 402511007 Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel cell carcinoma (disorder) 10149001 Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 13881000119100 Merkel cell carcinoma of lower limb (disorder) 13881000119100 Merkel cell carcinoma of lower limb (disorder) 352071000119103 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) | 402545000 | Basal cell carcinoma - second recurrence (disorder) |
| A02542002 | 402514004 | Basal cell carcinoma of obverse of pinna (disorder) |
| Basal cell carcinoma with sarcomatoid differentiation (morphologic abnormality) Basal cell carcinoma recurrent following radiotherapy (disorder) 69411000119107 History of basal cell carcinoma of eyelid (situation) 402511007 Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 1338141000119108 History of merkel cell carcinoma (situation) 133871000119103 Merkel cell carcinoma of lower limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 352071000119105 Merkel cell carcinoma of right lower limb (disorder) 351461000119100 Merkel cell carcinoma of skin (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 25480003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) | | Basal cell carcinoma recurrent following cryotherapy |
| 816972004 (morphologic abnormality) Basal cell carcinoma recurrent following radiotherapy (disorder) 69411000119107 History of basal cell carcinoma of eyelid (situation) 402511007 Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 13881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of left lower limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 50120004 Mycosis fungoides (morphologic abnormality) | 402542002 | |
| Basal cell carcinoma recurrent following radiotherapy (disorder) 69411000119107 History of basal cell carcinoma of eyelid (situation) 402511007 Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) 10149001 Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 138141000119108 History of merkel cell carcinoma (situation) 133871000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of left lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 524800003 Epithelioid cell sarcoma affecting skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) Mycosis fungoides (morphologic abnormality) | | |
| 402543007 (disorder) 69411000119107 History of basal cell carcinoma of eyelid (situation) 402511007 Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 138814000119108 History of merkel cell carcinoma (situation) 133881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 25480003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | 816972004 | |
| 69411000119107 History of basal cell carcinoma of eyelid (situation) 402511007 Basal cell carcinoma of conchal bowl of ear (disorder) Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) Merkel's cell (cell) Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 133841000119108 History of merkel cell carcinoma (situation) 133871000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of left lower limb (disorder) 352071000119105 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 25480003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | | |
| Basal cell carcinoma of conchal bowl of ear (disorder) | | |
| Basal cell carcinoma recurrent following Mohs' excision (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) 10149001 Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 138141000119108 History of merkel cell carcinoma (situation) 133881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) Epithelioid cell sarcoma of skin (disorder) Sarcomatous metastasis in skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) Mycosis fungoides (morphologic abnormality) | | |
| 402540005 (disorder) Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) 10149001 Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 133881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of right lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | 402511007 | · · · |
| Excision of postauricular basal cell carcinoma with closure (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) 10149001 | 402540005 | • |
| 703499006 (procedure) Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) 10149001 Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 138141000119108 History of merkel cell carcinoma (situation) 133881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | 402540005 | |
| Basal cell carcinoma - multiple recurrences (more than three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) 10149001 Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 138141000119108 History of merkel cell carcinoma (situation) 133881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | 702400006 | |
| three times) (disorder) Excision of basal cell carcinoma from right postauricular region with closure (procedure) 10149001 | 703499000 | |
| Excision of basal cell carcinoma from right postauricular region with closure (procedure) 10149001 | 402547008 | · |
| 736465001region with closure (procedure)10149001Merkel's cell (cell)253001006Merkel cell carcinoma (disorder)5052009Merkel cell carcinoma (morphologic abnormality)133841000119105Merkel cell carcinoma of face (disorder)138141000119108History of merkel cell carcinoma (situation)133881000119100Merkel cell carcinoma of lower limb (disorder)133871000119103Merkel cell carcinoma of upper limb (disorder)352071000119105Merkel cell carcinoma of right lower limb (disorder)351461000119100Merkel cell carcinoma of right lower limb (disorder)721541009Primary malignant sarcoma of skin (disorder)109386008Kaposi's sarcoma of skin (disorder)254800003Epithelioid cell sarcoma of skin (disorder)404093001Sarcomatous metastasis in skin (disorder)404155008Granulocytic sarcoma affecting skin (disorder)90120004Mycosis fungoides (morphologic abnormality) | 402347000 | |
| 10149001 Merkel's cell (cell) 253001006 Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 138141000119108 History of merkel cell carcinoma (situation) 133881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | 736465001 | |
| 253001006 Merkel cell carcinoma (disorder) 5052009 Merkel cell carcinoma (morphologic abnormality) 133841000119105 Merkel cell carcinoma of face (disorder) 138141000119108 History of merkel cell carcinoma (situation) 133881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | | |
| 5052009Merkel cell carcinoma (morphologic abnormality)133841000119105Merkel cell carcinoma of face (disorder)138141000119108History of merkel cell carcinoma (situation)133881000119100Merkel cell carcinoma of lower limb (disorder)133871000119103Merkel cell carcinoma of upper limb (disorder)352071000119105Merkel cell carcinoma of left lower limb (disorder)351461000119100Merkel cell carcinoma of right lower limb (disorder)721541009Primary malignant sarcoma of skin (disorder)109386008Kaposi's sarcoma of skin (disorder)254800003Epithelioid cell sarcoma of skin (disorder)404093001Sarcomatous metastasis in skin (disorder)404155008Granulocytic sarcoma affecting skin (disorder)90120004Mycosis fungoides (morphologic abnormality) | | |
| 133841000119105 Merkel cell carcinoma of face (disorder) 138141000119100 History of merkel cell carcinoma (situation) 133881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | | |
| 138141000119108 History of merkel cell carcinoma (situation) 133881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | | , 1 0 |
| 133881000119100 Merkel cell carcinoma of lower limb (disorder) 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | | |
| 133871000119103 Merkel cell carcinoma of upper limb (disorder) 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | | |
| 352071000119105 Merkel cell carcinoma of left lower limb (disorder) 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | | |
| 351461000119100 Merkel cell carcinoma of right lower limb (disorder) 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | | |
| 721541009 Primary malignant sarcoma of skin (disorder) 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | | |
| 109386008 Kaposi's sarcoma of skin (disorder) 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | 721541009 | |
| 254800003 Epithelioid cell sarcoma of skin (disorder) 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | 109386008 | |
| 404093001 Sarcomatous metastasis in skin (disorder) 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | 254800003 | |
| 404155008 Granulocytic sarcoma affecting skin (disorder) 90120004 Mycosis fungoides (morphologic abnormality) | | |
| 90120004 Mycosis fungoides (morphologic abnormality) | | |
| | | Mycosis fungoides (disorder) |

| 765328000 | Classic mycosis fungoides (disorder) |
|-----------------|-----------------------------------------------------------|
| 404115006 | Bullous mycosis fungoides (disorder) |
| 94714002 | Mycosis fungoides of spleen (disorder) |
| 404117003 | Spongiotic mycosis fungoides (disorder) |
| 681291000119105 | History of mycosis fungoides (situation) |
| 418628003 | Follicular mycosis fungoides (morphologic abnormality) |
| 404113004 | Tumour stage mycosis fungoides (disorder) |
| 404118008 | Syrngotropic mycosis fungoides (disorder) |
| 404112009 | Granulomatous mycosis fungoides (disorder) |
| 404114005 | Erythrodermic mycosis fungoides (disorder) |
| 404110001 | Hypomelanocytic mycosis fungoides (disorder) |
| 404109006 | Folliculotropic mycosis fungoides (disorder) |
| 404108003 | Pokilodermatous mycosis fungoides (disorder) |
| 404107008 | Patch/plaque stage mycosis fungoides (disorder) |
| 404116007 | Mycosis fungoides with systemic infiltration (disorder) |
| 94708009 | Mycosis fungoides of intrapelvic lymph nodes (disorder) |
| 34700003 | Mycosis fungoides of intra-abdominal lymph nodes |
| 94707004 | (disorder) |
| 34707004 | Mycosis fungoides of lymph nodes of multiple sites |
| 188627002 | (disorder) |
| 100027002 | Lymphomatoid papulosis-associated mycosis fungoides |
| 404111002 | (disorder) |
| 707111002 | Lymphomatoid papulosis type B mycosis fungoides-like |
| 404104001 | (disorder) |
| | Mycosis fungoides of extranodal AND/OR solid organ site |
| 94715001 | (disorder) |
| 94709001 | Mycosis fungoides of intrathoracic lymph nodes (disorder) |
| | Mycosis fungoides of lymph nodes of head, face AND/OR |
| 94711005 | neck (disorder) |
| | Mycosis fungoides of lymph nodes of axilla AND/OR upper |
| 94710006 | limb (disorder) |
| | Mycosis fungoides of lymph nodes of multiple sites |
| 188627002 | (disorder) |
| | Mycosis fungoides of lymph nodes of inguinal region |
| 94712003 | AND/OR lower limb (disorder) |
| | Cutaneous T-cell lymphoma, no International Classifcation |
| | of Diseases for oncology subtype (morphologic |
| 28054005 | abnormality) |
| 40012207 | Primary cutaneous T-cell lymphoma (disorder) |
| 277613000 | Cutaneous/peripheral T-cell lymphoma (disorder) |
| 404128004 | CD-30 negative cutanoeus T-cell lymphoma (disorder) |
| | Primary cutaneous T-cell lymphoma - category |
| 419283005 | (morphologic abnormality) |
| | Primary cutaneous CD30 antigen positive T-cell |
| 128804002 | lymphoproliferative disorder (morphologic abnormality) |
| 45000000 | Primary cutaneous gamma-delta T-cell lymphoma |
| 450908002 | (morphologic abnormality) |
| 122571000119106 | History of primary cutaneous T-cell lymphoma (situation) |
| 44.004.0000 | Primary cutaneous large T-cell lymphoma - category |
| 419018000 | (morphologic abnormality) |

| 402880009 | Primary cutaneous large T-cell lymphoma (disorder) |
|-----------------|------------------------------------------------------------|
| | Subcutaneous panniculitic cutaneous T-cell lymphoma |
| 404133000 | (disorder) |
| 404128004 | CD-30 negative cutaneous T-cell lymphoma (disorder) |
| | Primary cutaneous acral CD8 positive T-cell lymphoma |
| 787198005 | (morphologic abnormality) |
| | Primary cutaneous anaplastic large T-cell lymphoma, CD30- |
| 397352006 | positive (morphologic abnormality) |
| | Primary cutaneous gamma-delta-positive T-cell lymphoma |
| 733627006 | (disorder) |
| | CD-30 negative anaplastic large T-cell cutaneous lymphoma |
| 404129007 | (disorder) |
| 122571000119106 | History of malignant cutaneous T-cell lymphoma (situation) |
| | CD-30 negative pleomorphic large T-cell cutaneous |
| 404130002 | lymphoma (disorder) |
| | CD-30 positive pleomorphic large T-cell cutaneous |
| 404126000 | lymphoma (disorder) |
| | Primary cutaneous T-cell lymphoma - category |
| 419283005 | (morphologic abnormality) |
| | Primary cutaneous gamma-delta T-cell lymphoma - |
| 450908002 | category (morphologic abnormality) |
| | Primary cutaneous CD8 positive aggressicve |
| 765136002 | epidermotropic cytotoxic T-cell lymphoma (disorder) |
| | Primary cutaneous CD30 antigen positive large T-cell |
| 128875000 | lymphoma (disorder) |
| | Primary cutaneous CD8 positive aggressicve |
| | epidermotropic cytotoxic T-cell lymphoma (morphologic |
| 733895005 | abnormality) |
| | Primary cutaneous T-cell lymphoma, large cell, CD30- |
| 419586003 | negative (morphological abnormality) |
| 118611004 | Sezary's disease (disorder) |
| 4950009 | Sezary's disease (morphologic abnormality) |
| 255101006 | Sezary disease of skin (disorder) |
| 95263006 | Sezary's disase of spleen (disorder) |
| 188632001 | Sezary's disase of intra-abdominal lymph nodes (disorder) |
| 188635004 | Sezary's disase of intrapelvic lymph nodes (disorder) |
| 188631008 | Sezary's disase of intrathoracic lymph nodes (disorder) |
| 188637007 | Sezary disease of lymph nodes of multiple sites (disorder) |
| | Sézary's disease of extranodal AND/OR solid organ site |
| 95264000 | (disorder) |
| | Sézary's disease of lymph nodes of axilla and upper limb |
| 188633006 | (disorder) |
| | Sézary's disease of lymph nodes of head, face AND/OR neck |
| 95260009 | (disorder) |
| | Sézary's disease of lymph nodes of inguinal region and |
| 188634000 | lower limb (disorder) |
| | Sézary's disease of lymph nodes of inguinal region AND/OR |
| 95261008 | lower limb (disorder) |
| 419392005 | Primary cutaneous lymphoma (morphologic abnormality) |